

## **Motif BioSciences**

Protocol No.: ICL-24-ABSSSI2

A Phase 3, randomized double-blind, multicenter study to evaluate the safety and efficacy of intravenous iclaprim versus vancomycin in the treatment of acute bacterial skin and skin structure infections suspected or confirmed to be due to Gram-positive pathogens. (REVIVE-2)

**Covance Study ID: 000000145670** 

STATISTICAL ANALYSIS PLAN

Draft Amendment 2.0 Date of Issue: 24 July2017

**Author: Alyssa Liu** 

**Motif BioSciences** 125 Park Avenue, 25<sup>th</sup> Floor, Suite 2622 New York, NY 10017 Covance Clinical Development Services 206 Carnegie Center Princeton, NJ 08540

Version: Draft Amendment 2.0 Motif BioSciences Protocol No. ICL-24-ABSSSI2 Date of Issue: 24 July2017 Covance Study ID: 000000145416

## **APPROVALS**

The undersigned agree that all required reviews of this document are complete, and approve this Statistical Analysis Plan as final. Programming of the tables, figures and listings based upon the specifications within this document can proceed.

| and document can proceed. | |
|---|---|
| Covance Approval: | |
| Tofoles Opean | 24 July 2017 |
| Signature | Date // |
| Toyoko Oguri/Senior Manager, Biostatistical and Statistical Programming | |
| Printed Name/Title | |
| Motif BioSciences Approval: | |
| Man jed Markes | July 24, 2017 |
| Signature / | Date / |
| Rajesh Shukla/Vice President of Clinical Operations | |
| Printed Name/Title | |

**Version: Draft Amendment 2.0**Motif BioSciences Protocol No. ICL-24-ABSSSI2

Date of Issue: 24 July2017 Covance Study ID: 000000145416

# **VERSION HISTORY**

| Version Number | Version Date | Summary and rational of change(s) |
|---|---|---|
| Final 1.0 | 17-Aug-2016 | |
| Amendment 1.0 | 12-Jan-2017 | Section 2.3 (Sample Size and Power) • Revised power assumption related to TOC visit. |
| | | <ul> <li>Section 3.2 (Secondary Efficacy Endpoints)</li> <li>The order of PP population and mCE population was changed.</li> <li>Two definitions of "Persistent Infection" and "Recurrent Infection" were added when defining clinical failure.</li> </ul> |
| | | Section 5 (Analysis Population) • The order of PP population and mCE population was changed. |
| | | <ul> <li>Section 6.2 (Handling of Dropouts or Missing Data)</li> <li>Added mITT efficacy analyses for primary endpoint, while patients who do not have an adequate assessment at the appropriate visit assumed as non-responders.</li> </ul> |
| | | Section 7.2 (Patient Disposition and Data Sets Analysed) • The order of PP population and mCE population was changed. |
| | | <ul> <li>Section 7.4 (Demographics and Other Baseline Characteristics)</li> <li>The order of PP population and mCE population was changed.</li> <li>Added two demographic variables, diabetes (present or absent) and geographic region (US vs ex-US).</li> </ul> |
| | | Section 7.7 (Measurements of Treatment Compliance and Exposure) • Clarify the treatment is started in the AM and completed in the PM when patients are administered with iclaprim q12h for 5 to 14 days. |
| | | Section 7.8.2.2 (Time to Resolution of Signs and Symptoms of ABSSSI) • The order of PP population and mCE population was changed. |
| | | <ul> <li>Section 7.8.3 (Exploratory Analysis)</li> <li>For primary endpoint, added exploratory analysis for ITT population with ≥50%, ≥75%, and ≥90% reduction in lesion size at ETP compared from baseline.</li> <li>For the secondary endpoint of resolution or near resolution of ABSSSI at EOT and TOC, added exploratory analysis for ITT population with at least 50% and at least 75% reduction in lesion size at both EOT and TOC compared from baseline.</li> <li>If it is concluded that Iclaprim is non-inferior to Vancomycin (i.e., the lower bound of two-sided 95% confidence interval of group difference in early clinical response is greater than -0.1), it may be concluded that Iclaprim is superior to Vancomycin if the entire 95% confidence interval is &gt;0. Superiority may also be</li> </ul> |

Date of Issue: 24 July2017 Covance Study ID: 000000145416

## Statistical Analysis Plan

**Version: Draft Amendment 2.0** Motif BioSciences Protocol No. ICL-24-ABSSSI2

Version Number **Summary and rational of change(s) Version Date** concluded for resolution of ABSSSI at TOC in a similar manner. Section 7.8.4 (Subgroup Analysis) • Added two demographic variables for subgroup analysis: diabetes (present or absent) and geographic region (US vs ex-

| | | US). |
|---|---|---|
| | | <ul> <li>Section 7.9.1 (Adverse Events)</li> <li>Added another summary of TEAEs by diabetes (present or absent).</li> <li>Added the definition of SAE.</li> </ul> |
| | | Section 7.9.2 (Laboratory Evaluations) • Parameter of CRP was updated from category of haematology to chemistry. |
| | | Section 7.10 (Interim Analysis) • Clarified analysis for the primary endpoint under blinded interim data was using at least 20% reduction in lesion size at ETP when compared to baseline visit. |
| | | Section 7.10.2 (Laboratory Evaluations) • Add another kind of shift table between baseline and post-baseline change, only applied for liver enzyme and renal function tests. |
| Amendment 1.0 | 15–Feb-2017 | Table 1 Summary of Assessments was deleted. Same information is given in the text and it is a copy from protocol. |
| | | Section 4 (Pharmacokinetics/ Pharmacodynamics Variables) |
| | | <ul> <li>Deleted "After the study is complete, the database locked, and<br/>the data unblinded, patients randomized to iclaprim will have<br/>their samples assayed."</li> </ul> |
| | | Section 5 (Analysis Population) |
| | | Added details to Per Protocol population definition. |
| | | • Table 1 reformatted to separate protocol deviation types that would exclude a patient from some visits and visits from deviation types that excludes a patient from all visits. |
| | | <ul> <li>Deleted Type I A and Type III antiarrhythmic drugs from list<br/>of prohibited medications that would exclude a patient from<br/>per protocol analysis.</li> </ul> |
| | | Added mITT subpopulation, strep-enriched mITT for exploratory analysis. |
| | | Added PP population for EMA analysis. |
| | | Section 5.6.1 Important Protocol Deviations Leading to Exclusion from the mPP Analysis. |
| | | This section was deleted because it provides some |
| | | COVANCE INC. CONFIDENTIAL |

**Version: Draft Amendment 2.0**Motif BioSciences Protocol No. ICL-24-ABSSSI2

**Date of Issue: 24 July2017** Covance Study ID: 000000145416

| Version Number | Version Date | Summary and rational of change(s) |
|---|---|---|
| | | information as in PP population. |
| | | Section 6.1 (Time Points and Visit Widows) |
| | | Baseline for microbiology analysis was added. |
| | | 7.4 (Demographic and Other Baseline Characteristics) |
| | | <ul> <li>Blood culture at baseline was defined;</li> </ul> |
| | | Geographic region subgroups were revised |
| | | 7.9.2 (Secondary Efficacy Analysis) |
| | | • Added <i>S. pyogenes</i> -enriched mITT population and PP population for EMA to repeat the primary efficacy analysis. |
| | | 7.9.2.1 (Resolution or Near Resolution of ABSSSI) |
| | | • Added S. pyogenes-enriched mITT at TOC to the analysis |
| | | 7.9.2.2 (Signs and Symptoms of ABSSSI) |
| | | <ul> <li>Descriptive summary statistics for signs and symptoms will<br/>be limited to baseline display only.</li> </ul> |
| | | 7.9.2.3 (Bacteriological response) |
| | | • By-pathogen and by-patient bacteriological outcome section were moved from Section 3 to this section. |
| | | <ul> <li>Added more description of analyses.</li> </ul> |
| | | <ul> <li>Added summary of MIC frequency and interpretation.</li> </ul> |
| | | 7.10.1 (Adverse Events) |
| | | • Treatment-emergent adverse event definition was clarified. |
| Amendment 2.0 | 10-Mar-2017 | 6.1 (Time Points and Visit Windows) |
| | | Added definition of baseline for microbiology data. |
| | | 6.2 (Handling of Dropouts or Missing Data) |
| | | <ul> <li>Deleted general principle for imputing dates and clarified the<br/>imputing details refer to mockup.</li> </ul> |
| | | 7.6 (Prior and Concomitant Medications) |
| | | Added the definition of prior medication. |
| | | 7.9.2.2 (Signs and Symptoms of ABSSSI) |
| | | • Clarified patients are free of specific signs or symptoms at baseline should be out of that time-to-event analysis. |

**Version: Draft Amendment 2.0** 

**Date of Issue: 24 July2017** Covance Study ID: 000000145416 Motif BioSciences Protocol No. ICL-24-ABSSSI2

| | 7.9.3 (Exploratory Analysis) |
|---|---|
| | <ul> <li>Revised the definition for one exploratory analysis and added<br/>another exploratory analysis.</li> </ul> |
| | 7.10.1 (Adverse Events) |
| | • Treatment-emergent adverse event definition was clarified. |
| 11 July 2017 | <ul> <li>7.9.3.1 (Exploratory Analysis Excluding Lesion Size Criteria)</li> <li>New section to describe analysis excluding the criteria for lesion size reduction for the following exploratory analyses: <ul> <li>Resolution or near resolution of ABSSSI</li> <li>Clinical outcome</li> <li>By-pathogen bacteriological response</li> <li>By-patient bacteriological response</li> </ul> </li> </ul> |
| | 7.4 (Demographic and Other Baseline Characteristics) |
| | Age is obtained from IXRS rather than derived. |
| | <ul> <li>Defined Gram-positive pathogen groups.</li> </ul> |
| | <ul> <li>Defined categories of severe infection.</li> </ul> |
| | 7.9.2.1 (Resolution or Near Resolution of ABSSSI) |
| | <ul> <li>Add categories of cure criteria in each analysis</li> </ul> |
| | 7.2.9.2 (Signs and Symptoms of ABSSSI) |
| | <ul> <li>Add categories of intensity to each sign and symptom.</li> </ul> |
| | 7.9.4 (Subgroup Analysis) |
| | <ul> <li>Add categories of severe infection.</li> </ul> |
| | 7.10.1 (Adverse Events) |
| | <ul> <li>Add summary of SAE &gt; 1%</li> </ul> |
| | 7.10.2 (Laboratory Evaluations) |
| | • Add grade 0 (<= ULN) |
| | Add description of urinalysis categorical summary |
| 21 July 2017 | 7.9.3.1 (Exploratory Analysis Excluding Lesion Size Criteria) |
| | <ul> <li>Revised definition of persistent and recurrent infection</li> </ul> |
| | <ul> <li>Clarified definition of unplanned significant procudures<br/>(throughout the SAP)</li> </ul> |

**Version: Draft Amendment 2.0**Motif BioSciences Protocol No. ICL-24-ABSSSI2

## **Date of Issue: 24 July2017** Covance Study ID: 000000145416

## **TABLE OF CONTENTS**

| Al | PPRC | OVALS | 2 |
|---|---|---|---|
| V | ERSI | ON HISTORY | 3 |
| <b>G</b> ] | LOSS | SARY OF ABBREVIATIONS | 9 |
| 1 | SOI | URCE DOCUMENTS | 11 |
| 2 | | OTOCOL DETAILS | |
| _ | 2.1 | Study Objectives | |
| | 2.2 | Overall Study Design | |
| | 2.3 | Sample Size and Power | |
| 3 | EFF | FICACY AND SAFETY VARIABLES | |
| | 3.1 | Primary Efficacy Endpoint | |
| | 3.2 | Secondary Efficacy Endpoints | |
| | 3.3 | Safety Variables | |
| 4 | PHA | ARMACOKINETIC/PHARMACODYNAMIC VARIABLES | 15 |
| 5 | ANA | ALYSIS POPULATIONS | 15 |
| | <b>5.1</b> | Safety Population | 15 |
| | <b>5.2</b> | Intent-to-treat (ITT) population | 15 |
| | <b>5.3</b> | Microbiological intent-to-treat (mITT) population | 15 |
| | <b>5.4</b> | Per Protocol (PP) Population | 16 |
| | | 5.4.1 Important Protocol Deviations Leading to Exclusion from the PP Analysis | |
| | <b>5.5</b> | Modified clinically evaluable (mCE) population | |
| | <b>5.6</b> | PP microbiological evaluable (mPP) population | |
| | <b>5.7</b> | S. pyogenes-enriched mITT (S. pyogenes mITT) population | |
| | <b>5.8</b> | PP population for EMA sensitivity analysis | 18 |
| 6 | DA | ΓA HANDLING | |
| | 6.1 | Time Points and Visit Windows | |
| | <b>6.2</b> | Handling of Dropouts or Missing Data | 19 |
| 7 | STA | ATISTICAL METHODS | 19 |
| | <b>7.1</b> | General Principles | 19 |
| | <b>7.2</b> | Patient Disposition and Data Sets Analyzed | 20 |
| | <b>7.3</b> | Protocol Deviations | |
| | 7.4 | Demographics and Other Baseline Characteristics | |
| | 7.5 | Medical History | |
| | <b>7.6</b> | Prior and Concomitant Medications | |
| | 7.7 | Significant Procedures | |
| | <b>7.8</b> | Measurements of Treatment Compliance and Exposure | 22 |

| Version: | Draft A | mendm | ent 2. | 0 | | |
|-----------|----------|---------|--------|------|-------|-------|
| Motif Bio | Sciences | Protoco | ol No. | ICL- | 24-AB | SSSI2 |

Date of Issue: 24 July2017 Covance Study ID: 000000145416

| | <b>7.9</b> | Efficac | ·y | 22 |
|---|---|---|---|---|
| | | | Primary Efficacy Analysis | |
| | | 7.9.2 | Secondary Efficacy Analysis | 22 |
| | | 7.9.3 | Exploratory Analysis | 24 |
| | | 7.9.4 | Subgroup Analysis | 26 |
| | 7.10 | Safety | | 27 |
| | | | Adverse Events | |
| | | 7.10.2 | Laboratory Evaluations | 28 |
| | | 7.10.3 | Vital Signs | 29 |
| | | 7.10.4 | Electrocardiograms | 29 |
| | | 7.10.5 | Physical Examination | 30 |
| | <b>7.11</b> | Interin | n Analysis | 30 |
| 8 | REF | ERENC | CES | 30 |
| 9 | APP | ENDIC | ES | 31 |
| | | | - Prohibited Medicines | |
| | | | - Schedule of Events | |
| | | | - Table, Figure and Listing Shells | |
| TA | ABLE | S: | | |
| Ta | ble 1: | Importa | ant Protocol Deviations Leading to Exclusion from the PP population | 17 |
| Ta | ble 2: | Laborat | ory Evaluations | 28 |
| FI | GUR | ES: | | |
| Fi | oure 1 | · Study ] | Design | 13 |

**Version: Draft Amendment 2.0**Motif BioSciences Protocol No. ICL-24-ABSSSI2

**Date of Issue: 24 July2017** Covance Study ID: 000000145416

## **GLOSSARY OF ABBREVIATIONS**

| Abbreviation | Term |
|--------------|-----------------------------------------------------|
| ABSSSI | acute bacterial skin and skin structure infection |
| AE | adverse event |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase |
| ASO | anti-streptolysin O |
| AST | aspartate aminotransferase |
| ATC | Anatomical Therapeutic Chemical |
| BMI | Body Mass Index |
| BUN | blood urea nitrogen |
| CBC | complete blood count |
| CCLS | Covance Central Laboratory Services |
| CI | confidence interval |
| $CO_2$ | carbon dioxide |
| CPK | creatine phosphokinase |
| CrCL | creatinine clearance |
| CRF | case report form |
| CRP | C-reactive protein |
| CTMS | Clinical Trial Management System |
| CV | Conventional units for laboratory results |
| ECG | Electrocardiogram |
| eCRF | electronic case report form |
| EOT | End of Therapy |
| EMA | European Medicines Agency |
| ETP | early timepoint |
| GGT | gamma glutamyl transferase |
| hCG | beta-human chorionic gonadotropin |
| ITT | intent-to-treat |
| IXRS | Interactive Phone and Web Response System |
| LDH | lactate dehydrogenase |
| LFT | Liver Function Test |
| LFU | Late Follow-Up |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MIC | minimum inhibitory concentration |
| MRSA | Methicillin-resistant Staphylococcus aureus |
| MSSA | Methicillin-sensitive Staphylococcus aureus |
| mCE | Modified clinically evaluable population |
| mITT | microbiological intent-to-treat |
| mPP | Per-protocol microbiologically evaluable population |
| N | analysis population |

**Version: Draft Amendment 2.0** 

Motif BioSciences Protocol No. ICL-24-ABSSSI2

**Date of Issue: 24 July2017** Covance Study ID: 000000145416

| Abbreviation | Term |
|--------------|--------------------------------------------|
| NI | non-inferiority |
| PK | pharmacokinetic |
| PP | Per-protocol population |
| PT | Preferred Term |
| Q12h | every 12 hours |
| QTc | QT interval corrected for heart rate |
| QTcB | QTc corrected according to Bazett |
| QTcF | QTc corrected according to Fridericia |
| RBC | red blood cell |
| SAE | serious adverse event |
| SCr | serum creatinine |
| SD | standard deviation |
| SI Units | International System of Units |
| SOC | system organ class (MedDRA classification) |
| TEAE | treatment-emergent adverse event |
| TFLs | Tables, Figures and Listings |
| TOC | Test of Cure |
| UA | Urinalysis |
| WBC | white blood cells |

Version: Draft Amendment 2.0

Motif BioSciences Protocol No. ICL-24-ABSSSI2

Date of Issue: 24 July2017

Covance Study ID: 000000145416

#### 1 SOURCE DOCUMENTS

The Statistical Analysis Plan (SAP) was written based on the following documentation:

| Document | Date | Version |
|----------------------|-------------|----------------|
| Protocol | 21 Oct 2015 | Final 1.0 |
| Protocol Amendment 1 | 3 Dec 2015 | Amendment 1.0 |
| eCRF | 3 Feb 2016 | Production 3.0 |

#### 2 PROTOCOL DETAILS

#### 2.1 Study Objectives

Primary Objective:

The primary objective of this study is to demonstrate that iclaprim is non-inferior to vancomycin in achieving a  $\geq$  20% reduction in lesion size at 48 to 72 hours (early timepoint, ETP) compared to baseline in all randomized patients (intent-to-treat, ITT).

Secondary Objectives:

The secondary objectives of this study are to demonstrate non-inferiority of iclaprim compared to vancomycin in the ITT, microbiological ITT (mITT), modified clinically evaluable (mCE), per protocol (PP), and microbiological PP (mPP) populations for the following:

- 1. Resolution or near resolution of acute bacterial skin and skin structure infection (ABSSSI) (clinical cure, defined by a ≥ 90% reduction in lesion size from the size at baseline, no increase in lesion size since ETP, and no requirement for additional antibiotics [except aztreonam and metronidazole] or unplanned significant surgical procedures [excluding procedures that reflect failure of antimicrobial therapy] after ETP other than bedside wound care) at Test of Cure (TOC) visit (7 to14 days after the end of treatment);
- 2. Resolution or near resolution ( $\geq 90\%$ ) of ABSSSI at End of Therapy (EOT);
- 3. Resolution or near resolution (≥ 90%) of ABSSSI at EOT and TOC among patients with severe infection at baseline defined by meeting one or more of the following criteria:
  - a. fulfilled the published definition for systemic inflammatory response syndrome (SIRS) by having  $\geq 2$  of the following findings: body temperature  $> 38^{\circ}\text{C}$  or  $< 36^{\circ}\text{C}$ , heart rate > 90 bpm, respiration rate > 20 breaths/minute, and WBC  $> 12000/\text{mm}^3$  or  $< 4000/\text{mm}^3$  or > 10% bands;
  - b. Evaluated as having severe tenderness or severe erythema at the infection site; or
  - c. Positive blood cultures at baseline.
- 4. Time to resolution of systemic and local signs and symptoms of ABSSSI.

Additional secondary objectives are to:

- 5. Assess microbiological outcome in the mITT, mCE, and mPP populations at EOT and TOC;
- 6. Establish the pharmacokinetic (PK) profile for iclaprim using population pharmacokinetics; and
- 7. Establish the safety profile of iclaprim in patients with ABSSSI.

#### 2.2 Overall Study Design

This is a multicenter, randomized, double-blind study of the efficacy and safety of iclaprim compared to vancomycin. Patients will receive either iclaprim or vancomycin for 5 to 14 days, which comprises the range of total treatment duration. Patients will be evaluated daily up to ETP, then every 48 to 72 hours through the end of treatment. If the last dose of study drug falls on a day when an evaluation was not

Covance Study ID: 000000145416

#### **Statistical Analysis Plan**

Version: Draft Amendment 2.0 Motif BioSciences Protocol No. ICL-24-ABSSSI2

planned, an additional evaluation visit will need to be performed on that day (i.e. All EOT evaluations should be performed on the last day [+2 days] of drug dose). Patients will also be evaluated at the TOC visit (7 to 14 days post-EOT) for both efficacy and safety, and will have a Late Follow-Up (LFU) phone

call (28 to 32 days post-first dose) for safety only. Note, however, that patients with high liver function tests (LFTs) and unresolved adverse events (AEs) at TOC must be seen in person for an additional visit at LFU. The total duration of participation in the study for each patient is 29 to 33 days.

After completing screening procedures, including obtaining cultures from a clinical specimen prior to antibacterial therapy, a total of 600 patients (300 per treatment group) will be randomized (1:1) to receive either: (1) iclaprim 80 mg every 12 hours or (2) vancomycin 15 mg/kg. The duration of treatment for both groups will be 5 days (minimum duration) to 14 days (maximum duration). Assignment to study drug will be performed using a central randomization system. Approximately 80 active centers will be recruited.

Figure 1 displays a diagram of the study design.

The investigators, clinical study personnel, sponsor, and the patients will remain blinded with respect to the study drug treatment allocation. The unblinded pharmacist or his/her designee will be responsible for preparation of infusions. To account for the variable vancomycin dosing intervals, normal saline dummy infusions will be used to maintain the blind for patients who require a vancomycin dosing frequency other than every 12 hours (Q12h).

Concomitant antibiotics aztreonam and metronidazole used in compliance with their respective prescribing information are allowed at the discretion of the investigator during the study drug phase.

Systemic antibiotics (other than aztreonam and metronidazole) or topical antibiotics at the site of the ABSSSI under investigation, steroids >20 mg/day prednisolone or equivalent; and Type I A and Type III-antiarrhythmic drugs are prohibited.

#### 2.3 Sample Size and Power

For non-inferiority (NI) testing with a 1-sided alpha of 0.025, assuming a 75% early clinical response rate in each group and a 10% NI bound delta, a sample size of 295 ITT patients per treatment group is required for 80% power. In addition, using similar methods of NI testing with a 1-sided alpha of 0.025, assuming a 90% clinical response rate at TOC in vancomycin and iclaprim group and a 10% NI bound delta, a sample size of 300 patients in the ITT population per treatment group is required for 98% power.

A total of 600 patients (approximately 300 per treatment group) will be randomized (1:1) for this study.

**Date of Issue: 24 July 2017**Covance Study ID: 000000145416



Note: A window of +/-2 hours is acceptable for infusion of study medication.

- 1. ETP assessment is 48 to 72 hours post-first dose
- 2. If the last dose of study drug falls on a day when an evaluation was not planned, an additional evaluation visit will need to be performed on that day (ie. All EOT evaluations should be performed on the last day [+/- 2 days] of drug dose).
- 3. If duration of therapy is 14 days, LFU may overlap with TOC. In this case, all LFU evaluations may take place at the TOC visit. Vn=Visit n; ETP=Early Time Point; EOT=End of Therapy; TOC=Test of Cure; LFU=Late Follow-up

Version: Final Amendment 2.0

Date of Issue: 24 July 2017 Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

#### 3 EFFICACY AND SAFETY VARIABLES

#### 3.1 **Primary Efficacy Endpoint**

The primary efficacy endpoint is the proportion of randomized patients who achieve an early clinical response (defined as reduction in the lesion size  $\geq$  20% compared to baseline) at 48 to 72 hours (ETP) and will be evaluated in ITT population.

#### 3.2 Secondary Efficacy Endpoints

The primary efficacy endpoint will be repeated in mITT, PP, mCE and mPP populations.

The secondary endpoints are:

- 1. Resolution or near resolution of ABSSSI (i.e., Clinical Cure, defined by a > 90% reduction in lesion size from baseline, no increase in lesion size since ETP, and no requirement for additional antibiotics [except aztreonam and metronidazole] or unplanned significant surgical procedures [excluding procedures that reflect failure of antimicrobial therapy] after ETP other than bedside wound care) at TOC for iclaprim (80 mg q12h) compared with vancomycin (weight-based dose) for ITT, mITT, PP, mCE, and mPP populations
- 2. Resolution or near resolution (≥ 90%) of ABSSSI at EOT for ITT, mITT, PP, mCE, and mPP populations
- 3. Resolution or near resolution (≥ 90%) of ABSSSI at EOT and TOC among patients with severe infection at baseline for ITT, mITT, mCE, PP, and mPP populations
- 4. Time to resolution of signs and symptoms of ABSSSI from start of treatment for ITT, mITT, PP, mCE, and mPP populations
- 5. Patient-level bacteriological response rate at EOT and TOC for mITT, mCE, and mPP populations
- 6. Pathogen-level bacteriological response rate at EOT and TOC for mITT, mCE, and mPP populations

The clinical outcome will be evaluated at EOT and TOC (7 to 14 days post-EOT) programmatically for ITT, PP and mPP populations, and categorized as cure, failure, or indeterminate defined as follows:

- Cure: defined by a > 90% reduction in lesion size from baseline, no increase in lesion size since ETP, and no requirement for additional antibiotics (except aztreonam and metronidazole) or unplanned significant surgical procedures (excluding procedures that reflect failure of antimicrobial therapy);
- Failure: reduction in lesion size that is < 20% for ETP and < 90% for EOT and TOC compared to baseline, death related to the infection, persisting or recurrent infection, need for unplanned surgical procedure (i.e., procedures that reflect failure of antimicrobial therapy), or administration of rescue antibiotic therapy for the index infection before or at assessed visits or recurrence of index infection;
- Indeterminate: data inadequate for assessment of efficacy (there are no post-baseline local or systemic signs and symptoms data available to make this assessment [e.g., patient lost to follow up] after < 2 days of treatment or < 4 doses and no EOT evaluation), lost to follow-up prior to ETP, withdrawal of consent, receipt of effective antibiotic therapy for a cause other than the index infection before assessed visits, or death not attributed to the index ABSSSI or complication of ABSSSI.

#### **Statistical Analysis Plan**

Motif RioSciences Protocol No. ICL-24-ABSSSI2

Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

**Note**: If a patient starts an antibiotic for an infection other than the primary ABSSSI at EOT visit date, they will still be included as clinical cure or clinical failure dependent on the size of the lesion at EOT. The same rule will be applied to the evaluation of clinical outcome at TOC visit.

The definition of "Persistent Infection" and "Recurrent infection" when defining clinical failure are listed as follows:

- (1) Persistent infection occurs if a patient receives additional antibiotics for treatment of primary ABSSSI (except aztreonam and metronidazole) at EOT compared to baseline. The same rule applies when evaluating clinical failure at TOC visit.
- (2) Recurrent infection occurs if a patient does not receive additional antibiotics (except aztreonam and metronidazole) at EOT and receives additional antibiotics (except aztreonam and metronidazole) at TOC for treatment of primary ABSSSI.

#### 3.3 Safety Variables

Safety endpoints are AEs, serious adverse events (SAEs), electrocardiogram (ECG) results, liver function tests, hematology, coagulation, serum chemistry including creatinine and creatinine clearance, urinalysis (UA), vital signs, and physical examinations.

#### 4 PHARMACOKINETIC/PHARMACODYNAMIC VARIABLES

Pharmacokinetic samples will be obtained from patients on 3 occasions: following the first dose of study medication, at ETP, and at EOT.

Iclaprim plasma concentrations will be used to determine population PK parameters with a non-linear mixed effect model. The potential influence of clinical characteristics (age, size, sex, hepatic function, renal function, concomitant medications, etc.) on PK parameters will be evaluated. Further details will be provided in a separate population PK analysis plan.

#### 5 ANALYSIS POPULATIONS

The ITT population will be the primary population for analysis of primary endpoint. Microbiological response will be evaluated for mITT, mCE and mPP populations. All other efficacy analyses will be performed for each of the ITT, mITT, PP, mCE and mPP populations. All safety analysis will be performed in the Safety population. Enrolled patients are those who signed the inform consent form.

#### 5.1 Safety Population

All patients who receive any study drug during the trial will be included in the Safety population. It is the primary population for safety analyses. Patients will be analyzed according to the treatment they receive.

#### 5.2 Intent-to-treat (ITT) population

All randomized patients will be included in the ITT population. It is the primary population for efficacy analyses. Patients will be analyzed in the treatment group to which they are randomized.

## 5.3 Microbiological intent-to-treat (mITT) population

All randomized patients who have a Gram-positive baseline bacteria pathogen identified as the cause of ABSSSI will be included in mITT population.

Covance Study ID: 000000145416

#### Statistical Analysis Plan

Version: Final Amendment 2.0 Motif BioSciences Protocol No. ICL-24-ABSSSI2

A Gram-positive bacteria pathogen is identified as the cause of ABSSSI if the Gram-positive pathogen is identified from the lesion sample, and is subsequently confirmed by Covance Central Laboratory Services

(CCLS).

#### 5.4 Per Protocol (PP) Population

The PP population will consist of all patients in the ITT population who receive at least 80% of their planned doses and provide adequate data for assessment for each of the following time points: ETP, EOT, and TOC. This population excludes patients with Gram-negative bloodstream infections at baseline who are discontinued in order to treat the Gram-negative pathogen.

The data are considered adequate for inclusion in the PP population when the assessment of lesion size and clinical signs and symptoms are both performed at corresponding time point. To be included in the PP population, a patient must not have important protocol deviations.

#### 5.4.1 Important Protocol Deviations Leading to Exclusion from the PP Analysis

Only those important protocol deviations considered to have a major effect on efficacy will lead to complete exclusion of the patient from the PP population. For the purposes of this study, the following criteria (Table 1) have been identified as important protocol deviations leading to exclusion from the PP population as it is considered that the occurrences of any of these criteria might have an important influence on the primary efficacy endpoint.

The majority of the important protocol deviations leading to exclusion from the PP population will be determined programmatically from the data. Those criteria which require clinical or medical monitoring interpretation will be reviewed prior to database lock, following discussion with the medical monitor and Sponsor.

Covance Study ID: 000000145416

#### Statistical Analysis Plan


Table 1: Important Protocol Deviations Leading to Exclusion from the PP population

| Type | Important Protocol Deviations Leading to Exclusion from the PP population | Method of Identification |
|---|---|---|
| Discontinuation of study drug | Patients with Gram-negative bloodstream infections who are discontinued in order to treat the Gram-negative pathogen. | Programmatic check on blood culture results and patient disposition status. Manual review will be performed for identifying patients who discontinue the study drug. |
| Noncompliance | Received less than 80% of the planned study drug. | Programmatic check based on the exposure and drug accountability data. Manual review will be performed for identifying patients who miss the study drug. |
| Errors in<br>Treatment<br>Allocation | Patients that receive a wrong treatment at 1 or more study visits due to packaging or dispensing errors | Programmatic check based on unblinded IXRS database after the study is unblinded. The check will be done by comparing the package number that IXRS had assigned to the patient against the package number actually used. |
| Clinical Trial<br>Management<br>System (CTMS) | Covance Clinical will provide the list of protocol deviations based on the clinical monitoring | Manual review: This list will be reviewed and the important protocol deviations that will lead to exclusion from the PP population will be identified. |
| Туре | Important Protocol Deviations<br>Leading to Exclusion at Affected<br>Visits | Method of Identification |
| Missing the required clinical evaluation | No adequate data at ETP, EOT and TOC | <b>Programmatic</b> check the missing assessment of lesion size, and the signs and symptoms at time points ETP, EOT and TOC |
| Prohibited medications | Systemic antibiotics (other than aztreonam and metronidazole) or topical antibiotics at the site of the ABSSSI under investigation, and steroids >20 mg/day prednisolone or equivalent (See Appendix A). | Manual review: List of preceding and concomitant medications will be reviewed by the study physician for potential prohibited medications occurring during the study up to and including TOC. |

All important protocol deviations leading to exclusion from the PP population occurring during the study will be reviewed and approved by the Sponsor prior to database lock and unblinding. Should additional important protocol deviations leading to exclusion from the PP population, not anticipated at the time of preparing this SAP, be identified during the study (and prior to unblinding), they will be documented in a SAP amendment and included in all relevant protocol deviation reviews and approvals.

If a patient is one or more visits, the rule to determine if they are included in Per-protocol population for different time-point is summarized in the table below. For overall analysis, such as demographic summary, patients are included in the overall Per-protocol population if they are included in PP analysis at any visit.

#### Statistical Analysis Plan


Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

| ETP visit | EOT visit | TOC visit | Per-protocol Assessment |
|---|---|---|---|
| Missing | | | Patient is excluded from all visits even if EOT or TOC are not missing because lesion size difference from ETP cannot be determined. |
| Not missing | Missing Missing | | Evaluable at ETP only. |
| Not missing | Missing Not missing Evaluable at | | Evaluable at ETP and TOC, excluded from EOT. |
| Not missing | Not missing | Missing | Evaluable at ETP and EOT, excluded from TOC. |
| Missing | Missing | Missing | Non-evaluable at all visits |

When analyzing efficacy endpoints, the following two rules will be applied to determine the clinical outcome for Per-protocol analysis:

- 1. If a rescue antibiotic is taken at a visit for clinical failure in ITT analysis, then the patient is still included for Per-protocol analysis at that timepoint and the outcome of failure is carried forward to subsequent visits and the patient is included at each of those visits for PP population.
- 2 If antibiotic is taken for a cause other than the index infection before assessed visits, the clinical outcome for this patient is Indeterminate for ITT population; however, this patient is excluded from PP population at that visit and subsequent visits.

#### 5.5 Modified clinically evaluable (mCE) population

The mCE population will consist of all patients excluded from the PP population only because they have received prohibited concomitant or preceding antibiotics therapy active against Gram-positive pathogens.

#### 5.6 PP microbiological evaluable (mPP) population

All mITT patients who receive at least 80% of their planned doses and provide adequate data for assessment for each of the following time points: ETP, EOT, and TOC.

#### 5.7 S. pyogenes-enriched mITT (S. pyogenes mITT) population

S. pyogenes mITT include all mITT patients and patients who have infection site culture negative and ASO titer positive for S. pyogenes at baseline or TOC.

#### 5.8 PP population for EMA sensitivity analysis

All PP patients without excluding any results at visits because of missing results at ETP.

#### 6 DATA HANDLING

#### 6.1 Time Points and Visit Windows

All analyses will use the nominal study visit as defined in the Study Schedule and eCRF. The study visit designations throughout tables and listings are listed as Baseline, Visit 2 (0-24 HRS), VISIT 2 (25-48 HRS), VISIT 2 (49-72 HRS), ETP, EOT, TOC, every 48 to 72 hours until EOT for Visit 4 and LFU. For microbiology data, baseline is defined within  $\pm 24$  hours for first study treatment.

Covance Study ID: 000000145416

#### Statistical Analysis Plan


| Study Visit in Protocol | Visit designations in tables and listings |
|---|---|
| Baseline/Screening/Visit 1 or Visit 2 (0-24 HRS) | Baseline |
| Visit 1 | Visit 1 |
| Daily until ETP for Visit 2 | Visit 2.1, Visit 2.2 and Visit 2.3 |
| ETP for Visit 3 | ETP |
| Every 48 to 72 hours until EOT for Visit 4 | Visit 4.1, Visit 4.2, Visit 4.3 and Visit 4.4 |
| EOT for Visit 5 | EOT |
| TOC for Visit 6 | TOC |
| LFU phone call | LFU |

### 6.2 Handling of Dropouts or Missing Data

For all ITT and mITT efficacy analyses, including the analysis of the primary endpoint, patients who do not have an adequate assessment at the appropriate visit will be assumed to be non-responders.

The safety evaluations will be performed on observed data only. Missing data will not be imputed for safety analyses except following rules to determine onset or stop dates of AEs or concomitant medications (see Section 1.4 in Appendix C – Table, Figure and Listing Shells for more details).

The imputed dates will not be listed. Study day relative to the first dose of treatment associated with missing or partial dates will not be displayed in AE listings.

The imputed dates of a medication will only be used to determine whether that medication will be classified as prior medication or concomitant medication.

#### 7 STATISTICAL METHODS

#### 7.1 General Principles

All data processing, summarization and analyses will be performed using Hosted SAS Environment / Version 9.3 (or later) of the SAS® (SAS Institute, Cary, NC) statistical software package.

Unless specified otherwise, data will be displayed using the following treatment group labels, in the order presented:

- Iclaprim
- Vancomycin
- Total (if applicable)

All data collected will be presented in listings by treatment group, country, center, patient, and visit (where applicable), unless otherwise specified.

Data will be presented in summary tables by treatment group, assessment and visit (where applicable). The category "Missing" will be presented if the number missing is greater than zero for at least one treatment group.

Descriptive summary statistics for continuous variables will include the number of observations (N), mean, standard deviation (SD), median and range.

Covance Study ID: 000000145416

#### Statistical Analysis Plan


Descriptive summary statistics for categorical variables will include frequency counts and percentages. Unless stated otherwise in the table shells, the denominator for percentage calculations will be the number of patients in the analysis population.

Dates will be displayed as DDMMMYYYY.

All significance tests will use a significance level of 5% for two-sided tests and a significance level of 2.5% for one-sided tests.

#### 7.2 Patient Disposition and Data Sets Analyzed

Patient disposition will be listed and summarized by treatment group and overall, and will include the number and percentage of patients:

- enrolled:
- randomized (ITT population);
- treated (Safety populations);
- other study populations (mITT, PP, mCE, mPP, S. pyogenes mITT, safety).

In addition, the number and percentage of patients who complete the study, who discontinue from study early, including a breakdown of the primary reasons for discontinuation, will be presented for ITT and Safety populations. The number and percentage of patients who complete the treatment will be analyzed in a similar manner.

A summary of patient enrollment by country and center will also be provided by treatment group and overall for the ITT population.

The number of patients who complete study or complete each visit of ETP, TOC and TOC will be analyzed by treatment groups and study populations.

#### 7.3 Protocol Deviations

All important protocol deviations leading to exclusion from the PP population (see Section 5.4.1) will be listed and summarized by treatment group for the ITT and mITT populations.

The deviations will be identified before data are unblinded.

## 7.4 Demographics and Other Baseline Characteristics

Demographic and baseline characteristics will be listed and summarized by treatment group and overall for ITT, mITT, PP, mCE, mPP and safety populations. Standard descriptive statistics will be presented for the continuous variables of:

- age (years obtained from IXRS)
- weight (kg);
- height (cm);
- body mass index (BMI; kg/m²) calculated as (weight/height²) where weight is in kilograms and height is in meters;
- lesion size (cm<sup>2</sup>)

The total counts and percentages of patients will be presented for the categorical variables of:

- age group (grouped as 18-39 years, 40-64 years, and 65 years and older);
- sex;
- race;
- ethnicity;

#### **Statistical Analysis Plan**

Motif RioSciences Protocol No. ICL -24-ABSSSI2

Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

- creatinine clearance (CrCL) in mL/min (grouped as ≥ 90, 60-89, 30-59, 15-29, and < 15 or hemodialysis);
- lesion type (major cutaneous abscess, cellulitis/erysipelas, and wound infection);
- Receipt of prior antibiotics (obtained from IXRS as Yes, No);
- Blood culture at baseline (positive, if anaerobic or aerobic blood culture has pathogen; negative, if culture taken and organism isolated but there is no pathogen or no organism was isolated)
- Gram-positive pathogen in infection site (multiple ABSSSI Gram-positive pathogen only, single Gram-positive pathogen only, single or multiple ABSSSI Gram-positive pathogens and Gram-negative pathogens);
- Methicillin-resistant *Staphylococcus aureus* (MRSA) vs Methicillin-sensitive *Staphylococcus aureus* (MSSA);
- Infection site pathogen (multiple pathogens vs single pathogen);
- Streptococcus pyogenes determined from ASO and either blood or infection site culture results from baseline (ASO positive only (> 330 IU/mL), culture positive only, ASO positive and culture positive, ASO negative (<= 330 IU/mL) and culture negative).
- severe infection (met the criteria of SIRS, has severe tenderness or severe erythema, has positive blood culture at baseline), defined in Section 2.1
- diabetes (yes if patient have medical history for diabetes, or baseline glucose > 200 mg/dL, or concomitant medications of either insulin or oral hypoglycemic; or no no medical history for diabetes, baseline glucose <= 200 mg/dL, no concomitant medications of either insulin or oral hypoglycemic.)
- geographic region (US, Europe, Latin America).

Other baseline measurements, such as type of culture specimen / culture result, lesion type, blood culture by visit, baseline pathogens, vital signs, ECG, and laboratory evaluations, will be summarized by treatment group with the post-baseline measurements.

#### 7.5 Medical History

Medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 18.1 (or a later version if updated during the study). All medical history will be listed, and the number and percentage of patients with any medical history will be summarized for ITT population by system organ class (SOC) and preferred term (PT) for each treatment group and overall.

#### 7.6 Prior and Concomitant Medications

Medications received prior to or concomitantly with treatment will be coded by Covance using the WHO Drug Dictionary, Version WHODRUG Enhanced 201509, DDEB2 (or a later version if updated during the study), Anatomical Therapeutic Chemical (ATC) Classification codes.

Prior medications are those taken prior to the first dose date of treatment and within the preceding 30 days of the Informed Consent.

Concomitant medications are those with a start date on or after the first dose date of treatment, or those with a start date before the first dose date of treatment and a stop date on or after the first dose date of treatment, or with a start date before the first dose date of treatment and are reported as ongoing.

If a medication cannot be classified as "prior" or "concomitant" after applying imputation rules for missing/incomplete dates, it will be classified as concomitant.

Covance Study ID: 000000145416

#### Statistical Analysis Plan


The number and percentage of patients using each medication will be displayed together with the number and percentage of patients using at least one medication within each therapeutic class (ATC-Level 2), chemical subgroup (ATC-Level 4), and generic term.

Separate summaries will be presented for prior medications, concomitant medication excluding antibiotics, and concomitant antibiotic medications for ITT population. A patient listing of all prior and concomitant medications will be provided for ITT population.

#### 7.7 Significant Procedures

The number and percentage of patients receiving any significant procedures, such as debridement or incision and drainage will be displayed by study visits and treatment groups for ITT population.

#### 7.8 Measurements of Treatment Compliance and Exposure

Percentage compliance is calculated as:

100 \* actual number of doses received / planned number of doses.

For example, patients are administered iclaprim q12h for 5 to 14 days, so the planned number of doses is 2 times the number of days in treatment period if the treatment is started in the AM. If a patient was treated for < 5 days, the planned number of dosing days will be considered as 5 days. If a patient was treated for > 5 days, the planned number of dosing days is the actual number of days dosed. Missed doses will not be included in the actual number of doses for the compliance calculation.

The number and percentage of compliant patients will be presented for the Safety population, where compliant is defined as percentage compliance greater  $\geq 80.0\%$ . The category of percentage compliance < 80.0% will also be presented. The treatment compliance will be tabulated with three categories with number and percentage of patients: < 80%, 80% to 100%, >100%.

The total treatment duration is defined as: Date of last dose – Date of first dose + 1 if treatment is started in the AM and completed in the PM. Treatment duration (days) will be summarized using descriptive statistics (n, mean, SD, median, minimum, and maximum) by treatment group for the Safety population.

#### 7.9 Efficacy

#### 7.9.1 Primary Efficacy Analysis

The primary efficacy analysis will be the NI (at significance level 0.025) of iclaprim (group 1) to vancomycin (group 2) for the proportion of ITT patients with a  $\geq$ 20% reduction in lesion size at ETP compared to baseline. The NI bound will be 10%. Let P1 be the proportion for iclaprim and P2 be the proportion for vancomycin. Equivalently, if the lower bound of the two-sided 95% confidence interval (CI) for P1 – P2 is greater than -0.100 based on the Z test with unpooled variance estimate, NI will be concluded.

#### 7.9.2 Secondary Efficacy Analysis

The primary NI efficacy analysis will be repeated in the mITT, mCE, PP, mPP populations, *S. pyogenes* enriched mITT population and PP population for EMA.

The secondary endpoints are resolution or near resolution of ABSSSI (i.e., clinical cure) at TOC for iclaprim compared with vancomycin, resolution or near resolution ( $\geq$ 90%) of ABSSSI at EOT, resolution or near resolution ( $\geq$ 90%) of ABSSSI at EOT and TOC among patients with severe infection at baseline,

Covance Study ID: 000000145416

#### **Statistical Analysis Plan**


time to resolution of signs and symptoms of ABSSSI, by-patient bacteriological response rate at EOT and

# TOC, and by-pathogen bacteriological response rate at EOT and TOC.

#### 7.9.2.1 Resolution or Near Resolution of ABSSSI

For resolution or near resolution of ABSSSI at TOC, the NI test described in Section 7.9.1 will be used to demonstrate the non-inferiority of iclaprim to vancomycin in the ITT population EMA primary endpoint. The same NI test will be repeated for mITT, mCE, PP, mPP and *S. pyogenes* enriched mITT population at TOC. All above tests will then be repeated for resolution or near resolution of ABSSSI at EOT. Additionally, the number and percentage of patients in each cure criteria will be displayed.

The NI test will be performed for resolution or near resolution of ABSSSI at TOC as well as EOT among patients with severe infection at baseline in ITT population, and repeated for mITT, PP populations.

A summary of clinical outcome, including the number and percent of patients with cure, failure and indeterminate outcomes at EOT and at TOC will be produced for the ITT, mITT, PP, and mPP.

### 7.9.2.2 Signs and Symptoms of ABSSSI

Baseline signs (tender to palpitations, erythema, edema, purulent drainage/discharge, fluctuance, induration, ulceration, and necrotic tissue) and baseline symptoms (localized pain, swelling, chills, and fever) will be summarized by intensity (none, mild, moderate and severe) using descriptive statistics.

Time (in days) to resolution of each of the signs and symptoms of ABSSSI is defined as: first date with no specified sign/symptom of ABSSSI recorded on eCRF post treatment – date of first dose + 1. For patients who are not free of the specified sign/symptom until the end of study, the last day recorded available sign/symptom on eCRF will be used as the censoring day. For patients free of any specific signs or symptoms at baseline (i.e. "none" of results for sign/symptom), please exclude these patients when analyzing time to resolution of that specific sign or symptom.

For each of the signs and symptoms, the hazard ratio of iclaprim vs vancomycin will be estimated in a Cox proportional hazard model for time to resolution of the specified sign/symptom, with the treatment group as the only covariate. The Kaplan-Meier (KM) method will be applied to estimate the distribution of the resolution time of each signs or symptom for each treatment group. The 95% CI of the hazard ratio will also be reported. This Cox regression will be performed in the ITT, mITT, PP populations.

#### 7.9.2.3 Bacteriological response

Bacteriological response will be assessed at the patient level and at the microbiological level on the basis of results of the cultures, the susceptibilities of identified organisms, and the clinical outcome of the patient for the mITT, mCE and mPP populations.

For each assessment (ETP, EOT, and TOC), the by-pathogen bacteriological response for each causative organism identified at baseline will be defined as follows:

- Eradication: baseline causative organism cannot be isolated from any culture(s) at the assessment.
- Presumed eradication: The patient is a clinical cure at the assessment, and there is no appropriate material for culture from the original site of infection.
- Persistence: The baseline causative pathogen (based on susceptibility profile or molecular typing) is isolated at the assessment.
- Presumed persistence: The patient is a clinical failure at the assessment, and no appropriate material is available for culture from the original site of ABSSSI.
- Indeterminate: Clinical response was Indeterminate at the assessment and no appropriate material is available for culture from the original site of ABSSSI.

#### **Statistical Analysis Plan**

Motif BioSciences Protocol No. ICL -24-ABSSSI2

Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

• Superinfection: A pathogen is isolated at the assessment that is different from the baseline causative pathogen.

• Recurrent infection: A pathogen is isolated only after the EOT visit that is different from the baseline pathogen(s).

By-pathogen bacteriological response categories will be summarized in a frequency table for each causative baseline pathogen per treatment group.

The by-patient bacteriological response will be determined according to the following definitions:

- Eradication: All baseline Gram-positive causative organism(s) have a response of Eradication.
- Presumed eradication: All baseline Gram-positive causative organism(s) have a response of Presumed Eradication or a combination of responses of Eradication and Presumed Eradication.
- Persistence: All or some baseline Gram-positive causative organism(s) have a response of Persistence or a combination of responses of Persistence and Presumed Persistence.
- Presumed persistence: All or some baseline Gram-positive causative organism(s) have a response of Presumed Persistence.
- Indeterminate: All baseline causative organism(s) have a response of Indeterminate.
- Superinfection: Any patient classified as a clinical failure who has a pathogen isolated during therapy that is different from the baseline causative pathogen.
- Recurrent infection: Any patient classified as a clinical failure who has a pathogen isolated after the EOT visit only, that is different from the baseline pathogen(s).

The by-patient bacteriological response will be determined by ordering the pathogen outcome for the patient by medical importance: persistence, presumed persistence, superinfection, recurrent infection, presumed eradication, and eradication. Patient bacteriological outcome is determined by the pathogen outcome of higher importance. For the combined rate of eradication or presumed eradication, 95% CI will be calculated per treatment group and for the difference as specified for the primary endpoint analysis, and number and percentages for all underlying by-patient bacteriological response categories will be tabulated.

Minimum inhibitory concentrations (MIC) will be summarized using EUCAST and CSLI methods for vancomycin and iclaprim antibiotics for mITT population. The number and corresponding percentage for interpretation of the MIC result will be summarized for three categories: susceptible, Intermediate or resistance.

### 7.9.3 Exploratory Analysis

- Mortality rate within 28 days of first dose of treatment will be summarized overall and by treatment group for the ITT population.
- For early clinical response of ABSSSI, the NI test described for the primary endpoint analysis will be used to evaluate the proportion of ITT patients with a  $\geq$  50%,  $\geq$  75%, and  $\geq$  90% reduction in lesion size at ETP compared to baseline.
- For improvement of ABSSSI at EOT and TOC, the NI test described for the primary endpoint analysis will be used to evaluate the proportion of ITT patients with a ≥ 50% and ≥ 75% reduction in lesion size at EOT and TOC.

#### Statistical Analysis Plan


Totif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

### 7.9.3.1 Exploratory Analysis Excluding Lesion Size Criteria

The criteria for lesion size reduction will be excluded for the following exploratory analyses.

- 1. Resolution or near resolution of ABSSSI excluding both criteria for lesion size reduction (≥ 90% reduction in lesion size from baseline and no increase in lesion size since ETP) at TOC for ITT, mITT, mCE and PP populations.
- 2. Resolution or near resolution of ABSSSI excluding both criteria for lesion size reduction (≥ 90% reduction in lesion size from baseline and no increase in lesion size since ETP) at EOT for ITT populations.
- 3. Resolution or near resolution of ABSSSI excluding both criteria for lesion size reduction (≥ 90% reduction in lesion size from baseline and no increase in lesion size since ETP) at TOC among patients with severe infection at baseline for ITT and PP population.
- 4. Resolution or near resolution of ABSSSI excluding both criteria for lesion size reduction (≥ 90% reduction in lesion size from baseline and no increase in lesion size since ETP) at TOC by subgroups for ITT and PP population.
- 5. Resolution or near resolution of ABSSSI excluding the criteria for no increase in lesion size since ETP at TOC for ITT population.
- 6. Clinical outcome excluding both criteria for lesion size reduction (≥ 90% reduction in lesion size from baseline and no increase in lesion size since ETP) will be evaluated at EOT and TOC programmatically for ITT and PP populations and categorized as cure, failure or indeterminate as follows:
  - Cure: defined by no requirement for additional antibiotics for treatment of primary ABSSSI (except aztreonam and metronidazole) or unplanned significant surgical procedures (excluding procedures that reflect failure of antimicrobial therapy);
  - Failure: death related to the infection, persisting or recurrent infection, need for unplanned significant surgical procedure (i.e., procedures that reflect failure of antimicrobial therapy), administration of rescue antibiotic therapy for the index infection before or at assessed visits;
  - Indeterminate: data inadequate for assessment of efficacy (there are no post-baseline local or systemic signs and symptoms data available to make this assessment [e.g., patient lost to follow up] after < 2 days of treatment or < 4 doses and no EOT evaluation), withdrawal of consent, receipt of effective antibiotic therapy for a cause other than the index infection before assessed visits, or death not attributed to the index ABSSSI or complication of ABSSSI.

**Note**: If a patient starts an antibiotic for an infection other than the primary ABSSSI at EOT visit date, they will still be included as clinical cure or clinical failure. The same rule will be applied to the evaluation of clinical outcome at TOC visit.

- Persistent infection occurs if a patient receives additional antibiotics for treatment of primary ABSSSI (except aztreonam and metronidazole) at EOT compared to baseline. The same rule applies when evaluating clinical failure at TOC visit.
- Recurrent infection occurs if a patient does not receive additional antibiotics (except aztreonam and metronidazole) at EOT and receives additional antibiotics (except aztreonam and metronidazole) at TOC for treatment of primary ABSSSI.

#### **Statistical Analysis Plan**

Motif BioSciences Protocol No. ICL -24-ABSSSI2

Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

- 7. Pathogen-level bacteriological response rate at TOC for mITT and mPP populations, where presumed eradication and presumed persistence will be defined without the lesion size criteria for the clinical cure and clinical failure.
- 8. Patient-level bacteriological response rate at EOT for mITT and mCE populations and TOC for mITT and mPP populations, where superinfection and recurrent infection will be defined without the lesion size criteria for clinical failure.
- 9. Patient-level combined bacteriological response rate at EOT for mCE population and TOC for mITT and mPP populations.
- If it is concluded that Iclaprim is non-inferior to Vancomycin (i.e., the lower bound of two-sided 95% confidence interval of group difference in early clinical response is greater than -0.1), it may be concluded that Iclaprim is superior to Vancomycin if the entire 95% confidence interval is >0. Superiority may also be concluded for resolution of ABSSSI at TOC in a similar manner.

#### 7.9.4 Subgroup Analysis

The primary endpoint, the proportion of patients with a  $\geq$ 20% reduction in lesion size at ETP compared to baseline and the key secondary endpoint, proportion of patients with a clinical cure at TOC, will be presented for ITT and PP populations.

- age group (grouped as 18-39 years, 40-64 years, and 65 years and older);
- sex;
- race (white vs non-white);
- creatinine clearance (CrCL) in mL/min (grouped as ≥ 90, 60-89, 30-59, 15-29, and < 15 or hemodialysis);
- blood culture at baseline (positive, if anaerobic or aerobic blood culture has pathogen; negative, if culture taken and organism isolated but there is no pathogen or no organism was isolated)
- MRSA vs MSSA;
- multiple pathogens vs single pathogen;
- Streptococcus pyogenes determined from ASO and either blood or infection site culture results from baseline (ASO positive only, culture positive only, ASO positive and culture positive, ASO negative and culture negative).
- diabetes (yes if patient have medical history for diabetes, or baseline glucose > 200 mg/dL, or concomitant medications of either insulin or oral hypoglycemic; or no no medical history for diabetes, baseline glucose ≤ 200 mg/dL, no concomitant medications of either insulin or oral hypoglycemic.)
- severe infection (met the criteria of SIRS, has severe tenderness or severe erythema, has positive blood culture at baseline), defined in Section 2.1;
- geographic region (US, Europe and Latin America).

The difference in the proportions of the two treatment groups and 95% CI will be calculated for each subgroup, and forest plots will be used to display these intervals graphically.


Motif BioSciences Protocol No. ICL-24-ABSSSI2

Date of Issue: 24 July 2017

Covance Study ID: 000000145416

#### **7.10** Safety

#### 7.10.1 Adverse Events

All adverse events (AEs) recorded on the eCRF will be coded using the MedDRA dictionary Version 18.1 (or a later version if updated during the study) and classified as either pre-treatment AEs or treatment – emergent AEs (TEAEs) as follows:

- Pre-treatment AEs are events that start prior to the date of first dose of treatment.
- TEAEs are events with start date on or after the date of first dose of treatment (using dates and times as recorded on the medication administration log) through TOC visit, or events with start date prior to the date of first dose of treatment whose severity worsens on or after the date of first dose of treatment. SAEs will be reported through end of study as TEAE.

If any incomplete date/time of AE onset or start of first infusion is not sufficient to exclude that the AE is treatment emergent, then the AE will be considered to be a TEAE.

All AE data will be listed by treatment group with Pre-treatment AEs and TEAEs presented separately. Treatment-emergent status will be flagged in the listing. In addition, corresponding listings of SAEs, AEs leading to discontinuation of treatment and AEs resulting in death will be produced.

The severity of all AEs is recorded as mild, moderate, or severe. If severity is missing for a TEAE, it will be considered severe only in the overall category in the summary tables.

The relationship between an AE and treatment is assessed as related, probably related, probably not related, or not related. A drug-related AE is an AE considered by the investigator as related or probably related to the study drugs, or with unknown/missing relationship to treatment.

Each AE must be assessed and recorded in the eCRF as serious or not serious. Serious AEs must be reported as described in the protocol

An overview table will summarize the number and percentage of patients with at least one of the following TEAEs for Safety population, where patients with more than one TEAE in a particular category are counted only once in that category:

- any TEAE;
- any TEAE by severity (mild, moderate, severe);
- drug-related TEAEs;
- TEAEs leading to discontinuation of the study drug;
- SAEs;
- drug-related SAEs;
- SAEs leading to death.

The number and percentage of patients reporting each TEAE, including TEAE by age (< 65 and  $\geq$  65), TEAEs by CrCL ( $\geq$  90, 60-89, 30-59, 15, 29, and < 15 or hemodialysis), TEAEs by diabetes (present or absent), TEAEs leading to discontinuation, SAEs, drug related SAEs, and SAEs leading to death, will be summarized for each treatment group and overall, by SOC (sorted alphabetically) and PT (sorted by descending overall total) for Safety population. The analogous summaries will also be given for study drug related TEAEs, all TEAEs by severity and for all SAEs. TEAEs with missing severity will not be included in the counts of patients within a SOC or PT. For counting the number of events, the same rule for multiple events in one category will be applied as specified above. There will also be summaries of the

#### Statistical Analysis Plan

Motif BioSciences Protocol No. ICL -24-ABSSSI2

Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

most common TEAEs (> 5%) and SAEs (> 5%, > 1%) by PT in descending order of frequency in the iclaprim group.

No statistical comparisons of AEs, deaths, AE leading to discontinuation, or SAEs between treatment groups will be performed.

#### 7.10.2 Laboratory Evaluations

Data for the following hematology, blood chemistry, and urinalysis analytes received from central laboratory as well as LFT results (Table 2) recorded in the eCRF will be listed (see Appendix B for the scheduled data collection) and summarized by treatment group and visit. Data received from local laboratories will be listed with the original units. If data for any additional analytes are also received then these will be listed only.

All central laboratory data will be reported in International System of Units (SI Units) and Conventional Units (CV Units). Out-of-reference-range values will be flagged as high (H) or low (L) in the data listings.

**Table 2: Laboratory Evaluations** 

| Table 2. Laboratory Evaluations | | |
|---|---|---|
| Hematology (CBC) | Chemistry [Fasted] (Chem-20) | Urinalysis (UA) |
| Hematocrit | Albumin | pH and specific gravity |
| Hemoglobin | ALP | Glucose |
| MCH | ALT | Ketones |
| MCHC | AST | Occult blood |
| MCV | BUN | Proteins |
| Platelet count | Chloride | Microscopic examination |
| Red Blood Cell Count | Creatinine | of sediment (including |
| White Blood Cell Count | GGT | RBCs and WBCs) |
| White Blood Cell Differential | Glucose | Bilirubin/Urobilinogen |
| (% & ABS): | LDH | |
| Basophils | Potassium | |
| Eosinophils | Sodium | |
| Lymphocytes | Magnesium | |
| Monocytes | Total Bilirubin | |
| Neutrophils | Total CO <sub>2</sub> (measured as bicarbonate) | |
| | Total protein | |
| | CPK | |
| | CRP | |
| Source: Protocol Appendix A – Cl | inical Laboratory Evaluations | |

Laboratory test variables will be summarized by treatment group and visit using descriptive statistics (number of patients, mean, SD, minimum, maximum, as well as mean change from baseline, standard error for mean change, minimum, median, and maximum). For each laboratory analyte, the baseline value will be defined as last scheduled or unscheduled value collected prior to the first dose of treatment. The descriptive statistics will be summarized for both SI and CV units.

#### **Statistical Analysis Plan**

Motif BioSciences Protocol No. ICL -24-ABSSSI2

Motif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

The number and percentage of patients with values below, within and above the corresponding extended normal range will be tabulated per visit. Shift tables (i.e., cross-tabulations of below the lower limit of the normal range, within the limits of the normal range and above the upper limit of the normal range at baseline versus scheduled visits) will be presented by laboratory test.

In addition, shift tables for 6 liver enzyme tests (AST, ALT, alkaline phosphatase, GGT, total and direct bilirubin) and 3 renal function tests (BUN, creatinine, creatinine clearance) for post-baseline change in grade categories  $\leq$  ULN,  $\leq$  3x ULN, > 3x-5x ULN, > 5x-10x ULN, > 10x-20x ULN, > 20x ULN will be presented. For bilirubin, the category is presented as two categories, < 2x ULN, > 2x ULN. The maximum change through all study will be presented as overall results and results will also be presented by visit.

Urinalysis tests with categorical results will be summarized by frequency patients n each category. All laboratory data, including data obtained from laboratory tests not required by the protocol will not be summarized, but will be listed.

#### 7.10.3 Vital Signs

The following vital signs will be listed and summarized by treatment group and visit (see Appendix B for the scheduled data collection).

- systolic and diastolic blood pressure (mmHg);
- heart rate (bpm);
- respiration rate (breaths/min);
- body temperature (°C).

Vital signs data and changes from baseline in vital signs will be summarized by visit using standard descriptive statistics for the Safety population. The baseline value will be defined as last scheduled or unscheduled value collected prior to the first dose of treatment. Assessments carried out on day of first treatment administration are considered to have taken place before the treatment administration, if the corresponding times have not been recorded. For post-baseline, only data from scheduled visits will be included in the summary tables.

#### 7.10.4 Electrocardiograms

The following quantitative ECG measurements will be taken and read centrally during the study (see Appendix B for the scheduled data collection):

- heart rate (bpm);
- RR interval (msec);
- PR interval (msec);
- QRS interval (msec);
- QT interval (msec);
- Bazett corrected QT (QTcB) interval (msec);
- Fridericia corrected QT (QTcF) interval (msec).

Triplicate ECG measurements will be listed for every ECG measurement, and the median value of the triplicate measurements will be summarized using descriptive statistics.

Based on 12-lead triplicate ECG results as reported on the case report form (CRF) that are read centrally the number and percentage of patients whose median QTcF value is > 500 msec and/or is >60 msec

#### Statistical Analysis Plan


otif BioSciences Protocol No. ICL-24-ABSSSI2 Covance Study ID: 000000145416

different from the predose baseline value will be provided for every visit. For every visit with ECG measured, the median QTcF and QTcB values will be summarized with descriptive statistics for the following categories:

- > 450 msec;
- > 480 msec;
- > 500 msec;
- increase from baseline > 30 msec;
- increase from baseline > 60 msec.

The central ECG measurements at all pre-planned visits and time points and changes from baseline in ECG will be listed and summarized by treatment group and visit using standard descriptive statistics for the Safety population.

The baseline value will be defined as last scheduled or unscheduled median value collected prior to the first dose of treatment. Assessments carried out on day of first treatment administration are considered to have taken place before the treatment administration, if the corresponding times have not been recorded. For post-baseline, only data from scheduled visits will be included in the summary tables.

#### 7.10.5 Physical Examination

Physical examination results (normal/abnormal) and details of abnormalities will be listed for each patient (see Appendix B for the scheduled data collection).

#### 7.11 Interim Analysis

When 75% of the randomized patients have undergone the 48- to 72-hour (ETP) response assessment, a blinded interim analysis is planned to estimate the percentage of patients in the study who classify as having a reduction in the lesion size  $\geq$ 20% at the 48- to 72-hour visit compared to baseline. Based on the observed overall percentage, the sample size will be re-estimated as  $N_1$  using z-test with unpooled variance estimate. The new total sample size will be the maximum of 300 and  $N_1$ , following Friede T et al (2007). The sponsor may increase the total sample size to attempt to ensure that an adequate number of ITT patients are included in the study. Since the review is blinded and the efficacy analyses will not be reviewed by treatment group, no adjustment of p-values is required. Nevertheless, the sponsor will take steps to minimize the distribution of results to avoid introducing any bias.

#### **8 REFERENCES**

Friede T, Mitchell C, Müller-Velten R. *Blinded Sample Size Reestimation in Non-Inferiority Trials with Binary Endpoints*. Biometrical Journal. 2007; 49: 903-916.

Version: Final Amendment 2.0Date of Issue: 24 July 2017Motif BioSciences Protocol No. ICL-24-ABSSSI2Covance Study ID: 000000145416

#### 9 APPENDICES

#### **Appendix A – Prohibited Medicines**

The following medications are prohibited:

- Systemic antibiotics (other than aztreonam and metronidazole) or topical antibiotics at the site of the ABSSSI under investigation;
- Steroids >20 mg/day prednisolone or equivalent;
- Type IA and Type III anti-arrhythmic drugs; and
- Local antiseptics.


Covance Study ID: 000000145416

Date of Issue: 24 July 2017

#### Appendix B – Schedule of Events

| Procedure | Baseline/ | Daily until ETP | ETP | Every 48 to 72 | EOT/ | TOC | LFU |
|---|---|---|---|---|---|---|---|
| | Screening/ | Visit 2 | (48 to 72 | hours until | Early Termination | 7 to 14 days | 28 to 32 days |
| | Randomization | | hours post- | EOT | Visit 5 | post-EOT | post-first dose |
| | Visit 1 | | first dose) | Visit 4 | (treatment duration: | Visit 6 | Phone Call <sup>2</sup> |
| | (up to 24 hours | | Visit 3 | | minimum 5 days, maximum | | |
| | prior to first dose) <sup>1</sup> | | | | 14 days) | | |
| Informed consent | X | | | | | | |
| Medical history | X | | | | | | |
| Prior medications (preceding 30 days) | X | | | | | | |
| Concomitant medications | | X | X | X | X | X | |
| Review of inclusion & exclusion criteria | X | | | | | | |
| Complete physical examination <sup>3</sup> | X | | | | | | |
| Limited physical examination <sup>4</sup> | | X | X | X | X | X | |
| Assessment of signs & symptoms of ABSSSI with | X | | X | | X | X | |
| digital photography <sup>5</sup> | | 37 | | 37 | | | |
| Assessment of signs & symptoms of ABSSSI without digital photography <sup>5</sup> | | X | | X | | | |
| Evaluation of adverse events <sup>6</sup> | X | X | X | X | X | X | X |
| Significant procedures (incision & drainage, debridement, amputation, suture removal, etc.) | | X | X | X | X | X | |
| Creatinine clearance (estimated) | X | | | | | | |
| LFT safety | X | X | X | | X | X | |
| C-reactive protein | X | | X | | X | X | |
| Hematology <sup>7</sup> | X | | X | X | X | X | |
| Clinical chemistry <sup>7</sup> | X | | X | X | X | X | |
| Urinalysis <sup>7</sup> | X | | X | X | X | X | |
| Serum pregnancy test (females of childbearing potential) <sup>8</sup> | X | | | | | | |
| Blood cultures (aerobic/anaerobic) | $X^9$ | $X^{10}$ | X <sup>11</sup> | X <sup>11</sup> | | | |
| Study medication administration <sup>12</sup> | | X | X | $X^{13}$ | $X^{14}$ | | |
| Blood sample for PK analysis | | X <sup>15</sup> | $X^{16}$ | | $X^{16}$ | | |
| ECG (at each timepoint 3 ECGs at least 1 minute apart will be performed) | X | X <sup>17</sup> | $X^{18}$ | | | | |
| Infection site cultures <sup>19</sup> | X | | X | | X | X | |
| ASO antibody titers | X | | | | | X | |
| Draw trough levels <sup>20</sup> | | | | $X^{21}$ | | | |
| Central randomization | X | | | | | | |
| Clinical efficacy assessment | | | | | X | X | |
| Day 28 mortality | | | | | - | - | X |

Abbreviations: ASO = anti-streptolysin O; EOT = End of Therapy; ETP = Early Timepoint; LFT=liver function test; LFU = Late Follow-up; TOC = Test of Cure.

<sup>&</sup>lt;sup>1</sup> Must be performed during the baseline visit and completed within 24 hours of study entry (first dose of study drug).

<sup>&</sup>lt;sup>2</sup> Patients with high LFTs and unresolved AEs at TOC will be required to come in for an additional visit at LFU (for LFTs, blood samples will be obtained to document normalization). If duration of therapy

Motif BioSciences Protocol No. ICL-24-ABSSSI2

**Date of Issue: 24 July 2017** Covance Study ID: 000000145416

is 14 days, LFU may overlap with TOC. In this case, all LFU evaluations may take place at the TOC visit.

- <sup>3</sup> Complete physical examination, including vital signs (includes determination of body temperature), height, weight, and a review by body systems.
- <sup>4</sup> Limited physical examination, including vital signs (includes determination of body temperature) and excluding weight and height.
- <sup>5</sup> Eight signs (tenderness to palpitation, erythema, edema, purulent drainage/discharge, fluctuance, induration, ulceration, and necrotic tissue) and four symptoms (localized pain, swelling, chills, and fever) of infection will be assessed at each evaluation and graded on a scale of 0 to 3 (0=none, 1=mild, 2=moderate, or 3=severe). The extent of the infection (to include width, length, and depth and diagram of the infection site) will be determined via photography at baseline, ETP, EOT, and TOC only. Photography procedures outlined in protocol Appendix B will be followed. Acetate based planimetric tracing will follow the procedures outlined in Appendix C. (Planimetry measurements are based upon automatic detection of pixels inside of the traced skin infection area. Pixels are converted to calibrated units based on the scanned resolution [e.g., 300 DPI]. Skin infection measurements will be provided in cm<sup>2</sup>.). Patients who have a worsening of clinical signs and symptoms of ABSSSI during study medication treatment such that additional or alternative systemic antibacterial therapy is warranted must be withdrawn from study medication.
- <sup>6</sup> All adverse events will be recorded throughout the study period, up to and including the LFU phone call.
- <sup>7</sup> Hematology comprises a complete blood count (RBC count, WBC count with differential counts, platelet count, hemoglobin, and hematocrit), MCH, MCHC, MCV, and CRP. Clinical chemistry comprises creatinine, BUN, AST, ALT, alkaline phosphatase, total bilirubin, albumin, total protein, glucose, sodium, potassium, chloride, bicarbonate, LDH, GGT, and CPK. Urinalysis comprises determination of pH, specific gravity, presence of blood, glucose, protein, ketones, and bile, and microscopic examination of sediment.
- <sup>8</sup> Serum pregnancy test must be obtained immediately prior to randomization. If obtaining the serum pregnancy result would cause a delay in treatment, the patient can be entered on the basis of a negative urine pregnancy test result. The urine pregnancy test must be sensitive to at least 50 mU/mL of beta-hCG, pending results of the serum test. The patient must inform the investigator if she becomes pregnant, and study medication must be withdrawn.
- <sup>9</sup> Obtain two sets of blood cultures (aerobic and anaerobic) 10 minutes apart from two separate peripheral sites.
- <sup>10</sup> If patient has a blood culture that grows a Gram-negative pathogen from Visit 1 blood cultures, the patient must be withdrawn from study medication and started on the appropriate antibiotics for complicated bacteremia. If patient has signs of bacteremia, obtain two sets of aerobic/anaerobic blood cultures 10 minutes apart that are collected at different sites.
- <sup>11</sup> If patient has a blood culture that grows a Gram-negative pathogen from Visit 2 blood cultures, the patient must be withdrawn from study medication and started on the appropriate antibiotics for complicated bacteremia. If patient has a blood culture that grows a Gram-positive pathogen from Visit 1 and/or Visit 2 blood cultures, another 2 sets of blood cultures must be obtained at both Visit 3 and Visit 4. If these are positive, the patient must be withdrawn from study medication and started on the appropriate antibiotics for complicated bacteremia.
- 12 A window of +/- 2 hours is acceptable for infusion of study medication. For patients randomized to receive vancomycin, vancomycin dosing will be adjusted based on trough levels to maintain a trough of either 10 to 15 mg/L for patients with an organism whose MIC is ≤1 mg/L or 15 to 20 mg/L for patients with an organism whose MIC is >1 mg/L. Dose adjustments made due to trough monitoring will need to be performed in such a manner as to ensure that the blind is maintained.
- <sup>13</sup> If the last dose of study drug falls on a day when an evaluation was not planned, an additional evaluation visit will need to be performed on that day (i.e., all EOT evaluations should be performed on the last day [+2 days] of drug dose).
- <sup>14</sup> If clinically indicated (i.e., investigator may decide on a given day that a patient no longer needs treatment. In these cases, medication will not be administered, but all other EOT assessments must be performed.)
- 15 On Day 1, before the start of first study medication infusion and within 5 to 15 minutes, 1 to 3 hours, and 5 to 7 (ensure last PK sample is taken prior to next dose) hours after the infusion.
- 16 Before the start of study medication infusion at ETP and EOT, and within 5 to 15 minutes, 1 to 3 hours, and 5 to 7 hours (ensure last PK sample is taken prior to next dose) after the ETP and EOT infusions.
- <sup>17</sup> On Day 1, before the start of first study medication infusion and within 10 minutes of the end of the first study medication infusion. If the median QTcF value is >500 msec and/or is >60 msec different from the predose baseline value, follow-up ECG tests should be performed every 1 to 2 hours until they are below these threshold values.
- <sup>18</sup> At ETP, an ECG should be performed before the start of study medication infusion and within 10 minutes of the end of the study medication infusion.
- <sup>19</sup> Prior to randomization, all patients (regardless of the disease type) should have appropriate cultures obtained. Deep culture samples, such as from a biopsy, needle aspiration, surgically obtained specimens, or punch biopsies of an area contiguous to the infected wound should be obtained. Swabs are not acceptable; cultures will be performed locally, where isolates will be retained for transport to a central microbiology laboratory for susceptibility testing according to CLSI-approved methodology. Note that only target pathogens will be sent to the central microbiology laboratory (therefore, contaminants/Gram-negative isolates [from mixed wound infections] in blood cultures do not need to be sent). If the patient is discontinued from the study due to treatment failure, a clinical specimen will
- be obtained at that time only. Additional clinical specimens will be obtained, if clinically feasible and if the patient has persistent clinical signs or symptoms, at ETP, EOT, and TOC. <sup>20</sup> For vancomycin patients with a CrCL < 25mL/min, a daily level should be obtained and the unblinded team should monitor and re-dose the patient when that level is below 20 mg/L.
- <sup>21</sup> Vancomycin patients with a CrCL ≥25 mL/min should have their vancomycin level checked with the 5<sup>th</sup> dose due to difficulty interpreting levels checked prior to achieving steady state.


**Date of Issue: 24 July 2017** Covance Study ID: 000000145416 Motif BioSciences Protocol No. ICL-24-ABSSSI2

## Appendix C – Table, Figure and Listing Shells

The table, figure, and listing shells and corresponding Table of Contents will be created in a separate file.

# TABLES, FIGURES, AND LISTINGS SHELLS

A Phase 3, randomized, double-blind, multicenter study to evaluate the safety and efficacy of intravenous iclaprim versus vancomycin in the treatment of acute bacterial skin structure infections suspected or confirmed to be due to Gram-positive pathogens. (REVIVE-2)

TFL Status: Final 1.0 TFL Date: 2016-08-16T22:39:26

Study Drug: iclaprim

Sponsor Reference: Protocol ICL-24-ABSSSI2 Covance Study No: 000000145670

#### 1. INTRODUCTION

The table, figure, and listing (TFL) shells presented in this document are mock-ups and may be subject to minor format modifications once the actual data are used. The data represented in this document are used for example purposes only and do not reflect the actual study data captured. The overall contents in any individual TFL shell will not change, although additional tables may be added if necessary, thus changing the table number scheme. Significant changes will be approved by the responsible Covance Clinical Pharmacology project team member and communicated to the Sponsor.

## 1.1 General Programming Specifications

All TFLs will follow the following rules:

Papersize will be Letter, with the following margins in Inches:

#### Landscape

top 1.5 left 1 bottom 1.73 right 1

## **Portrait**

Top 1.5 left 1.5 Bottom 1.5 right 1.23
Every TFL will have a footnote containing program location, name, run date and run time (optional), the name of the last person who ran the program, and the status of the output:

Dry run – Draft – Final Draft – Final (others as needed)

Dates will be presented in the format ddMonyyyy

The presentation order of the statistics will be:

Mean, SD, median, minimum, maximum, N. The abbreviations Med, Min, Max may be used, if necessary.

Rules for significant digits in safety data tables are as follows: if the raw value has x decimal places, then the mean and the median will have x+1 decimal places, the standard deviation will have x+2 decimal places.

N will be presented as whole numbers.

Percentages will always be displayed with 1 decimal place. For percentages < 0.1%, <0.1% will be displayed.

### 1.2 Derived Parameters

Individual derived parameters and appropriate summary statistics will be reported to three significant figures.

# 1.3 Tables Summarizing Categorical Data

Tables that summarize categorical data will be created per these specifications:

- 1. If the number of events is zero, data will be presented as "0".
- 2. If the categories of a parameter are ordered, all categories between the maximum possible category and the minimum category will be included, even if n=0 for a given category.
- 3. If the categories are not ordered, only those categories for which there is at least one subject represented will be included.

4. A "missing" category will be included for any parameter for which information is missing. This will ensure that the population size totals are consistent across different parameters.

#### 1.4 Tables for Imputing Onset and Stop Dates of Adverse Events (AEs) and Concomitant Medications

The general principle for imputing dates is as follows:

If an adverse event start date is completely missing or partially missing, then it assumed that the start date occurs at the earliest time on-treatment whenever possible.

If a concomitant medication onset date is completely missing, then the date is not imputed. Otherwise, if the concomitant medication onset date is partially missing, then it is assumed that the start date occurs at the earliest time on-treatment whenever possible.

If a concomitant medication or adverse event stop date is completely missing or partially missing, then the stop date is imputed to maximize the duration of the event or concomitant treatment. It should be noted that imputation of stop dates only applies to concomitant medications that are not ongoing and adverse events that are not ongoing (ie outcome is not resolved).

| Sce | nario | |
|---|---|---|
| Onset date | Stop date | Imputation rule |
| Partially<br>Missing | Complete | Imputation of onset date: A. If partial date has day and month missing: |
| Wilssing | | If year of the partial date < year of the first dose date, assign December 31 <sup>st</sup> to the missing fields. If year of the partial date = year of the first dose date, assign the first dose date to the missing fields. |

| | | If year of the partial date > year of the first dose date, assign January 1 <sup>st</sup> to the missing fields. Note: if first dose date is missing, then use randomization date in the above imputations. B. If partial date has missing day only: If the month and year of the partial date < month and year of the first dose date, assign last day of the onset month to the missing day. If the month and year of the partial date = month and year of the first dose date, assign the day of first dose to the missing day. If the month and year of the partial date > month and year of the first dose date, assign first day of the onset month to the missing day. |
|---|---|---|
| | | If the imputed onset date (after A or B above) is after the stop date, the onset date will be imputed to be equal to the stop date. |
| Complete | Partially<br>Missing | Imputation of stop date (if not reported as ongoing): C. If partial date has day and month missing: If year of partial date < year of the last known alive date (LKAD), assign December 31st to the missing fields. If year of partial date = year of the LKAD, assign the LKAD date to the missing fields If year of partial date > year of the LKAD, the missing day and month will NOT be imputed. D. If partial date has missing day only: If the month and year of the partial data < the month and year of the LKAD, assign the last day of the onset month to the missing day. If the month and year of the partial date = the month and year of the LKAD, assign the LKAD to the missing day. If the month and year > the month and year of the LKAD, the missing day will NOT be imputed. LKAD is defined as the date of death or the last day recorded on the log form. |
| | | If the imputed stop date (after C or D above) is before the onset date, the stop date will be imputed to be equal to the onset date. |
| Partially<br>Missing | Partially<br>Missing | Impute onset date per A and B above Impute stop date (if not reported as ongoing) per C and D above If imputed onset date > imputed stop date, then set onset date = stop date = minimum of (imputed onset date per A and B, imputed stop date per C and D) |


| Partially<br>Missing | Completely<br>Missing | Impute onset date per A and B above. |
|---|---|---|
| | | Impute stop date (if not reported as ongoing) as the LKAD; see definition above. |
| | | If imputed onset date > imputed stop date, then set onset date = stop date = minimum of (imputed onset date per A and B, imputed stop date above) |
| Completely<br>Missing | Partially<br>Missing | Adverse Events Impute onset date as the first dose date; if first dose date is missing, then use randomization date |
| | | If imputed onset date > imputed stop date, then set onset date = stop date = minimum of (imputed onset date above, imputed stop date per C and D) |
| | | Concomitant Medications Do not impute onset date |
| | | Impute stop date (if not reported as ongoing) per C and D above |
| Completely<br>Missing | Complete | Adverse Events Impute onset date as the first dose date; if first dose date is missing, then use randomization date. |
| | | If imputed onset date > stop date, then set onset date = (complete) stop date |
| | | Concomitant Medications Do not impute onset date. |
| Complete | Completely<br>Missing | Impute stop date (if not reported as ongoing) as the LKAD; see definition above. |
| | wiissing | If onset date > imputed stop date, then set stop date = (complete) onset date |
| Completely | Completely | Adverse Events |

| Missing | Missing | Impute onset date as the first dose date; if first dose date is missing, then use randomization date. |
|---|---|---|
| | | Impute stop date (if not reported as ongoing) as the LKAD; see definition above. |
| | | Concomitant Medications Do not impute onset date. |
| | | Impute stop date (if not reported as ongoing) as the LKAD; see definition above. |

## 2. TABLE OF CONTENTS

| | Introduction - | |
|---|---|---|
| | Table of Contents - | |
| Table 14.1.1 | Overall Summary of Study Populations - Enrolled Patients | |
| Table 14.1.2.1 | Summary of Study Completion - ITT Population | |
| Table 14.1.2.2 | Summary of Study Completion - Safety Population | . 1' |
| Table 14.1.2.3 | Summary of Treatment Completion - ITT Population | |
| Table 14.1.2.4 | Summary of Treatment Completion - Safety Population | . 10 |
| Table 14.1.3 | Study Sample Sizes by Country and Center - Enrolled Patients | 20 |
| Table 14.1.4 | Number of Patients Assessed at Visits with Efficacy Assessment - All Randomized Patients | 2 |
| Table 14.1.5.1 | Summary of Major Protocol Violations/Deviations - ITT Population | 2 |
| Table 14.1.5.2 | Summary of Major Protocol Violations/Deviations - mITT Population | |
| Table 14.1.6 | Summary of Patients Validity - All Randomized Patients | |
| Table 14.1.7.1 | Summary of Demography - ITT Population | |
| Table 14.1.7.2 | Summary of Demography - mITT Population | |
| Table 14.1.7.3 | Summary of Demography - PP Population | |
| Table 14.1.7.4 | Summary of Demography - mPP Population | |
| Table 14.1.7.5 | Summary of Demography - mCE Population | |
| Table 14.1.7.6 | Summary of Demography - Safety Population | |
| Table 14.1.8.1 | Baseline Disease Characteristics - ITT Population | 25 |
| Table 14.1.8.2 | Baseline Disease Characteristics - mITT Population | |
| Table 14.1.8.3 | Baseline Disease Characteristics - PP Population | |
| Table 14.1.8.4 | Baseline Disease Characteristics - mPP Population | |
| Table 14.1.8.5 | Baseline Disease Characteristics - mCE Population | |
| Table 14.1.8.6 | Baseline Disease Characteristics - Safety Population | |
| Table 14.1.9 | Summary of Medical History - ITT Population | 30 |
| Table 14.1.10.1 | Prior Medications - ITT Population | |
| Table 14.1.10.2 | Concomitant Medication Excluding Antibiotics - ITT Population | |
| Table 14.1.10.3 | Concomitant Antibiotic Medication - ITT Population | |
| Table 14.1.10.4 | Summary of Significant Procedures by Visit - ITT Population | |
| Table 14.1.11.1.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Tender to Palpitation - ITT Population | |
| Table 14.1.11.1.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Tender to Palpitation - PP Population | |
| Table 14.1.11.1.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Tender to Palpitation - mCE Population | 3 |
| Table 14.1.11.2.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Erythema - ITT Population | 3 |
| Table 14.1.11.2.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Erythema - PP Population | |
| Table 14.1.11.2.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Erythema - mCE Population | |
| Table 14.1.11.3.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Edema - ITT Population | |

| Table 14.1.11.3.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Edema - PP Population | 36 |
|---|---|---|
| Table 14.1.11.3.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Edema - mCE Population | 36 |
| Table 14.1.11.4.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Purulent Drainage/Discharge - ITT Population | 36 |
| Table 14.1.11.4.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Purulent Drainage/Discharge - PP Population | 36 |
| Table 14.1.11.4.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Purulent Drainage/Discharge - mCE Population | 36 |
| Table 14.1.11.5.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Fluctuance - ITT Population | 36 |
| Table 14.1.11.5.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Fluctuance - PP Population | |
| Table 14.1.11.5.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Fluctuance - mCE Population | 36 |
| Table 14.1.11.6.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Induration - ITT Population | 36 |
| Table 14.1.11.6.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Induration - PP Population | 36 |
| Table 14.1.11.6.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Induration - mCE Population | 36 |
| Table 14.1.11.7.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Ulceration - ITT Population | 36 |
| Table 14.1.11.7.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Ulceration - PP Population | 36 |
| Table 14.1.11.7.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Ulceration - mCE Population | |
| Table 14.1.11.8.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Necrotic Tissue - ITT Population | |
| Table 14.1.11.8.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Necrotic Tissue - PP Population | |
| Table 14.1.11.8.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Necrotic Tissue - mCE Population | |
| Table 14.1.11.9.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Localized Pain - ITT Population | 36 |
| Table 14.1.11.9.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Localized Pain - PP Population | |
| Γable 14.1.11.9.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Localized Pain - mCE Population | |
| Γable 14.1.11.10.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Swelling - ITT Population | |
| Table 14.1.11.10.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Swelling - PP Population | |
| Table 14.1.11.10.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Swelling - mCE Population | 37 |
| Гable 14.1.11.11.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Chills - ITT Population | |
| Гable 14.1.11.11.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Chills - PP Population | |
| Γable 14.1.11.11.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Chills - mCE Population | |
| Γable 14.1.11.12.1 | Clinical Signs and Symptoms of ABSSSI by Visit: Fever - ITT Population | 37 |
| Table 14.1.11.12.2 | Clinical Signs and Symptoms of ABSSSI by Visit: Fever - PP Population | |
| Table 14.1.11.12.3 | Clinical Signs and Symptoms of ABSSSI by Visit: Fever - mCE Population | 37 |
| Table 14.1.12.1 | Type of Culture Specimen and Culture Results by Visit - ITT Population | |
| Table 14.1.12.2 | Summary of Culture Specimen for Lesion Type by Visit - ITT Population | 39 |
| Table 14.1.12.3 | Microbiological Assessment of Primary Infection Site - Gram Stain - ITT Population | 40 |
| Гable 14.1.12.4 | Blood Culture Results by Visit - ITT Population | 41 |
| Table 14.1.12.5 | Gram-positive Pathogens Occurring in Patients at Baseline - ITT Population | |
| Table 14.1.12.6 | Frequency Distribution of MIC by Baseline Pathogen - ITT Population | 43 |
| Table 14.1.13.1 | Summary of Treatment Compliance - ITT Population | 44 |
| Table 14.1.13.2 | Summary of Treatment Exposure: Duration in Days - Safety Population | |
| Гable 14.2.1 | Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - ITT Population | |
| Гable 14.2.2.1 | Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - mITT Population | 46 |
| Гable 14.2.2.2 | Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - mCE Population | |
| Table 14.2.2.3 | Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - PP Population | 47 |

| Table 14.2.2.4 | Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - mPP Population | 4 |
|---|---|---|
| Table 14.2.3.1 | Resolution or Near Resolution of ABSSSI at TOC - ITT Population | 48 |
| Table 14.2.3.2 | Resolution or Near Resolution of ABSSSI at TOC - mITT Population | |
| Table 14.2.3.3 | Resolution or Near Resolution of ABSSSI at TOC - mCE Population | 49 |
| Table 14.2.3.4 | Resolution or Near Resolution of ABSSSI at TOC - PP Population | |
| Table 14.2.3.5 | Resolution or Near Resolution of ABSSSI at TOC - mPP Population | |
| Table 14.2.4.1 | Resolution or Near Resolution of ABSSSI at EOT - ITT Population | 49 |
| Table 14.2.4.2 | Resolution or Near Resolution of ABSSSI at EOT - mITT Population | |
| Table 14.2.4.3 | Resolution or Near Resolution of ABSSSI at EOT - mCE Population | |
| Table 14.2.4.4 | Resolution or Near Resolution of ABSSSI at EOT - PP Population | 50 |
| Table 14.2.4.5 | Resolution or Near Resolution of ABSSSI at EOT - mPP Population | 50 |
| Table 14.2.5.1 | Summary of Clinical Response at EOT and TOC - PP Population | 5 |
| Table 14.2.5.2 | Summary of Clinical Response at EOT and TOC - mPP Population | <b>5</b> ! |
| Table 14.2.6.1 | Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - ITT Population | 52 |
| Table 14.2.6.2 | Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - mITT Population | 52 |
| Table 14.2.6.3 | Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - mCE Population | |
| Table 14.2.6.4 | Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - PP Population | 53 |
| Table 14.2.6.5 | Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - mPP Population | 53 |
| Table 14.2.7.1 | Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - ITT Population | 53 |
| Table 14.2.7.2 | Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - mITT Population | |
| Table 14.2.7.3 | Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - mCE Population | |
| Table 14.2.7.4 | Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - PP Population | |
| Table 14.2.7.5 | Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - mPP Population | 54 |
| Table 14.2.8.1 | Time to Resolution of Signs and Symptoms of ABSSSI - ITT Population | 55 |
| Table 14.2.8.2 | Time to Resolution of Signs and Symptoms of ABSSSI - mITT Population | |
| Table 14.2.8.3 | Time to Resolution of Signs and Symptoms of ABSSSI - mCE Population | 50 |
| Table 14.2.8.4 | Time to Resolution of Signs and Symptoms of ABSSSI - PP Population | 56 |
| Table 14.2.8.5 | Time to Resolution of Signs and Symptoms of ABSSSI - mPP Population | |
| Table 14.2.9.1 | Percent of Resolution of Signs and Symptoms of ABSSSI - ITT Population | 5′ |
| Table 14.2.9.2 | Percent of Resolution of Signs and Symptoms of ABSSSI - mITT Population | 5′ |
| Table 14.2.9.3 | Percent of Resolution of Signs and Symptoms of ABSSSI - mCE Population | 5′ |
| Table 14.2.9.4 | Percent of Resolution of Signs and Symptoms of ABSSSI - PP Population | |
| Table 14.2.9.5 | Percent of Resolution of Signs and Symptoms of ABSSSI - mPP Population | |
| Table 14.2.10.1.1 | By Patient Bacteriological Response Rate at EOT - mITT Population | |
| Table 14.2.10.1.2 | By Patient Combined Bacteriological Response Rate at EOT - mITT Population | 60 |
| Table 14.2.10.2.1 | By Patient Bacteriological Response Rate at EOT - mCE Population | |
| Table 14.2.10.2.2 | By Patient Combined Bacteriological Response Rate at EOT - mCE Population | |
| Table 14.2.10.3.1 | By Patient Bacteriological Response Rate at EOT - mPP Population | |
| Table 14.2.10.3.2 | By Patient Combined Bacteriological Response Rate at EOT - mPP Population | |
| Table 14.2.11.1.1 | By Patient Bacteriological Response Rate at TOC - mITT Population | |
| Table 14.2.11.1.2 | By Patient Combined Bacteriological Response Rate at TOC - mITT Population | 60 |

| Table 14.2.11.2.1 | By Patient Bacteriological Response Rate at TOC - mCE Population | 59 |
|---|---|---|
| Table 14.2.11.2.2 | By Patient Combined Bacteriological Response Rate at TOC - mCE Population | 61 |
| Table 14.2.11.3.1 | By Patient Bacteriological Response Rate at TOC - mPP Population | 59 |
| Table 14.2.11.3.2 | By Patient Combined Bacteriological Response Rate at TOC - mPP Population | 61 |
| Table 14.2.12.1 | By Pathogen Bacteriological Response Rate at EOT - mITT Population | 62 |
| Table 14.2.12.2 | By Pathogen Bacteriological Response Rate at EOT - mCE Population | 62 |
| Table 14.2.12.3 | By Pathogen Bacteriological Response Rate at EOT - mPP Population | |
| Table 14.2.13.1 | By Pathogen Bacteriological Response Rate at TOC - mITT Population | |
| Table 14.2.13.2 | By Pathogen Bacteriological Response Rate at TOC - mCE Population | 62 |
| Table 14.2.13.3 | By Pathogen Bacteriological Response Rate at TOC - mPP Population | 62 |
| Table 14.2.14 | Mortality Rate within 28 Days of First Dose of Treatment - ITT Population | 63 |
| Table 14.2.15.1 | Proportions of Patients with a >=20% Reduction in Lesion Size at ETP by Subgroups - ITT Population | 64 |
| Table 14.2.15.2 | Proportions of Patients with a >=20% Reduction in Lesion Size at ETP by Subgroups - PP Population | 65 |
| Table 14.2.16.1 | Resolution or Near Resolution of ABSSSI at TOC by Subgroups - ITT Population | 65 |
| Table 14.2.16.2 | Resolution or Near Resolution of ABSSSI at TOC by Subgroups - PP Population | 66 |
| Table 14.3.1.1 | Overall Summary of Treatment-emergent Adverse Events (TEAEs) - Safety Population | 67 |
| Table 14.3.1.2 | Summary of Treatment-emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term - Safety Population | 69 |
| Table 14.3.1.3 | Summary of Treatment-emergent Adverse Events (TEAEs) by Maximum Severity, MedDRA System Organ Class and Preferred Term - Safety | |
| | Population | 71 |
| Table 14.3.1.4 | Summary of Study Drug-Related Treatment-emergent Adverse Events (TEAEs) by System Organ Class and Preferred Term - Safety Population | 70 |
| Table 14.3.1.5 | Summary of Treatment-emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug by MedDRA System Organ Class and | |
| | Preferred Term - Safety Population | 70 |
| Table 14.3.1.6 | Summary of Treatment-emergent Adverse Events (TEAEs) by Age Group, MedDRA System Organ Class and Preferred Term - Safety Population | |
| Table 14.3.1.7 | Summary of Treatment-emergent Adverse Events (TEAEs) by Creatinine Clearance, MedDRA System Organ Class and Preferred Term - Safety | |
| | Population | 74 |
| Table 14.3.1.8 | Summary of Treatment-emergent Adverse Events (TEAEs) with Frequency > 5% by MedDRA Preferred Term - Safety Population | |
| Table 14.3.1.9 | Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Class and Preferred Term - Safety Population | 70 |
| Table 14.3.1.10 | Summary of Study Drug-related Serious Adverse Events (SAEs) by MedDRA System Organ Class and Preferred Term - Safety Population | 70 |
| Table 14.3.1.11 | Summary of Serious Adverse Events (SAEs) Leading to Death by MedDRA System Organ Class and Preferred Term - Safety Population | 70 |
| Table 14.3.1.12 | Summary of Serious Adverse Events (SAEs) with Frequency > 5% by MedDRA Preferred Term - Safety Population | 75 |
| Table 14.3.2.1 | Listing of Treatment-emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug - Safety Population | 77 |
| Table 14.3.2.2 | Listing of Serious Adverse Events (SAEs) - Safety Population | 78 |
| Table 14.3.2.3 | Listing of Serious Adverse Events (SAEs) Leading to Death - Safety Population | 79 |
| Table 14.3.4.1 | Summary of Laboratory Test Results and Change from Baseline by Visit: Hematology - Safety Population | 80 |
| Table 14.3.4.2 | Summary of Laboratory Test Results and Change from Baseline by Visit: Chemistry including Creatinine Clearance - Safety Population | 81 |
| Table 14.3.4.3 | Summary of Laboratory Test Results and Change from Baseline by Visit: Urinalysis - Safety Population | 81 |
| Table 14.3.4.4 | Shift Table of Laboratory Test Results: Hematology - Safety Population | 82 |
| Table 14.3.4.5 | Shift Table of Laboratory Test Results: Chemistry including Creatinine Clearance - Safety Population | 82 |
| Table 14.3.4.6 | Shift Table of Laboratory Test Results: Urinalysis - Safety Population | 83 |
| Table 14.3.4.7 | Liver Function Test - CTCAE Toxicity Grade - Safety Population | 84 |
| Table 14.3.4.8 | Laboratory Abnormality - Safety Population | |

| Table 14.3.5.1 | Summary of Vital Signs - Body Temperature (°C) - Safety Population | 87 |
|---|---|---|
| Table 14.3.5.2 | Summary of Vital Signs - Heart Rate (bmp) - Safety Population | |
| Table 14.3.5.3 | Summary of Vital Signs - Respiratory Rate (breaths/min) - Safety Population | |
| Table 14.3.5.4 | Summary of Vital Signs - Systolic Blood Pressure (mmHg) - Safety Population | |
| Table 14.3.5.5 | Summary of Vital Signs - Diastolic Blood Pressure (mmHg) - Safety Population | 88 |
| Table 14.3.6.1 | Summary of ECG Measurements by Visit - heart rate - Safety Population | 89 |
| Table 14.3.6.2 | Summary of ECG Measurements by Visit - RR interval - Safety Population | 90 |
| Table 14.3.6.3 | Summary of ECG Measurements by Visit - PR Interval - Safety Population | 90 |
| Table 14.3.6.4 | Summary of ECG Measurements by Visit - QRS Interval - Safety Population | 90 |
| Table 14.3.6.5 | Summary of ECG Measurements by Visit - QT Interval - Safety Population | 90 |
| Table 14.3.6.6 | Summary of ECG Measurements by Visit - QTcB Interval - Safety Population | 90 |
| Table 14.3.6.7 | Summary of ECG Measurements by Visit - QTcF Interval - Safety Population | 90 |
| Table 14.3.6.8 | Summary of ECG Interpretations by Visit - Safety Population | 91 |
| Table 14.3.6.9 | Summary of Marked QT/QTc Prolongation by Visit - Safety Population | <u>92</u> |
| Table 14.3.6.10 | Summary of ECG QTc Interval Prolongation Evaluated Using Median QTcB, by Visit - Safety Population | 93 |
| Table 14.3.6.11 | Summary of ECG QTc Interval Prolongation Evaluated Using Median QTcF, by Visit - Safety Population | 94 |
| Figure 14.2.1.1 | Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI - ITT Population | 95 |
| Figure 14.2.1.2 | Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI - mITT Population | 96 |
| Figure 14.2.1.3 | Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI - mCE Population | 96 |
| Figure 14.2.1.4 | Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI - PP Population | 96 |
| Figure 14.2.1.5 | Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI - mPP Population | 96 |
| Figure 14.2.2.1 | Forest Plots for Subgroup Analysis of the Difference in Early Clinical Response Rate at ETP between Iclaprim and Vancomycin group - ITT | |
| | Population | 97 |
| Figure 14.2.2.2 | Forest Plots for Subgroup Analysis of the Difference in Early Clinical Response Rate at ETP between Iclaprim and Vancomycin group - PP | |
| | Population | 98 |
| Figure 14.2.3.1 | Forest Plots for Subgroup Analysis of the Difference in Clinical Cure Rate at TOC between Iclaprim and Vancomycin group - ITT Population | <mark>98</mark> |
| Figure 14.2.3.2 | Forest Plots for Subgroup Analysis of the Difference in Clinical Cure Rate at TOC between Iclaprim and Vancomycin group - PP Population | <mark>98</mark> |
| Listing 16.2.1.1 | Patients Enrolled - Enrolled Patients | |
| Listing 16.2.1.2 | Patients Disposition - ITT Population | 100 |
| Listing 16.2.1.3 | End of Treatment - ITT Population | 101 |
| Listing 16.2.2.1 | Inclusion and Exclusion Criteria - All enrolled Patients | 102 |
| Listing 16.2.2.2 | Protocol Deviations - ITT Population | |
| Listing 16.2.3 | Study Population - ITT Population | |
| Listing 16.2.4.1 | Demographics - ITT Population | 105 |
| Listing 16.2.4.2 | Baseline Characteristics - ITT Population | 106 |
| Listing 16.2.4.3 | Medical History - ITT Population | |
| Listing 16.2.4.4 | Prior and Concomitant Medication - ITT Population | 108 |
| Listing 16.2.5.1 | Study Drug Administration - Safety Population | |
| Listing 16.2.5.2 | Overall Compliance - Safety Population | |
| Listing 16.2.5.3 | Population Pharmacokinetic - Safety Population | |
| Listing 16.2.6.1 | Blood Culture Results - ITT Population | 112 |

| Listing 16.2.6.2 | Signs and Symptoms of ABSSSI - ITT Population | 113 |
|---|---|---|
| Listing 16.2.6.3 | Signs and Symptoms of ABSSSI - ITT Population | 114 |
| Listing 16.2.6.4.1 | Microbiological Assessment - Patient Level - ITT Population | 115 |
| Listing 16.2.6.4.2 | Microbiological Assessment - Pathogen Level - ITT Population | 116 |
| Listing 16.2.6.5 | Microbiological Assessment of Primary Infection Site - Gram Stain Results - ITT Population | 117 |
| Listing 16.2.6.6 | Microbiological Assessment of Primary Infection Site - Gram Stain Results - ITT Population Significant Surgical Procedures - ITT Population Death - ITT Population Unblinding - ITT Population Unblinding Dose - ITT Population Adverse Events - Safety Population | 118 |
| Listing 16.2.6.7 | Death - ITT Population | 119 |
| Listing 16.2.6.8.1 | Unblinding - ITT Population | 120 |
| Listing 16.2.6.8.2 | Unblinding Dose - ITT Population | 121 |
| Listing 16.2.7 | Adverse Events - Safety Population | 122 |
| Listing 16.2.8.1 | Laboratory Findings in Local Labs at Baseline - Hematology - Safety Population | 123 |
| Listing 16.2.8.2 | Laboratory Findings in Local Labs at Baseline - Chemistry - Safety Population | 124 |
| Listing 16.2.8.3 | Laboratory Findings in Local Labs at Baseline - Urinalysis - Safety Population | 125 |
| Listing 16.2.8.4 | Laboratory Findings in Central Labs by Visit - Hematology - Safety Population | 126 |
| Listing 16.2.8.5 | Laboratory Findings in Central Labs by Visit - Chemistry - Safety Population | 127 |
| Listing 16.2.8.6 | Laboratory Findings in Central Labs by Visit - Urinalysis - Safety Population | 128 |
| Listing 16.2.9 | Vital Signs - Safety Population | 129 |
| Listing 16.2.10.1 | ECG Results - Safety Population | 130 |
| Listing 16.2.10.2 | ECG Assessment - Safety Population | 131 |
| Listing 16.2.11 | Physical Examination Results - Safety Population | 130 |

Table 14.1.1
Overall Summary of Study Populations
Enrolled Patients

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Patients Enrolled | | | XXX |
| Patients Randomized [a] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients Treated | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ITT Population [b] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Microbiological ITT (mITT) Population [c] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Per Protocol (PP) Population [d] PP Microbiologically Evaluable (mPP) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| population [e] Modified Clinically Evaluable (mCE) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Population [f] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Safety Population [g] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Completed Study [h] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

<sup>[</sup>a] The denominator for percentage in each treatment group is the number of total patients randomized.

<sup>[</sup>b] The ITT Population consists of all randomized patients, analysed according to treatment a patient was randomized to. The percentage is based on patients randomized in each treatment group.

<sup>[</sup>c] The mITT Population consists of all randomized patients who had a Gram+ baseline bacterial pathogen identified as the cause of ABSSSI, analysed according to treatment randomized to. The percentage is based on patients randomized in each treatment group.

<sup>[</sup>d] The PP Population consists of all randomized patients who received at least 80% of their planned doses and have adequate assessment for each of the following timepoints: ETP, EOT and TOC, analysed according to treatment received at Visit 1. The percentage is based on patients randomized in each treatment group.

<sup>[</sup>e] The mPP Population consists of mITT patients who received at least 80% of their planned doses and had adequate assessment for each of the following timepoints: ETP, EOT and TOC, analysed according to treatment received at Visit 1. The percentage is based on patients randomized in each treatment group.

<sup>[</sup>f] The mCE Population consists of PP and all patients who may have been excluded from PP due to receipt of prohibited medications, including concomitant antibiotics or high dose steroids. The percentage is based on patients randomized in each treatment group.

[g] The Safety Population consists of all patients who received any study drug during the trial, analysed according to treatment received at Visit 1. The percentage is based on patients randomized in each treatment group.

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

[h] The percentage is calculated from all enrolled patients who signed inform consent in each treatment group. Programming Notes:

Enrolled = informed consent. Counts for enrolled patients will only be presented in the total column.

Program Name: Date Generated: Page x of y

Document Version: 2016-08-16T22:39:26 

Table 14.1.2.1
Summary of Study Completion
ITT Population

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Patients who completed study | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Primary reason for early discontinuation | on of | | |
| study | | | |
| Adverse Event | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Pregnancy | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Death | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Lost To Follow-up | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Non-Compliance With Study Drug | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Investigator Decision | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Protocol Violation | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Study Terminated By Sponsor | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Screen Failure | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Withdrew Consent | xxx (xx.x) | xxx (xx.x) | xxx ( xx.x) |
| Other | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Gram-positive bacteremia | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Gram-negative bacteremia | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

Note: Percentages of patients with each primary reason calculated based on the number of patients not completing the study; all other percentages are calculated based on the ITT Population within each treatment group.

Programming Notes:

Obtain reasons for early discontinuation from CRF.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.1.2.2 Summary of Study Completion - Safety Population Add:

Footnote: Note: Percentages of patients with each primary reason calculated based on the number of patients not completing the study; all other percentages are calculated based on the Safety Population within each treatment group.

Delete:

Footnote: Note: Percentages of patients with each primary reason calculated based on the number of patients not completing the study; all other percentages are calculated based on the ITT Population within each treatment group.


Table 14.1.2.3

Summary of Treatment Completion
ITT Population

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Patients who discontinued treatment | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Primary reason for discontinuation of | | | |
| treatment: | | | |
| Adverse Event | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Investigator Decision | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Pregnancy | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Protocol Deviation | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Withdrew Consent | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Lost to Follow-Up | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Sponsor Decision | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Unblinding | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Lack of Efficacy | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Screen Failure | xxx ( xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death | xxx ( xx.x) | xxx (xx.x) | xxx (xx.x) |
| Other | xxx ( xx.x) | xxx (xx.x) | xxx (xx.x) |

Note: Percentages of patients with each primary reason calculated based on the number of patients not completing the study; all other percentages are calculated based on the ITT Population within each treatment group.

Programming Notes:

Obtain reasons for early discontinuation from CRF.

Program Name: Date Generated:

Page x of y

Repeat for the following displays:

Table 14.1.2.4 Summary of Treatment Completion - Safety Population Add:

Footnote: Note: Percentages of patients with each primary reason calculated based on the number of patients not completing the study; all other percentages are calculated based on the Safety Population within each treatment group.

Delete:

Footnote: Note: Percentages of patients with each primary reason calculated based on the number of patients not completing the study; all other percentages are calculated based on the ITT Population within each treatment group.

Table 14.1.3
Study Sample Sizes by Country and Center
Enrolled Patients

| Region | Country | Center | Number of<br>Patients<br>enrolled | Treatment<br>group | Randomized | Valid<br>for ITT | Valid<br>for<br>mITT | Valid<br>for PP | Valid<br>for<br>mPP | Valid<br>for<br>mCE | Valid<br>for<br>Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Overall | | | XX | Total | XX | xx | xx | XX | xx | xx | XX |
| 0.01011 | | | **** | Iclaprim | XX | XX | XX | XX | XX | XX | XX |
| | | | | Vancomycin | XX | XX | XX | XX | XX | XX | XX |
| North America | xxxxxxxxxx | Xxxxxx | xx | Total | xx | XX | xx | XX | XX | xx | xx |
| | | | | Iclaprim | XX | XX | XX | XX | XX | XX | XX |
| | | | | Vancomycin | xx | XX | XX | XX | XX | XX | xx |
| | xxxxxxxxxx | Xxxxxx | XX | Total | xx | XX | xx | XX | XX | xx | xx |
| | | | | Iclaprim | XX | XX | XX | XX | XX | XX | XX |
| | | | | Vancomycin | XX | XX | XX | XX | XX | XX | XX |
| Europe | xxxxxxxxxx | Xxxxxx | XX | Total | xx | XX | xx | XX | XX | xx | xx |
| | | | | Iclaprim | XX | XX | XX | XX | XX | XX | XX |
| | | | | Vancomycin | XX | XX | XX | XX | XX | XX | XX |

Program Name: Page x of y

Date Generated:

| Analysis<br>Population | Treatment<br>group | N | Number<br>completed<br>study | Number<br>completed<br>ETP | Number<br>completed<br>EOT | Number<br>completed<br>TOC | Number of Discontinua tion of treatment |
|---|---|---|---|---|---|---|---|
| T.M.M. | m-1-1 | | | | | | |
| ITT | Total | XX | XX | XX | XX | XX | XX |
| | Iclaprim | XX | XX | XX | XX | XX | XX |
| | Vancomycin | XX | XX | XX | XX | XX | XX |
| mITT | Total | XX | XX | xx | XX | xx | XX |
| | Iclaprim | XX | XX | XX | XX | XX | xx |
| | Vancomycin | XX | XX | xx | XX | XX | XX |
| PP | Total | XX | XX | XX | XX | xx | xx |
| | Iclaprim | XX | XX | XX | XX | XX | XX |
| | Vancomycin | XX | XX | XX | XX | XX | XX |
| | vancomycin | 2121 | 2121 | 2121 | 7171 | 7171 | **** |
| mPP | Total | XX | XX | XX | XX | XX | xx |
| | Iclaprim | XX | XX | XX | XX | XX | XX |
| | Vancomycin | XX | XX | XX | XX | XX | XX |
| mCE | Total | xx | XX | XX | XX | xx | xx |
| | Iclaprim | XX | XX | XX | XX | XX | XX |
| | Vancomycin | XX | XX | XX | XX | XX | XX |
| | <u> -</u> | | | | | | |
| Safety | Total | XX | XX | XX | XX | XX | XX |
| | Iclaprim | XX | XX | XX | XX | XX | XX |
| | Vancomycin | XX | XX | XX | XX | XX | XX |

Program Name: Page x of y

Date Generated:

Table 14.1.5.1

Summary of Major Protocol Violations/Deviations

ITT Population

| Protocol Violation | <pre>Iclaprim (N = xxx) n (%)</pre> | Vancomycin (N = xxx) n (%) | Total<br>(N = xxx)<br>n (%) |
|---|---|---|---|
| Subjects with at Least 1 Major Protocol Violation | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Major Protocol Violation 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

etc

The violations/deviations were identified prior to data unblinding. Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.1.5.2 Summary of Major Protocol Violations/Deviations - mITT Population

Table 14.1.6
Summary of Patients Validity
All Randomized Patients

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Patients valid for ITT analysis | | | |
| (Randomized Patients) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients valid for Safety analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients valid for mITT analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients valid for PP analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients valid for mPP analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients valid for mCE analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| xcluded from Safety analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Never took study drug | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| scluded from mITT analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Non-Gram-positive pathogen at baseline | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ASO titer positive for S. pyogenes | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| xcluded from PP analysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Non-compliance with study drug | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No efficacy data for any ETP evaluation | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No efficacy data for any EOT evaluation | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No efficacy data for any TOC evaluation | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

<repeat for each population defined in SAP>

Note: Patients in ITT and mITT are grouped according to the randomized treatment group. Patients in PP, mPP, mCE and safety populations are analysed as treated.

Programming Notes:

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

The values of categorical variables are sorted in coded order. Multiple reasons for exclusion from the analysis are possible. All data sets defined in the SAP are to be included in the table. Display reason(s) for exclusion from the population as defined in SAP.

Program Name: Date Generated: Page x of y


Table 14.1.7.1 Summary of Demography ITT Population

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Age (Years) [a] | | | |
| n | XXX | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | xxx, xxx | xxx, xxx | xxx, xxx |
| Age Categories (years) n (%) | | | |
| n | xxx | XXX | XXX |
| 18-39 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 40-64 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 65+ | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Sex, n (%) | | | |
| n | xxx | xxx | XXX |
| Male | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Female | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Race, n (%) | | | |
| n | xxx | XXX | XXX |
| American Indian or Alaska Native | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Asian | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Black or African American | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| White | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Other | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Multi-racial | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Ethnicity, n (%) | | | |
| n | XXX | XXX | XXX |
| Hispanic or Latino | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No Hispanic or Latino | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Not Reported | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

| Unknown | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
|---|---|---|---|
| (kg) | | | |
| n | xxx | xxx | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xxx, xxx | xxx, xxx | xxx, xxx |
| (m) | | | |
| n | xxx | xxx | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | xxx, xxx | xxx, xxx | xxx, xxx |
| (kg/m2) | | | |
| n | xxx | XXX | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | XX.X | XX.X | XX.X |
| Min, Max | XXX, XXX | XXX, XXX | XXX, XXX |
| | (kg) n Mean (SD) Median Min, Max (m) n Mean (SD) Median Min, Max (kg/m2) n Mean (SD) Median Mean (SD) | (kg) n xxx Mean (SD) xx.x (xx.xx) Median xx.x Min, Max xxx (m) xxx n xxx Mean (SD) xx.x Median xxx (kg/m2) xxx n xxx Mean (SD) xx.x Median xx.x Median xx.x | (kg) n xxx xxx Mean (SD) xx.x (xx.xx) xx.x (xx.xx) Median xx.x xx.x Min, Max xxx, xxx xxx, xxx (m) xxx xxx Mean (SD) xx.x (xx.xx) xx.x Median xxx xxx Min, Max xxx xxx xxx (kg/m2) xxx xxx xxx n xxx xxx xxx Mean (SD) xxxx xxxx xxx Median xxx xxxx xxx |

Note: Denominators for percentages are based on the number of patients with non-missing data in each treatment group for the relevant variable.

[a] Age is calculated as (calendar months from birth to informed consent -  $I(day\ of\ informed\ consent < day\ of\ birth))/12$ , and will be reported as whole years.

Program Name: Date Generated: Page x of y

Repeat for the following displays: Table 14.1.7.2 Summary of Demography - mITT Population

Table 14.1.7.3 Summary of Demography - PP Population

Table 14.1.7.4 Summary of Demography - mPP Population

Table 14.1.7.5 Summary of Demography - mCE Population

Table 14.1.7.6 Summary of Demography - Safety Population

Table 14.1.8.1
Baseline Disease Characteristics
ITT Population

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = XXX) |
| | n (응) | n (%) | n (%) |
| Lesion Type | | | |
| Major Cutaneous Abscess, n (%) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| | xxx ( xx.x) | , , | · |
| Cellulitis/ Erysipelas, n (%) | , , | xxx ( xx.x) | xxx ( xx.x) |
| Wound Infection, n(%) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Lesion Size at Baseline (cm²) | | | |
| n | xxx | xxx | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | xx.x | xx.x | XX.X |
| Min,Max | xxx, xxx | xxx, xxx | XXX, XXX |
| Receipt of Prior Antibiotics | | | |
| (based on IVRS) | | | |
| Yes | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No | xxx ( xx.x) | xxx ( xx.x) | XXX ( XX.X) |
| 140 | AAA ( AA•A) | AAA ( AA.A) | AAA ( AA.A) |
| Blood Culture at Baseline | | | |
| Positive | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |
| Negative | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |
| CrCL (mL/min) | | | |
| N | XXX | XXX | XXX |
| >=90 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 60-89 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 30-59 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 15-29 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| <15 or hemodialysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Any Severe Infection[a] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram-positive Pathogen | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram-positive PLUS Gram-negative Pathogen | , , | xxx ( xx.x) | xxx (xx.x) |

| MRSA | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
|---|---|---|---|
| MSSA | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Multiple Pathogens | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Single Pathogen | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Only S. pyogenes by ASO | | | |
| Titer and Blood Culture at baseline | | | |
| ASO positive only | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Culture positive only | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ASO and Culture both positive | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ASO and Culture both negative | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

CrCL=Creatinine Clearance, MRSA=Methicillin-resistant Staphylococcus aureus, MSSA=Methicillin-sensitive Staphylococcus aureus
Note: Denominators for percentages are based on the number of patients with non-missing data in each treatment group for the relevant variable.

- [a] Severe infection is defined as meeting one or more of the following criteria:
- a. fulfilled the published definition for systemic inflammatory response syndrome (SIRS) by having >=2 of the following findings: body temperature >38°C or <36°C, heart rate >90 bpm, respiration rate >20 breaths/minute, and WBC >12000/mm3 or <4000/mm3 or >10% bands;
- b. Evaluated as having severe tenderness or severe erythema at the infection site; and
- c. Positive blood cultures at baseline

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.1.8.2 Baseline Disease Characteristics - mITT Population

Table 14.1.8.3 Baseline Disease Characteristics - PP Population

Table 14.1.8.4 Baseline Disease Characteristics - mPP Population

Table 14.1.8.5 Baseline Disease Characteristics - mCE Population

Table 14.1.8.6 Baseline Disease Characteristics - Safety Population

Table 14.1.9
Summary of Medical History
ITT Population

| | Iclaprim | Vancomycin | Total |
|------------------------------------|-------------|-------------|-------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Patients with Any Medical History? | | | |
| No | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Yes | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Medical History | | | |
| System Organ Class 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 3 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 4 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| System Organ Class 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Preferred Term 2 | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |
| Preferred Term 3 | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |
| Preferred Term 4 | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |

The denominator for percentages is the number of patients in the ITT Population for each treatment group.

Note: This table contains counts of patients. If a patient had more than one medical history within a preferred term, the patient is counted only once within a preferred term. If a patient had more than one medical history within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Note: MedDRA Version 18.1 used for coding.

Program Name: Date Generated: Page x of y

Table 14.1.10.1
Prior Medications
ITT Population

| ATC CLASS (ATC Level 2) SUBCLASS (ATC Level 4)/ GENERIC TERM | <pre>Iclaprim (N = xxx) n (%)</pre> | Vancomycin<br>(N = xxx)<br>n (%) | Total<br>(N = xxx)<br>n (%) |
|---|---|---|---|
| Number(%) of patients with at least one medication | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ANY MEDICATION CLASS | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Any medication | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ATC Class Term | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 1/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 2/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 3/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 4/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

<continue other ATC class and subclass>

Note: Patients in ITT are grouped according to the randomized treatment group.

Prior medications are those taken prior to the first dose date of treatment and within the preceding 30 days of the Informed Consent. Programming Notes:

Includes antibiotics started prior to first dose of study drug. Program Name: Date Generated:

Page x of y

 $\begin{array}{c} \text{Table 14.1.10.2} \\ \text{Concomitant Medication Excluding Antibiotics} \\ \text{ITT Population} \end{array}$ 

| ATC CLASS (ATC Level 2) | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| SUBCLASS (ATC Level 4)/ | (N = xxx) | (N = xxx) | (N = xxx) |
| GENERIC TERM | n (%) | n (%) | n (%) |
| Number(%) of patients with at least one medication | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ANY MEDICATION CLASS | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Any medication | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ATC Class Term | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 1/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 2/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 3/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 4/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

<continue other ATC class and subclass>

Note: Patients in ITT are grouped according to the randomized treatment group.

Note: Concomitant medications are those with a start date on or after the first dose date of treatment, or those with a start date before the first dose date of treatment and a stop date on or after the first dose date of treatment.

Program Name: Date Generated: Page x of y

Table 14.1.10.3

Concomitant Antibiotic Medication

ITT Population

| ATC CLASS (ATC Level 2) SUBCLASS (ATC Level 4)/ GENERIC TERM | <pre>Iclaprim (N = xxx) n (%)</pre> | Vancomycin (N = xxx) n (%) | Total (N = xxx) n (%) |
|---|---|---|---|
| Number(%) of patients with at least one medication | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ANY MEDICATION CLASS | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Any medication | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ATC Class Term | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 1/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 2/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 3/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| SUBCLASS 4/ GENERIC TERM | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

<continue other ATC class and subclass>

Note: Patients in ITT are grouped according to the randomized treatment group.

Note: Concomitant antibiotics are selected from medications that are checked as antibiotic in the CRF Program Name: Date Generated:

Page x of y

Table 14.1.10.4

Summary of Significant Procedures by Visit

ITT Population

| | <pre>Iclaprim (N = xxx) n (%)</pre> | Vancomycin (N = xxx) n (%) | Total<br>(N = xxx)<br>n (%) |
|---|---|---|---|
| Number (%) of patients receiving any significant procedures at Visit 2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Debridement | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Incision and drainage | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Other | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

<Repeat for all visits with significant procedures performed>

Note: Patients in ITT are grouped according to the randomized treatment group. Program Name:

Date Generated:

Page x of y

| | Iclaprim | Vancomycin | Total |
|----------------------|-------------|-------------|-------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| ender to Palpitation | n (%) | n (%) | n (%) |
| Baseline | | | |
| None | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Mild | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Moderate | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Severe | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 7isit 2 | | | |
| None | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Mild | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Moderate | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Severe | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

< Repeat for all visits where signs and symptoms were assessed >

Program Name:

Date Generated:

Page x of y

Repeat for the following displays:
Table 14.1.11.1.2

Clinical Signs and Symptoms of ABSSSI by Visit: Tender to Palpitation - PP Population

Table 14.1.11.2.1

Clinical Signs and Symptoms of ABSSSI by Visit: Tender to Palpitation - mCE Population

Table 14.1.11.2.1

Clinical Signs and Symptoms of ABSSSI by Visit: Erythema - ITT Population

Table 14.1.11.2.2

Clinical Signs and Symptoms of ABSSSI by Visit: Erythema - PP Population

Clinical Signs and Symptoms of ABSSSI by Visit: Erythema - mCE Population


Table 14.1.11.2.3

```
Table 14.1.11.3.1
                      Clinical Signs and Symptoms of ABSSSI by Visit: Edema - ITT Population
Table 14.1.11.3.2
                      Clinical Signs and Symptoms of ABSSSI by Visit: Edema - PP Population
Table 14.1.11.3.3
                      Clinical Signs and Symptoms of ABSSSI by Visit: Edema - mCE Population
Table 14.1.11.4.1
                      Clinical Signs and Symptoms of ABSSSI by Visit: Purulent Drainage/Discharge - ITT Population
Table 14.1.11.4.2
                      Clinical Signs and Symptoms of ABSSSI by Visit: Purulent Drainage/Discharge - PP Population
Table 14.1.11.4.3
                      Clinical Signs and Symptoms of ABSSSI by Visit: Purulent Drainage/Discharge - mCE Population
Table 14.1.11.5.1
                      Clinical Signs and Symptoms of ABSSSI by Visit: Fluctuance - ITT Population
Table 14.1.11.5.2
                      Clinical Signs and Symptoms of ABSSSI by Visit: Fluctuance - PP Population
Table 14.1.11.5.3
                      Clinical Signs and Symptoms of ABSSSI by Visit: Fluctuance - mCE Population
Table 14.1.11.6.1
                      Clinical Signs and Symptoms of ABSSSI by Visit: Induration - ITT Population
Table 14.1.11.6.2
                      Clinical Signs and Symptoms of ABSSSI by Visit: Induration - PP Population
Table 14.1.11.6.3
                      Clinical Signs and Symptoms of ABSSSI by Visit: Induration - mCE Population
Table 14.1.11.7.1
                      Clinical Signs and Symptoms of ABSSSI by Visit: Ulceration - ITT Population
Table 14.1.11.7.2
                      Clinical Signs and Symptoms of ABSSSI by Visit: Ulceration - PP Population
Table 14.1.11.7.3
                      Clinical Signs and Symptoms of ABSSSI by Visit: Ulceration - mCE Population
Table 14.1.11.8.1
                      Clinical Signs and Symptoms of ABSSSI by Visit: Necrotic Tissue - ITT Population
Table 14.1.11.8.2
                      Clinical Signs and Symptoms of ABSSSI by Visit: Necrotic Tissue - PP Population
Table 14.1.11.8.3
                      Clinical Signs and Symptoms of ABSSSI by Visit: Necrotic Tissue - mCE Population
Table 14.1.11.9.1
                      Clinical Signs and Symptoms of ABSSSI by Visit: Localized Pain - ITT Population
Table 14.1.11.9.2
                      Clinical Signs and Symptoms of ABSSSI by Visit: Localized Pain - PP Population
Table 14.1.11.9.3
                      Clinical Signs and Symptoms of ABSSSI by Visit: Localized Pain - mCE Population
```

| Table | 14.1.11.10.1 | Clinical | Signs | and | Symptoms | of | ABSSSI | bу | Visit: | Swelling - ITT Population |
|---|---|---|---|---|---|---|---|---|---|---|
| Table | 14.1.11.10.2 | Clinical | Signs | and | Symptoms | of | ABSSSI | bу | Visit: | Swelling - PP Population |
| Table | 14.1.11.10.3 | Clinical | Signs | and | Symptoms | of | ABSSSI | рà | Visit: | Swelling - mCE Population |
| Table | 14.1.11.11.1 | Clinical | Signs | and | Symptoms | of | ABSSSI | рÀ | Visit: | Chills - ITT Population |
| Table | 14.1.11.11.2 | Clinical | Signs | and | Symptoms | of | ABSSSI | bу | Visit: | Chills - PP Population |
| Table | 14.1.11.11.3 | Clinical | Signs | and | Symptoms | of | ABSSSI | by | Visit: | Chills - mCE Population |
| Table | 14.1.11.12.1 | Clinical | Signs | and | Symptoms | of | ABSSSI | bу | Visit: | Fever - ITT Population |
| Table | 14.1.11.12.2 | Clinical | Signs | and | Symptoms | of | ABSSSI | рÀ | Visit: | Fever - PP Population |
| Table | 14.1.11.12.3 | Clinical | Signs | and | Symptoms | of | ABSSSI | by | Visit: | Fever - mCE Population |

| | Iclaprim | Vancomycin | Total |
|-----------------------------------|-------------|-------------|-------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Baseline | | | |
| Was a specimen obtained for the c | ulture? | | |
| Yes | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Specimen type | | | |
| Aerobic blood culture | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Anaerobic blood culture | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Infection site culture | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Was culture performed? | | | |
| Yes | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Did the culture grow an organism? | | | |
| Yes | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Was the organism a pathogen? | | | |
| | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Yes | | | |

Program Name: Date Generated: Page x of y
$\begin{array}{c} \text{Table 14.1.12.2} \\ \text{Summary of Culture Specimen for Lesion Type by Visit} \\ \text{ITT Population} \end{array}$ 

| Lesion Type | Iclaprim | Vancomycin | Total |
|-------------------------|-------------|-------------|-------------|
| Specimen Type | (N = xxx) | (N = xxx) | (N = xxx) |
| Genus Species | n (%) | n (%) | n (%) |
| Baseline | | | |
| Major Cutaneous Abscess | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Aerobic Blood Culture | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Genus1 Species1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Genus1 Species2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| • • • | | | |
| Anaerobic Blood Culture | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Genus1 Species1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| ••• | | | |
| Infection Site Culture | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Genus1 Species1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| | , | , | |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Cellulitis/Erysipelas | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Aerobic Blood Culture | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Genusl Species1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| • • • | | | |
| • • • | | | |
| Wound Infection | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

Table 14.1.12.3

Microbiological Assessment of Primary Infection Site - Gram Stain
ITT Population

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Method of Collection | | | |
| Needle aspirate | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Biopsy | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |
| Tissue/fluid/pus surgically obtained | | | |
| in operating room | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Tissue/fluid/pus obtained during | , , | , , | • |
| during bedside procedure | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram Stain, n (%) | | | |
| Gram Stain Not Done | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| No Bacteria | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram-positive cocci (clusters) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram-positive cocci (chains) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram-negative cocci | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram-positive bacilli | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Gram-negative bacilli | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

Table 14.1.12.4

Blood Culture Results by Visit
ITT Population

| | Iclaprim | Vancomycin | Total | |
|---|---|---|---|---|
| | (N = XXX) | (N = xxx) | (N = xxx) | |
| | n (%) | n (%) | n (%) | |
| aseline | | | | |
| lood Cultures, n (%) | | | | |
| Positive | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) | |
| Negative | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) | |
| Missing Data/Not Done | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) | |
| isit 2 | | | | |
| •• | | | | |
| Repeat for all visits where cu | lture was performed > | | | |
| <u>*</u> | · | | | |
| rogram Name: | Date Generat | ed: | | Page x of y |

 $\begin{array}{c} \text{Table 14.1.12.5} \\ \text{Gram-positive Pathogens Occurring in Patients at Baseline} \\ \text{ITT Population} \end{array}$ 

| | <pre>Iclaprim (N = xxx) n (%)</pre> | Vancomycin (N = xxx) n (%) | Total (N = xxx) n (%) |
|---|---|---|---|
| Pathogen Pathogen 1 Pathogen 2 | XXX ( XX.X) | xxx ( xx.x) | xxx ( xx.x) |
| | XXX ( XX.X) | xxx ( xx.x) | xxx ( xx.x) |

•••

<Continue for other identified pathogens>

Note: Patients may have more than one pathogens.

Program Name: Date Generated:

Page x of y

Treatment Group: treatment 1

| Pathogen 1 | gen 1 Frequency of MIC (mcg/mL) (n, %, Cumulative %) | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Test [a] | 0.0625 | 0.125 | 0.25 | 0.5 | 1.0 | 2.0 | 4.0 | 8.0 | 16.0 | 32.0 | 64.0 | MIC50 | MIC90 |
| AMP, N=xx | XX<br>XX.X | xx<br>xx.x | XX<br>XX.X | xx<br>xx.x | XX<br>XX.X | xx<br>xx.x | XX<br>XX.X | xx<br>xx,x | XX<br>XX.X | xx<br>xx.x | xx<br>xx.x | XX.X | xx.x |
| | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | |

<Continue for other antibiotics tested>

<Continue for other pathogens identified at baseline>

N = number of isolates; MIC = Minimum Inhibitory Concentration; MIC50 = MIC at which 50% of isolates tested are inhibited; MIC90 = MIC at which 90% of isolates tested are inhibited.

- [a] Antibiotics Tested: AMP=Ampicillin, .....
- [b] MIC50 and MIC90 values are only reported when >=10 isolates were tested.

Table 14.1.13.1

Summary of Treatment Compliance
ITT Population

| | Iclaprim | Vancomycin | Total |
|-------------------|---------------|---------------|----------------|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| ompliance (%) | | | |
| n | XXX | xxx | XXX |
| Mean (SD) | xx.x ( xx.xx) | xx.x ( xx.xx) | xx.xx ( xx.xx) |
| Median | xx.x | XX.X | XX.X |
| Min | xx.x | XX.X | XX.X |
| Max | XX.X | xx.x | XX.X |
| Range | xxx, xxx | xxx, xxx | xxx, xxx |
| verall Compliance | | | |
| n | XXX | xxx | XXX |
| <80.0% | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 80.0% to 100.0% | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| >100.0% | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Note: Percentage compliance is calculated as (number of doses received / number of doses scheduled)\*100%. Compliance is defined as percentage compliance at least 80.0%.

Table 14.1.13.2

Summary of Treatment Exposure: Duration in Days
Safety Population

| | Iclaprim (N = xxx) n (%) | Vancomycin (N = xxx) n (%) |
|----------------|--------------------------|----------------------------|
| uration (days) | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min | XX.X | XX.X |
| Max | XX.X | XX.X |
| Range | XX.X, XX.X | XX.X, XX.X |

The denominator for percentages is the number of patients with non-missing data in the Safety Population for each treatment group. Note: Duration of exposure calculated as (date of last dose - date of first dose) + 1.

| | Iclaprim<br>(N = xxx)<br>n (%) | Vancomycin (N = xxx) n (%) | % Difference (Iclaprim - Vancomycin) |
|---|---|---|---|
| Early Clinical Response [a] 95% CI [b] p-value [c] | xxx ( xx.x)<br>(x.xx , x.xx) | xxx ( xx.x)<br>(x.xx , x.xx) | xx.x<br>(x.xx , x.xx)<br>x.xxx |

<sup>[</sup>a] Early Clinical Response is defined as >=20% reduction in lesion size at ETP.

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.2.1 Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - mITT Population Add:

The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

# Delete:

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

<sup>[</sup>b] The two-sided 95% CI is based on the exact binomial CI for the proportions of the 2 groups, and is based on the z-test with unpooled variance estimate for the difference in the 2 proportions. If the lower bound of 95% CI is greater than -0.10, NI is concluded.

<sup>[</sup>c] p-value is for the NI test with significance level of 0.025.

Table 14.2.2.2 Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - mCE Population Add:

The denominator for percentages is the number of patients with non-missing data in the mCE Population for each treatment group.

## Delete:

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.2.3 Proportions of Patients with a >=20% Reduction in Lesion Size at ETP - PP Population

The denominator for percentages is the number of patients with non-missing data in the PP Population for each treatment group.

## Delete:

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.2.4 Proportions of Patients with a  $\geq$ =20% Reduction in Lesion Size at ETP - mPP Population Add:

The denominator for percentages is the number of patients with non-missing data in the mPP Population for each treatment group.

#### Delete:

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

 $\begin{array}{c} {\tt Table \ 14.2.3.1} \\ {\tt Resolution \ or \ Near \ Resolution \ of \ ABSSSI \ at \ TOC} \\ {\tt ITT \ Population} \end{array}$ 

| | Iclaprim (N = xxx) n (%) | Vancomycin<br>(N = xxx)<br>n (%) | % Difference (Iclaprim - Vancomycin) |
|---|---|---|---|
| Clinical cure rate | xxx ( xx.x) | xxx ( xx.x) | XX.X |
| 95% CI [a] | (x.xx , x.xx) | (x.xx, x.xx) | (x.xx , x.xx) |
| p-value [b] | | | x.xxx |

[a] The two-sided 95% CI is based on the exact binomial CI for the proportions of the 2 groups, and is based on the z-test with unpooled variance estimate for the difference in the 2 proportions. If the lower bound of 95% CI is greater than -0.10, NI is concluded.

[b] p-value is for the NI test with significance level of 0.025.

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.3.2 Resolution or Near Resolution of ABSSSI at TOC - mITT Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.3.3 Resolution or Near Resolution of ABSSSI at TOC - mCE Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mCE Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.3.4 Resolution or Near Resolution of ABSSSI at TOC - PP Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the PP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.3.5 Resolution or Near Resolution of ABSSSI at TOC - mPP Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mPP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.4.1 Resolution or Near Resolution of ABSSSI at EOT - ITT Population

Table 14.2.4.2 Resolution or Near Resolution of ABSSSI at EOT - mITT Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.4.3 Resolution or Near Resolution of ABSSSI at EOT - mCE Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mCE Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.4.4 Resolution or Near Resolution of ABSSSI at EOT - PP Population

Add

Footnote: The denominator for percentages is the number of patients with non-missing data in the PP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.4.5 Resolution or Near Resolution of ABSSSI at EOT - mPP Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mPP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

| Clinical Response | Iclaprim | Vancomycin |
|-------------------|-------------|-------------|
| | (N = xxx) | (N = xxx) |
| | n (%) | n (%) |
| EOT | | |
| n [a] | | |
| Cure | xxx ( xx.x) | xxx ( xx.x) |
| Failure | xxx ( xx.x) | xxx ( xx.x) |
| Indeterminate | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) |
| COC | | |
| n [a] | | |
| Cure | xxx ( xx.x) | xxx ( xx.x) |
| Failure | xxx ( xx.x) | xxx ( xx.x) |
| Indeterminate | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx (xx.x) |

[a] Number of patients who completed the visit at the corresponding time point. Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.2.5.2 Summary of Clinical Response at EOT and TOC - mPP Population

| | Iclaprim (N = xxx) n (%) | Vancomycin (N = xxx) n (%) | % Difference (Iclaprim - Vancomycin) |
|---|---|---|---|
| Patients with severe infection, n | xxx | xxx | |
| Clinical cure | xxx ( xx.x) | xxx ( xx.x) | xx.x |
| 95% CI [a] | (x.xx, x.xx) | (x.xx, x.xx) | (x.xx , x.xx) |
| p-value [b] | | | X.XXX |

[a] The two-sided 95% CI is based on the exact binomial CI for the proportions of the 2 groups, and is based on the z-test with unpooled variance estimate for the difference in the 2 proportions. If the lower bound of 95% CI is greater than -0.10, NI is concluded.

[b] p-value is for the NI test with significance level of 0.025.

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.6.2 Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - mITT Population Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

## Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.6.3 Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - mCE Population Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mCE Population for each treatment group.

## Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.6.4 Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - PP Population Add.

Footnote: The denominator for percentages is the number of patients with non-missing data in the PP Population for each treatment group.

#### Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.6.5 Resolution or Near Resolution of ABSSSI at TOC among Patients with Severe Infection at Baseline - mPP Population Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mPP Population for each treatment group.

# Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.7.1 Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - ITT Population

Table 14.2.7.2 Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - mITT Population Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

## Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.7.3 Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - mCE Population Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mCE Population for each treatment group.

#### Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.7.4 Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - PP Population Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the PP Population for each treatment group.

## Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.7.5 Resolution or Near Resolution of ABSSSI at EOT among Patients with Severe Infection at Baseline - mPP Population Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mPP Population for each treatment group.

### Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

| Tender to Palpitation | Iclaprim | Vancomycin |
|--------------------------------|----------------|-----------------|
| | (N = xxx) | (N = xxx) |
| | n (%) | n (%) |
| Number of Patients with Events | xxx ( xx.x) | xxx ( xx.x) |
| Number of Patients Censored | xxx ( xx.x) | xxx ( xx.x) |
| Time to event (days) | | |
| Median [a] | XX.X | XX.X |
| 95% CI for Median [a] | (xx.xx, xx.xx) | (xx.xx , xx.xx) |
| 25% and 75% (Percentiles) | xx.x, xx.x | XX.X, XX.X |
| Range [b] | xx.x, xx.x | XX.X, XX.X |
| P-value (Log-Rank Test) | | x.xxx |
| Unadjusted Hazard Ratio [c] | | x.xx |
| 95% CI | | [x.xxx, x.xxx] |

<Repeat for other signs and symptoms of ABSSSI>

Time to resolution of signs and symptoms of ABSSSI is defined as: first date with no signs and symptoms of ABSSSI (in log form) post treatment - date of first dose + 1.

Note: Denominators for percentages are based on the number of patients in the ITT Population

- [a] Kaplan-Meier estimates.
- [b] Including censored observations.
- [c] Hazard ratio is estimated using Cox's Proportional Hazards Model for Iclaprim versus Vancomycin, and the confidence interval is based on inverting the Wald test. If the upper bound of 95% CI is less than 1.10, NI is concluded. The p-value is based on one-sided Wald test with significant level of 0.025.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.8.2 Time to Resolution of Signs and Symptoms of ABSSSI - mITT Population Add:

Note: Denominators for percentages are based on the number of patients in the mITT Population

Note: Denominators for percentages are based on the number of patients in the ITT Population

- Table 14.2.8.3 Time to Resolution of Signs and Symptoms of ABSSSI mCE Population Add:
- Note: Denominators for percentages are based on the number of patients in the mCE Population Delete:
- Note: Denominators for percentages are based on the number of patients in the ITT Population
- Table 14.2.8.4 Time to Resolution of Signs and Symptoms of ABSSSI PP Population Add:
- Note: Denominators for percentages are based on the number of patients in the PP Population Delete:
- Note: Denominators for percentages are based on the number of patients in the ITT Population
- Table 14.2.8.5 Time to Resolution of Signs and Symptoms of ABSSSI mPP Population Add:
- Note: Denominators for percentages are based on the number of patients in the mPP Population Delete:
- Note: Denominators for percentages are based on the number of patients in the ITT Population

 $\begin{array}{c} \text{Table 14.2.9.1} \\ \text{Percent of Resolution of Signs and Symptoms of ABSSSI} \\ \text{ITT Population} \end{array}$ 

| % of Resolution of Tender to | Iclaprim | Vancomycin | |
|---|---|---|---|
| Palpitation | (N = xxx) | (N = xxx) | |
| | n (%) | n (%) | |
| Baseline | | | |
| n | xxx | XXX | |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) | |
| Median | XX.X | XX.X | |
| Min,Max | XX.X, XX.X | xx.x, xx.x | |
| ETP | | | |
| ••• | | | |
| <continue for="" other="" td="" visits="" with<=""><td>the assessment&gt;</td><td></td><td></td></continue> | the assessment> | | |
| <pre><repeat and="" for="" other="" pre="" signs="" sym<=""></repeat></pre> | ptoms of ABSSSI> | | |
| n is the number of patients wi | th non-missing data i | n the ITT Population for each treatment group. | |
| Program Name: | Date | Generated: | Page x of y |
| Repeat for the following displa | vs: | | |
| | <del>-</del> | mptoms of ABSSSI - mITT Population | |
| Footnote: n is the number Delete: | of patients with non- | missing data in the mITT Population for each treatme | ent group. |
| Footnote: n is the number | of patients with non- | missing data in the ITT Population for each treatmen | nt group. |
| Table 14.2.9.3 Percent of Resol Add: | ution of Signs and Sy | mptoms of ABSSSI - mCE Population | |
| Footnote: n is the number Delete: | of patients with non- | missing data in the mCE Population for each treatmen | nt group. |
| Footnote: n is the number | of patients with non- | missing data in the ITT Population for each treatmen | nt group. |

 $\hbox{\tt Table 14.2.9.4 Percent of Resolution of Signs and Symptoms of ABSSSI - PP Population } \\$ 

Add

Footnote: n is the number of patients with non-missing data in the PP Population for each treatment group.

Delete:

Footnote: n is the number of patients with non-missing data in the ITT Population for each treatment group.

 $\hbox{\tt Table 14.2.9.5 Percent of Resolution of Signs and Symptoms of ABSSSI - mPP Population } \\$ 

Add:

Footnote: n is the number of patients with non-missing data in the mPP Population for each treatment group.

Delete:

Footnote: n is the number of patients with non-missing data in the ITT Population for each treatment group.

| | Iclaprim | Vancomycin |
|---------------------------------------|-------------|-------------|
| | (N = xxx) | (N = xxx) |
| | n (%) | n (%) |
| Number of Patients with Gram-positive | | |
| Pathogen response assessment | XXX | XXX |
| Bacteriological Response | | |
| Eradication | xxx ( xx.x) | xxx ( xx.x) |
| Presumed Eradication | xxx ( xx.x) | xxx (xx.x) |
| Persistence | xxx ( xx.x) | xxx ( xx.x) |
| Presumed Persistence | xxx ( xx.x) | xxx ( xx.x) |
| Indeterminate | xxx ( xx.x) | xxx ( xx.x) |
| Superinfection | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | XXX ( XX.X) |

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.10.2.1 By Patient Bacteriological Response Rate at EOT - mCE Population

Table 14.2.10.3.1 By Patient Bacteriological Response Rate at EOT - mPP Population

Table 14.2.11.1.1 By Patient Bacteriological Response Rate at TOC - mITT Population

Table 14.2.11.2.1 By Patient Bacteriological Response Rate at TOC - mCE Population

Table 14.2.11.3.1 By Patient Bacteriological Response Rate at TOC - mPP Population

| | Iclaprim<br>(N = xxx)<br>n (%) | Vancomycin (N = xxx) n (%) | % Difference (Iclaprim - Vancomycin) |
|---|---|---|---|
| Eradication/Presumed Eradication 95% CI [a] | xxx ( xx.x)<br>(xx.xx , xx.xx) | xxx ( xx.x)<br>(xx.xx , xx.xx) | xx.x |

Repeat for the following displays:

Table 14.2.10.2.2 By Patient Combined Bacteriological Response Rate at EOT - mCE Population

Add

Footnote: The denominator for percentages is the number of patients with non-missing data in the mCE Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

Table 14.2.10.3.2 By Patient Combined Bacteriological Response Rate at EOT - mPP Population

Footnote: The denominator for percentages is the number of patients with non-missing data in the mPP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

Table 14.2.11.1.2 By Patient Combined Bacteriological Response Rate at TOC - mITT Population

Table 14.2.11.2.2 By Patient Combined Bacteriological Response Rate at TOC - mCE Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mCE Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

Table 14.2.11.3.2 By Patient Combined Bacteriological Response Rate at TOC - mPP Population

Footnote: The denominator for percentages is the number of patients with non-missing data in the mPP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the mITT Population for each treatment group.

 $\begin{array}{c} \text{Table 14.2.12.1} \\ \text{By Pathogen Bacteriological Response Rate at EOT} \\ \text{mITT Population} \end{array}$ 

| | Iclaprim | Vancomycin |
|----------------------|-------------|-------------|
| | (N = xxx) | (N = xxx) |
| | n (%) | n (%) |
| Pathogen 1 | | |
| Eradication | xxx ( xx.x) | xxx ( xx.x) |
| Presumed Eradication | xxx ( xx.x) | xxx ( xx.x) |
| Persistence | xxx ( xx.x) | xxx ( xx.x) |
| Presumed Persistence | xxx ( xx.x) | xxx ( xx.x) |
| Indeterminate | xxx ( xx.x) | xxx ( xx.x) |
| Superinfection | xxx ( xx.x) | xxx ( xx.x) |
| Missing | xxx ( xx.x) | xxx ( xx.x) |

<Continue for all pathogens identified>

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.12.2 By Pathogen Bacteriological Response Rate at EOT - mCE Population

Table 14.2.12.3 By Pathogen Bacteriological Response Rate at EOT - mPP Population

Table 14.2.13.1 By Pathogen Bacteriological Response Rate at TOC - mITT Population

Table 14.2.13.2 By Pathogen Bacteriological Response Rate at TOC - mCE Population

Table 14.2.13.3 By Pathogen Bacteriological Response Rate at TOC - mPP Population

| | (N = xxx) | (N = xxx) | (N = XXX) |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| Patients Who Died within 28 Days :<br>of First Dose of Treatment | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

The denominator for percentages is the number of patients with non-missing date of first dose. Program Name:

Date Generated:

Page x of y

| | Total (N = xxx) | Iclaprim (N = xxx) | Vancomycin (N = xxx) | |
|---|---|---|---|---|
| | (N - XXX) | n (%) | n (%) | % Difference[a] (95% CI[b]) |
| .ge Group | | | | |
| 18-39 | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| 40-64 | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| 65+ | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| ex | | | | |
| Male | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| Female | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| Race | | | | |
| White | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| Non-white | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| Cr Clearance (mL/min) | | | | |
| >=90 | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| 60-89 | XXX | xxx (xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| 30-59 | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| 15-29 | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| <15 or hemodialysis | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| ositive Blood Culture | | | | |
| t Baseline | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| RSA | xxx | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| SSA | XXX | xxx ( xx.x) | xxx (xx.x) | xx.x (x.xx, x.xx) |
| ultiple pathogens | xxx | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| ingle pathogen | XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |

Patients with S. pyogenes

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

| xxx | xxx ( xx.x) | xxx ( xx.x) | xx.x ( $x.xx$ , $x.xx$ ) |
|---|---|---|---|
| XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| ction | | | |
| XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x (x.xx, x.xx) |
| XXX | xxx ( xx.x) | xxx ( xx.x) | xx.x ( $x.xx$ , $x.xx$ ) |
| | xxx<br>xxx<br>xxx<br>ction<br>xxx | xxx | xxx |

MRSA=Methicillin-resistant Staphylococcus aureus, MSSA=Methicillin-sensitive Staphylococcus aureus.

The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.2.15.2 Proportions of Patients with a >=20% Reduction in Lesion Size at ETP by Subgroups - PP Population

Footnote: The denominator for percentages is the number of patients with non-missing data in the PP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

Table 14.2.16.1 Resolution or Near Resolution of ABSSSI at TOC by Subgroups - ITT Population

<sup>[</sup>a] The difference is defined as the % of iclaprim - % of vancomycin.

<sup>[</sup>b] The two-sided 95% CI is based on the exact binomial CI for the proportions of the 2 groups, and is based on the z-test with unpooled variance estimate for the difference in the 2 proportions.

Table 14.2.16.2 Resolution or Near Resolution of ABSSSI at TOC by Subgroups - PP Population

Add:

Footnote: The denominator for percentages is the number of patients with non-missing data in the PP Population for each treatment group.

Delete:

Footnote: The denominator for percentages is the number of patients with non-missing data in the ITT Population for each treatment group.

| | Iclaprim | Vancomycin | Total |
|---|---|---|---|
| | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Patients with Any TEAEs [a] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Any TEAEs | | | |
| Patients with Mild TEAEs | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Moderate TEAEs | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Severe TEAEs | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Missing Severity | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Study Drug Related TEAEs [b] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with TEAE Leading to Discon- | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| tinuation of Study Drug | | | |
| Patients with Serious Adverse Events (SAEs) | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Study Drug Related SAEs [b] | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with SAE Leading to Death | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Patients with Study Drug Related SAE | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Leading to Death | | | |
| Patients with a SAE Leading to Study | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Drug Discontinuation | | | |
| Patients with a SAE Leading to Discon- | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| tinuation from Study | | | |

The denominator for percentages is the number of patients in the Safety Population

<sup>[</sup>a] TEAEs are defined as events with start date on or after the date of first dose of study drug through the end of study, or events with start date prior to the date of first dose of treatment whose severity worsens on or after the date of first dose of treatment through the end of study. Note that study drug exposure is 5-14 days.

<sup>[</sup>b] Included are AEs considered probably related or related to study drug and AEs with unknown or missing relationship to study drug.

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

Table 14.3.1.2

Summary of Treatment-emergent Adverse Events (TEAEs) by MedDRA System Organ Class and Preferred Term Safety Population

| System Organ Class | Iclaprim | Vancomycin | Total |
|-------------------------|-------------|-------------|-------------|
| Preferred Term | (N = xxx) | (N = xxx) | (N = xxx) |
| | n (%) | n (%) | n (%) |
| Patients with Any TEAEs | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| System Organ Class 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 3 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| etc. | | | |
| System Organ Class 2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 3 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| etc. | | | |

The denominator for percentages is the number of patients in the Safety Population

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Programming Notes:

SOC will be sorted alphabetically and PT will be sorted by descending overall total. Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

Table 14.3.1.4 Summary of Study Drug-Related Treatment-emergent Adverse Events (TEAEs) by System Organ Class and Preferred Term - Safety Population

#### Add:

Footnote: Note: Included are AEs considered related or probably related to study drug and AEs with unknown or missing relationship to study drug.

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term and for the episode with the maximum severity. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

#### Delete

Footnote: Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Table 14.3.1.5 Summary of Treatment-emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug by MedDRA System Organ Class and Preferred Term - Safety Population

Table 14.3.1.9 Summary of Serious Adverse Events (SAEs) by MedDRA System Organ Class and Preferred Term - Safety Population

Table 14.3.1.10 Summary of Study Drug-related Serious Adverse Events (SAEs) by MedDRA System Organ Class and Preferred Term - Safety Population

Table 14.3.1.11 Summary of Serious Adverse Events (SAEs) Leading to Death by MedDRA System Organ Class and Preferred Term - Safety Population

Table 14.3.1.3

Summary of Treatment-emergent Adverse Events (TEAEs) by Maximum Severity, MedDRA System Organ Class and Preferred Term Safety Population

| System Organ Class | Iclaprim | Vancomycin | Total |
|-------------------------|-------------|-------------|-------------|
| Preferred Term | (N = xxx) | (N = xxx) | (N = xxx) |
| Maximum Severity | n (%) | n (%) | n (%) |
| Patients with Any TEAEs | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Mild | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Moderate | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Severe | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing Severity | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| System Organ Class 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Mild | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Moderate | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Severe | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing Severity | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Mild | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Moderate | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Severe | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing Severity | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |
| Mild | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Moderate | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Severe | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Missing Severity | xxx ( xx.x) | xxx ( xx.x) | xxx (xx.x) |
| etc | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

The denominator for percentages is the number of patients in the Safety Population

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term and for the episode that is most related to the study drug. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Programming Notes:

SOC will be sorted alphabetically and PT will be sorted by descending overall total.

Program Name: Date Generated: Page x of y


Table 14.3.1.6 Summary of Treatment-emergent Adverse Events (TEAEs) by Age Group, MedDRA System Organ Class and Preferred Term Safety Population

| System Organ Class | Iclaprim | Vancomycin | Total |
|-------------------------|-------------|-------------|-------------|
| Preferred Term | (N = xxx) | (N = xxx) | (N = xxx) |
| Age Group | n (%) | n (%) | n (%) |
| Patients with Any TEAEs | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx (xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 18-64 | xxx (xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 65+ | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| System Organ Class 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 18-64 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 65+ | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 18-64 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 65+ | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 2 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 18-64 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Age 65+ | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| etc | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

The denominator for percentages is the number of patients in the Safety Population

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

# Programming Notes:

SOC will be sorted alphabetically and PT will be sorted by descending overall total. Program Name: Date Generated:

Page x of y

Table 14.3.1.7

Summary of Treatment-emergent Adverse Events (TEAEs) by Creatinine Clearance, MedDRA System Organ Class and Preferred Term Safety Population

| System Organ Class | Iclaprim | Vancomycin | Total |
|-------------------------|-------------|-------------|-------------|
| Preferred Term | (N = xxx) | (N = xxx) | (N = xxx) |
| CrCL(mL/min) | n (%) | n (%) | n (%) |
| Patients with Any TEAEs | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| >= 90 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 60-89 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 30-59 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 15-29 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| <15 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Hemodialysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| System Organ Class 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| >= 90 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 60-89 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 30-59 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 15-29 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| <15 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Hemodialysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Overall | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| >= 90 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 60-89 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 30-59 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| 15-29 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| <15 | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Hemodialysis | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| etc | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

The denominator for percentages is the number of patients in the Safety Population

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Programming Notes:

SOC will be sorted alphabetically and PT will be sorted by descending overall total.

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.3.1.12 Summary of Serious Adverse Events (SAEs) with Frequency > 5% by MedDRA Preferred Term - Safety Population


Table 14.3.1.8

Summary of Treatment-emergent Adverse Events (TEAEs) with Frequency > 5% by MedDRA Preferred Term Safety Population

| Preferred Term | Iclaprim (N = xxx) n (%) | Vancomycin (N = xxx) n (%) | Total (N = xxx) n (%) |
|---|---|---|---|
| Patients with Any TEAEs of<br>Frequency >10% | xxx ( xx.x) | xxx ( xx.x) | xxx ( xx.x) |
| Preferred Term 1<br>Preferred Term 2<br>Preferred Term 3<br>etc. | xxx ( xx.x)<br>xxx ( xx.x)<br>xxx ( xx.x) | xxx ( xx.x)<br>xxx ( xx.x)<br>xxx ( xx.x) | xxx ( xx.x)<br>xxx ( xx.x)<br>xxx ( xx.x) |

The denominator for percentages is the number of patients in the Safety Population PT is sorted in descending order of frequency in the iclaprim group

Note: This table contains counts of patients. If a patient experienced more than one episode of an adverse event, the patient is counted only once within a preferred term. If a patient experienced more than one adverse event within a system organ class, the patient is counted once for each preferred term and once for the system organ class.

Programming Notes:

SOC will be sorted alphabetically and PT will be sorted by descending overall total. Program Name:

Date Generated:

Table 14.3.2.1 Listing of Treatment-emergent Adverse Events (TEAEs) Leading to Discontinuation of Study Drug Safety Population

Treatment: Treatment 1

| Center | Patient | AE No. | System Organ Class/<br>Preferred Term/<br>Verbatim [a] | Onset Date (day)[b]/<br>End Date (day)[b]/<br>Duration (days) | TEAE/<br>Severity | Relationship<br>to Study<br>Drug/ADR? | Treatment<br>required?/<br>Action<br>Taken[c] | Outcome | SAE? |
|---|---|---|---|---|---|---|---|---|---|
| Xxxxxx | xxx | xx | ********************/ **************** | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/<br>xx | Yes/<br>Mild | Not related/<br>No | Yes/<br>No | Completely recovered | No |
| | | xx | *******************/ ***************** | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/<br>xx | No/<br>Moderate | Probably not<br>related/<br>No | No/<br>Discontinu<br>ed | Death | Yes |
| xxxxxx | xxx | XX | *******************/ ***************** | DDMMMYYYY (xx)/<br>Ongoing | Yes/<br>Severe | Probably<br>related/<br>Yes | Yes/<br>Interrupte<br>d | Ongoing | Yes |
| | | | | | | Related/<br>Yes | | Recovered to stability | No |

Sort by treatment group, subject, AE start date, end date, and preferred term.

Program Name: Date Generated:

<sup>[</sup>a] Coded using MedDRA Dictionary (Version 18.1)

<sup>[</sup>b] Relative to the day of first dose of study treatment.

<sup>[</sup>c] Action Taken: No =xxx; Stop = xxxxxx xxxx; Disc = xxxx xxxxxxxxx; Remedy = xxxx xxxxxxx xxxxxxxx. Programming Notes:

Table 14.3.2.2 Listing of Serious Adverse Events (SAEs) Safety Population

Treatment: Treatment 1

| Center | Patient | AE No. | System Organ Class/<br>Preferred Term/<br>Verbatim [a] | Onset Date (day)[b]/<br>End Date (day)[b]/<br>Duration (days) | TEAE/<br>Severity | Relationship<br>to Study<br>Drug/ADR? | Treatment<br>required?/<br>Action<br>Taken[c] | Outcome | SAE<br>Type<br>[d] |
|---|---|---|---|---|---|---|---|---|---|
| Xxxxxx | xxx | XX | ************************************** | DDMMMYYYY (xx)/ DDMMMYYYY (xx)/ xx | Yes/<br>Mild | Not related/ | Yes/<br>No | Completely recovered | LT |
| | | XX | ************************************** | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/<br>xx | No/<br>Moderate | Probably not<br>related/<br>No | No/<br>Discontinu<br>ed | Death | Death |
| xxxxx | xxx | XX | ************************************** | DDMMMYYYY (xx)/<br>Ongoing | Yes/<br>Severe | Probably<br>related/<br>Yes | Yes/<br>Interrupte<br>d | Ongoing | PD |
| | | | | | | Related/<br>Yes | | Recovered to stability | Hosp |
| | | | | | | | | | Other |

[a] Coded using MedDRA Dictionary (Version 18.1)

#### Programming Notes:

Sort by treatment group, subject, AE start date, end date, and preferred term. Program Name:

Date Generated: Page x of y

<sup>[</sup>b] Relative to the day of first dose of study treatment.

<sup>[</sup>c] Action Taken: No =xxx; Stop = xxxxxx xxxx; Disc = xxxx xxxxxxxxx; Remedy = xxxx xxxxxxx xxxxxxx.

<sup>[</sup>d] SAE Type: LT = Life-threatening; PD = Permanently Disabling; Hosp = Hospitalization/prolonged hospitalization; C = Congenital anomaly; CC = Current condition.

Table 14.3.2.3 Listing of Serious Adverse Events (SAEs) Leading to Death Safety Population

Treatment: Treatment 1

| Center | Patient | AE No. | System Organ Class/<br>Preferred Term/<br>Verbatim [a] | Onset Date (day)[b]/<br>End Date (day)[b]/<br>Duration (days) | TEAE/<br>Severity | Relationship<br>to Study<br>Drug/ADR? | Treatment<br>required?/<br>Action<br>Taken[c] | Date of<br>Death<br>(days)[a] | Cause<br>of<br>Death |
|---|---|---|---|---|---|---|---|---|---|
| Xxxxx | xxx | XX | ************************************** | DDMMMYYYY (xx)/ DDMMMYYYYY (xx)/ xx | Yes/<br>Mild | Not related/<br>No | Yes/<br>No | DDMMMYYYY<br>(xx) | Xxxxx |
| | | XX | ************************************** | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/<br>xx | No/<br>Moderate | Probably not<br>related/<br>No | No/<br>Discontinu<br>ed | DDMMMYYYY<br>(xx) | Xxxxx |
| xxxxxx | XXX | xx | ***********************/ ************* | | | | | | |

Sort by treatment group, subject, AE start date, end date, and preferred term.

<sup>[</sup>a] Coded using MedDRA Dictionary (Version 18.1)

<sup>[</sup>b] Relative to the day of first dose of study treatment.

| | | bareey roparacion |
|-------------------------------------|----------------|-------------------|
| Hematocrit (%) | | |
| | Iclaprim | Vancomycin |
| Study Visit | (N = xxx) | (N = XXX) |
| | n (%) | n (%) |
| Baseline | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min, Max | xx.x, xx.x | XX.X, XX.X |
| <pre><visit> Pre-dose</visit></pre> | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx (x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | XX.X, XX.X |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx (x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | XX.X, XX.X |
| (Visit> Post-dose | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx (x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | |
| n | xxx | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx (x.xxx) |
| Median | XX.X | XX.X |
| Min, Max | XX.X, XX.X | XX.X, XX.X |

#### [Continue for remaining post-baseline time points]

Note: This table only presents central lab (CCLS) results for patients with non-missing data at baseline and the time point of

Note: Low = below lower limit of normal range, Normal = within normal limits, High = above upper limit of normal range.

Programming Notes:

Repeat the table for other continuous Hematology variables. See SAP for variable list.

Note: Only the tests with continuous values will be summarized.

Program Name: Date Generated:

Page x of y

Repeat for the following displays:

Table 14.3.4.2 Summary of Laboratory Test Results and Change from Baseline by Visit: Chemistry including Creatinine Clearance - Safety Population

Add:

Note to Programmer: Repeat the table for other continuous Chemistry including Creatinine Clearance variables. See SAP for variable list.

Delete:

Note to Programmer: Repeat the table for other continuous Hematology variables. See SAP for variable list.

Table 14.3.4.3 Summary of Laboratory Test Results and Change from Baseline by Visit: Urinalysis - Safety Population

Note to Programmer: Repeat the table for other continuous Urinalysis variables. See SAP for variable list.

Note to Programmer: Repeat the table for other continuous Hematology variables. See SAP for variable list.

Table 14.3.4.4
Shift Table of Laboratory Test Results: Hematology
Safety Population

| | Iclaprim<br>(N = xxx)<br>Baseline | Vancomycin<br>(N = xxx)<br>Baseline |
|---|---|---|
| Hematocrit (%) | L N H Tot | L N H Tot |
| <pre><visit></visit></pre> | | |
| Low (L) | XXX XXX XXX | XXX XXX XXX XXX |
| Normal (N) | XXX XXX XXX | XXX XXX XXX XXX |
| High (H) | XXX XXX XXX | XXX XXX XXX XXX |
| Total (Tot) | XXX XXX XXX | XXX XXX XXX |
| <visit></visit> | | |
| Low (L) | XXX XXX XXX | XXX XXX XXX XXX |
| Normal (N) | XXX XXX XXX | XXX XXX XXX XXX |
| High (H) | XXX XXX XXX | XXX XXX XXX XXX |
| Total (Tot) | XXX XXX XXX XXX | XXX XXX XXX XXX |

<Continue for all visits>

Note: This table only presents results for patients with non-missing data at baseline and the time point of interest.

Note: Low = below lower limit of normal range, Normal = within normal limits, High = above upper limit of normal range.

Programming Notes:

Repeat the table for other Hematology variables. See SAP for variable list.

Program Name: Date Generated:

Page x of y

Repeat for the following displays:

Table 14.3.4.5 Shift Table of Laboratory Test Results: Chemistry including Creatinine Clearance - Safety Population

Note to Programmer: Repeat the table for other Chemistry including Creatinine Clearance variables. See SAP for variable list.

Note to Programmer: Use categories negative, positive, missing.

Delete:

Note to Programmer: Repeat the table for other Hematology variables. See SAP for variable list.

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

Table 14.3.4.6 Shift Table of Laboratory Test Results: Urinalysis - Safety Population Add:

Note to Programmer: Repeat the table for other Urinalysis variables. See SAP for variable list. Delete:  $\frac{1}{2}$ 

Note to Programmer: Repeat the table for other Hematology variables. See SAP for variable list.

Table 14.3.4.7 Liver Function Test - CTCAE Toxicity Grade Safety Population

| Laboratory Test (Unit) | Grade Criteria | Worst CTCAE<br>Grade | Iclaprim<br>(N = xxx) | Vancomycin (N = xxx) |
|---|---|---|---|---|
| | | 02000 | n (%) | n (%) |
| aseline | | | | |
| Number (%) of Patients | | | xxx ( xx.x) | xxx ( xx.x) |
| ALP (U/L) | 1.25-2.5x ULN | Grade 1 | xxx ( xx.x) | xxx ( xx.x) |
| | 2.6-5.0x ULN | Grade 2 | xxx ( xx.x) | xxx ( xx.x) |
| | 5.1-10.0x ULN | Grade 3 | xxx ( xx.x) | xxx ( xx.x) |
| | >10.0x ULN | Grade 4 | xxx ( xx.x) | xxx ( xx.x) |
| | | Grade 1-4 | xxx ( xx.x) | xxx ( xx.x) |
| ALT (U/L) | 1.25-2.5x ULN | Grade 1 | xxx ( xx.x) | xxx ( xx.x) |
| | 2.6-5.0x ULN | Grade 2 | xxx ( xx.x) | xxx ( xx.x) |
| | 5.1-10.0x ULN | Grade 3 | xxx ( xx.x) | xxx ( xx.x) |
| | >10.0x ULN | Grade 4 | xxx ( xx.x) | xxx ( xx.x) |
| | | Grade 1-4 | xxx ( xx.x) | xxx ( xx.x) |
| AST (U/L) | 1.25-2.5x ULN | Grade 1 | xxx ( xx.x) | xxx ( xx.x) |
| | 2.6-5.0x ULN | Grade 2 | xxx ( xx.x) | xxx ( xx.x) |
| | 5.1-10.0x ULN | Grade 3 | xxx ( xx.x) | xxx ( xx.x) |
| | >10.0x ULN | Grade 4 | xxx ( xx.x) | xxx ( xx.x) |
| | | Grade 1-4 | xxx (xx.x) | xxx ( xx.x) |
| Total bilirubin | 1.1-1.5x ULN | Grade 1 | xxx ( xx.x) | xxx ( xx.x) |
| (mg/dL) | 1.6-2.5x ULN | Grade 2 | xxx ( xx.x) | xxx ( xx.x) |
| , 5. , | 2.6-5.0x ULN | Grade 3 | xxx ( xx.x) | xxx (xx.x) |
| | >5.0x ULN | Grade 4 | xxx (xx.x) | xxx (xx.x) |
| | | Grade 1-4 | xxx ( xx.x) | xxx ( xx.x) |

Final 1.0

Statistical Analysis Plan Motif BioSciences Protocol ICL-24-ABSSSI2

ALP=alkaline phosphatase, ALT=alanine aminotransferase, AST=aspartate aminotransferase.

The percentages are based on patients with at least one laboratory value for that specific lab test at the corresponding visit.

Program Name:

Date Generated:

Page x of y


Table 14.3.4.8
Laboratory Abnormality
Safety Population

| Laboratory Variable | Iclaprim<br>(N = xxx) | Vancomycin<br>(N = xxx) |
|-----------------------|-----------------------|-------------------------|
| | Baseline | Baseline |
| | num/denom (%) | num/denom (%) |
| Visit 2 | | |
| Laboratory category 1 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| Parameter 1 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| Parameter 2 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| Parameter 3 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| Laboratory category 2 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| Parameter 1 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| Parameter 2 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| Parameter 3 | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |
| | xxx/xxx (xx.x%) | xxx/xxx (xx.x%) |

<Continue with additional category and analysts and for remaining post-baseline visits>

CNS=clinically not significant, CS=clinically significant.

Note: The denominator (denom) represents the number of patients at baseline with normal or abnormal CNS laboratory assessment who also had at least one valid laboratory value after start of treatment. Patients with missing or abnormal CS values at baseline are not included in the denominator.

Note: The numerator (num) represents the number of patients with at least one abnormal CS laboratory assessment after the start of treatment who had a normal or abnormal CNS laboratory assessment at baseline.

Note: Unscheduled visits were also considered in the summary.

 $\begin{array}{c} \text{Table 14.3.5.1} \\ \text{Summary of Vital Signs - Body Temperature (°C)} \\ \text{Safety Population} \end{array}$ 

| | Iclaprim | Vancomycin |
|---------------------------|----------------|----------------|
| Study Visit | (N = xxx) | (N = xxx) |
| beddy vibie | n (%) | n (%) |
| | ( • / | |
| Baseline | | |
| n | XXX | xxx |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | xx.x, xx.x |
| <visit> Pre-dose</visit> | | |
| n | xxx | xxx |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | XX.X, XX.X |
| Change from Baseline | | |
| n | XXX | xxx |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | xx.x, xx.x |
| <visit> Post-dose</visit> | | |
| n | xxx | xxx |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | xx.x, xx.x |
| Change from Baseline | | |
| n | xxx | xxx |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | xx.x, xx.x |

#### [Continue for remaining post-baseline time points]

Baseline values are defined as the last non-missing scheduled or unscheduled values collected prior to first dose of study drug.

Program Name:

Page x of y

Repeat for the following displays:

Table 14.3.5.2 Summary of Vital Signs - Heart Rate (bmp) - Safety Population

Delete:

Footnote: Baseline values are defined as the last non-missing scheduled or unscheduled values collected prior to first dose of study drug.

Table 14.3.5.3 Summary of Vital Signs - Respiratory Rate (breaths/min) - Safety Population

Footnote: Baseline values are defined as the last non-missing scheduled or unscheduled values collected prior to first dose of study drug.

Table 14.3.5.4 Summary of Vital Signs - Systolic Blood Pressure (mmHq) - Safety Population

Delete

Footnote: Baseline values are defined as the last non-missing scheduled or unscheduled values collected prior to first dose of study drug.

Table 14.3.5.5 Summary of Vital Signs - Diastolic Blood Pressure (mmHg) - Safety Population

Footnote: Baseline values are defined as the last non-missing scheduled or unscheduled values collected prior to first dose of study drug.

Table 14.3.6.1

Summary of ECG Measurements by Visit - heart rate

Safety Population

| heart rate (bpm) | | |
|---------------------------|----------------|----------------|
| | Iclaprim | Vancomycin |
| Study Visit | (N = xxx) | (N = XXX) |
| | n (%) | n (%) |
| Baseline | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | XX.X, XX.X |
| <visit> Pre-dose</visit> | | |
| n | xxx | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min, Max | xx.x, xx.x | XX.X, XX.X |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | xx.x, xx.x |
| <visit> Post-dose</visit> | | |
| n | xxx | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Min,Max | xx.x, xx.x | XX.X, XX.X |
| Change from Baseline | | |
| n | XXX | XXX |
| Mean (SD) | xx.xx ( x.xxx) | xx.xx ( x.xxx) |
| Median | XX.X | XX.X |
| Median | AA • A | |

## [Continue for remaining post-baseline time points]

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Table 14.3.6.2 Summary of ECG Measurements by Visit - RR interval - Safety Population

Table 14.3.6.3 Summary of ECG Measurements by Visit - PR Interval - Safety Population

Table 14.3.6.4 Summary of ECG Measurements by Visit - QRS Interval - Safety Population

Table 14.3.6.5 Summary of ECG Measurements by Visit - QT Interval - Safety Population

Table 14.3.6.6 Summary of ECG Measurements by Visit - QTcB Interval - Safety Population

Table 14.3.6.7 Summary of ECG Measurements by Visit - QTcF Interval - Safety Population

Table 14.3.6.8 Summary of ECG Interpretations by Visit Safety Population

| | <pre>Iclaprim (N = xxx) n (%)</pre> | Vancomycin (N = xxx) n (%) |
|---|---|---|
| seline | | |
| N | XXX | XXX |
| Normal (N) | xxx ( xx.x) | xxx ( xx.x) |
| Abnormal Not Clinical Significant (ANCS) | xxx ( xx.x) | xxx ( xx.x) |
| Abnormal Clinical Significant (ACS) | xxx ( xx.x) | xxx ( xx.x) |
| /isit> | | |
| N | xxx | XXX |
| Normal (N) | xxx ( xx.x) | xxx ( xx.x) |
| Abnormal Not Clinical Significant (ANCS) | xxx ( xx.x) | xxx ( xx.x) |
| Abnormal Clinical Significant (ACS) | xxx ( xx.x) | xxx ( xx.x) |

< Repeat for all visits where ECG performed >

The denominator for percentages is the number of patients with non-missing data in the Safety Population for each treatment group. Note: N: Normal; ANCS: Abnormal, Not Clinically Significant; ACS: Abnormal, Clinically Significant Page x of y Program Name: Date Generated:

 $\begin{array}{c} {\tt Table \ 14.3.6.9} \\ {\tt Summary \ of \ Marked \ QT/QTc \ Prolongation \ by \ Visit} \\ {\tt Safety \ Population} \end{array}$ 

| | Iclaprim | Vancomycin |
|--------------------------------|-------------|-------------|
| | (N = xxx) | (N = xxx) |
| | n (%) | n (%) |
| Baseline | | |
| n | xxx | xxx |
| Any marked QT/QTc prolongation | xxx ( xx.x) | xxx ( xx.x) |
| Visit 2 | | |
| n | XXX | XXX |
| Any marked QT/QTc prolongation | xxx ( xx.x) | xxx ( xx.x) |
| ETP | | |
| n | XXX | XXX |
| Any marked QT/QTc prolongation | xxx ( xx.x) | xxx ( xx.x) |

The marked QT/QTc prolongation is defined as median QTcF value >500 msec and/or >60 msec different from the pre-dose baseline value. Program Name:

Page x of y

| | Iclaprim | Vancomycin |
|----------------------------------------------|-------------|-------------|
| | (N = xxx) | (N = xxx) |
| | n (%) | n (%) |
| Baseline | | |
| n | XXX | xxx |
| Value > 450 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 480 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 500 ms | xxx ( xx.x) | xxx ( xx.x) |
| Visit 2 | | |
| n | XXX | XXX |
| Value > 450 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 480 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 500 ms | xxx ( xx.x) | xxx ( xx.x) |
| <pre>Increase &gt; 30 ms from baseline</pre> | xxx ( xx.x) | xxx ( xx.x) |
| Increase > 60 ms from baseline | xxx ( xx.x) | xxx ( xx.x) |
| ETP | | |
| n | | |
| Value > 450 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 480 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 500 ms | xxx ( xx.x) | xxx ( xx.x) |
| Increase > 30 ms from baseline | xxx ( xx.x) | xxx ( xx.x) |
| <pre>Increase &gt; 60 ms from baseline</pre> | xxx ( xx.x) | xxx ( xx.x) |

| | Iclaprim | Vancomycin |
|----------------------------------------------|-------------|-------------|
| | (N = xxx) | (N = xxx) |
| | n (%) | n (%) |
| Baseline | | |
| n | XXX | XXX |
| Value > 450 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 480 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 500 ms | xxx ( xx.x) | xxx ( xx.x) |
| Visit 2 | | |
| n | XXX | XXX |
| Value > 450 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 480 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 500 ms | xxx ( xx.x) | xxx ( xx.x) |
| Increase > 30 ms from baseline | xxx ( xx.x) | xxx ( xx.x) |
| Increase > 60 ms from baseline | xxx ( xx.x) | xxx ( xx.x) |
| ETP | | |
| n | | |
| Value > 450 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 480 ms | xxx ( xx.x) | xxx ( xx.x) |
| Value > 500 ms | xxx ( xx.x) | xxx ( xx.x) |
| Increase > 30 ms from baseline | xxx ( xx.x) | xxx ( xx.x) |
| <pre>Increase &gt; 60 ms from baseline</pre> | xxx ( xx.x) | xxx ( xx.x) |

Figure 14.2.1.1 Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI ITT Population



## Programming Notes:

The y-axis will be ticked at every 0.1, and x-axis will be ticked at every 2 days. The y-axis label will be "Probability of Resolution of Tender to Palpitation", and x-axis label will be "Days Since First Dose". The two lines will represent "iclaprim" and "vancomycin" using solid line and dashed line respectively.

<Continue for other signs and symptoms of ABSSSI>

Program Name:

Date Generated:

Page x of y

Repeat for the following displays:

- Figure 14.2.1.2 Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI mITT Population Add:
- Note to Programmer: The y-axis will be ticked at every 0.1, and x-axis will be ticked at every 2 days. The y-axis label will be "Probability of Resolution of ", and x-axis label will be "Days Since First Dose". The two lines will represent "iclaprim" and "vancomycin" using solid line and dashed line respectively.

Note to Programmer: The y-axis will be ticked at every 0.1, and x-axis will be ticked at every 2 days. The y-axis label will be "Probability of Resolution of Tender to Palpitation", and x-axis label will be "Days Since First Dose". The two lines will represent "iclaprim" and "vancomycin" using solid line and dashed line respectively.

- Figure 14.2.1.3 Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI mCE Population Add:
- Note to Programmer: The y-axis will be ticked at every 0.1, and x-axis will be ticked at every 2 days. The y-axis label will be "Probability of Resolution of ", and x-axis label will be "Days Since First Dose". The two lines will represent "iclaprim" and "vancomycin" using solid line and dashed line respectively.

  Delete:

Note to Programmer: The y-axis will be ticked at every 0.1, and x-axis will be ticked at every 2 days. The y-axis label will be "Probability of Resolution of Tender to Palpitation", and x-axis label will be "Days Since First Dose". The two lines will represent "iclaprim" and "vancomycin" using solid line and dashed line respectively.

- Figure 14.2.1.4 Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI PP Population Add:
- Note to Programmer: The y-axis will be ticked at every 0.1, and x-axis will be ticked at every 2 days. The y-axis label will be "Probability of Resolution of ", and x-axis label will be "Days Since First Dose". The two lines will represent "iclaprim" and "vancomycin" using solid line and dashed line respectively.

Note to Programmer: The y-axis will be ticked at every 0.1, and x-axis will be ticked at every 2 days. The y-axis label will be "Probability of Resolution of Tender to Palpitation", and x-axis label will be "Days Since First Dose". The two lines will represent "iclaprim" and "vancomycin" using solid line and dashed line respectively.

Figure 14.2.1.5 Kaplan-Meier Curves for Time to Resolution of Each Sign/Symptom of ABSSSI - mPP Population

Figure 14.2.2.1

Forest Plots for Subgroup Analysis of the Difference in Early Clinical Response Rate at ETP between Iclaprim and Vancomycin group ITT Population



MRSA=Methicillin-resistant Staphylococcus aureus, MSSA=Methicillin-sensitive Staphylococcus aureus

Statistical Analysis Plan
Motif BioSciences

Program Name: Date Generated: Page x of y

Repeat for the following displays:

Protocol ICL-24-ABSSSI2

Figure 14.2.2.2 Forest Plots for Subgroup Analysis of the Difference in Early Clinical Response Rate at ETP between Iclaprim and Vancomycin group - PP Population

Delete

Footnote: MRSA=Methicillin-resistant Staphylococcus aureus, MSSA=Methicillin-sensitive Staphylococcus aureus

Figure 14.2.3.1 Forest Plots for Subgroup Analysis of the Difference in Clinical Cure Rate at TOC between Iclaprim and Vancomycin group - ITT Population

Delete

Footnote: MRSA=Methicillin-resistant Staphylococcus aureus, MSSA=Methicillin-sensitive Staphylococcus aureus

Figure 14.2.3.2 Forest Plots for Subgroup Analysis of the Difference in Clinical Cure Rate at TOC between Iclaprim and Vancomycin group - PP Population

Delete:

Footnote: MRSA=Methicillin-resistant Staphylococcus aureus, MSSA=Methicillin-sensitive Staphylococcus aureus

Final 1.0

Listing 16.2.1.1
Patients Enrolled
Enrolled Patients

Treatment: Treatment 1

| Center | Patient | Date of Informed<br>Consent | Primary Reason for<br>Screen Failure |
|---|---|---|---|
| Xxxxxx | xxx | DDMMMYYYY | Reason 1 Reason 2 |
| Xxxxxx | xxx | DDMMMYYYY | |
| xxxxxx | xxx | DDMMMYYYY | |

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient

Program Name: Date Generated:

Listing 16.2.1.2
Patients Disposition
ITT Population

Treatment: Treatment 1

| Center | Patient | Completed<br>Study | Date of<br>Discontinuation or<br>Completion (Day)[a] | Primary Reason for<br>Discontinuation/<br>Other, specify | If AE,<br>Specify AE<br>No. | If Protocol<br>Violation,<br>Specify | Gram-positive<br>bacteremia? |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxx | No | DDMMMYYYY (xx) | Reason 1/ | | | Yes |
| Xxxxxx | XXX | No | DDMMMYYYY (xx) | Other/ | | | No |
| XXXXXX | xxx | Yes | DDMMMYYYY (xx) | *************************************** | | | |

[a] Relative to date of first dose of study treatment

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient

Variable "Completed Study"=Yes comes from 1st option of "Subject Status" on page "Disposition"

Program Name:

Date Generated:

Listing 16.2.1.3 End of Treatment ITT Population

Treatment: Treatment 1

| Center | Patient | Discontinuation of treatment? | Primary Reason for Discontinuation/Other, specify | If AE,<br>Specify AE<br>No. | Date of First Dose (Day)[a]/ Date of Last Dose (Day)[a] | FU phone call agreed by Patient? |
|---|---|---|---|---|---|---|
| xxxxxx | xxx | Yes | Reason 1/ | | DDMMMYYYY (1)/ | Yes |
| Xxxxxx | xxx | Yes | Other/ | | DDMMMYYYY (xx) DDMMMYYYY (1)/ | No |
| xxxxxx | xxx | No | XXXXXX | | DDMMMYYYY (xx)<br>DDMMMYYYY (1)/ | Yes |
| | | | | | DDMMMYYYY (xx) | |

LFU=Last Follow-up Visit.

[a] Relative to date of first dose of study treatment

Programming Notes:

Repeat for all treatments. Sort by center and patient

Listing 16.2.2.1
Inclusion and Exclusion Criteria
All enrolled Patients

Treatment: Treatment 1

| Center | Patient | Overall eligibility met? | If no, category of criterion | Identifier |
|---|---|---|---|---|
| Xxxxxx | XXX | Yes | | |
| XxxxxX | XXX | No | Inclusion | 5, 6 |
| XXXXXX | XXX | No | Exclusion | 2, 3 |

Refer to Protocol for full descriptions of the Inclusion and Exclusion Criteria.
[a] Relative to the day of first dose of study treatment

# Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient Program Name:

Date Generated:

Page x of y


Final 1.0

Listing 16.2.2.2
Protocol Deviations
ITT Population

Treatment: Treatment 1

| Center | Patient | Any Deviations? | Date | Deviation Category | Details of Deviation |
|---|---|---|---|---|---|
| xxxxxx | xxx | Yes | DDMMMYYYY | xxxxxxxxxxxx | xxxxxxxxxxxxxxx |

Note: Deviations were identified and categorized prior to unblinding. Patients may have more than one violation leading to exclusion from ITT Population

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient

Listing 16.2.3 Study Population ITT Population

Treatment: Treatment 1

| Center E | Patient | Completed<br>Treatment | Completed<br>Study | ITT | mITT | PP | mPP | mCE | Safety |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx > | xxx | Yes<br>No | Yes<br>No | Yes<br>No | Yes<br>No | Yes<br>No | Yes<br>No | Yes<br>No | Yes<br>No |

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient

Final 1.0

Listing 16.2.4.1 Demographics ITT Population

Treatment: Treatment 1

| Center | Patient | Date of Birth | Age (Years) | Sex | Race/<br>Other,<br>specify | Ethnicity |
|---|---|---|---|---|---|---|
| xxxxx | XXX | DDMMMYYYY | XX | Male | Race1 | Ethnicity1 |
| XXXXXX | xxx | DDMMMYYYY | xx | Female | Race2<br>Other/<br>xxxxx | Ethnicity2 |

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient

Program Name: Date Generated:

Listing 16.2.4.2
Baseline Characteristics
ITT Population

Treatment: Treatment 1

| Center | Patient | Lesion Type | Gram-positive pathogen? | CrCL (mL/min) | Date of<br>Randomization<br>(Day)[a] | Randomization<br>Number |
|---|---|---|---|---|---|---|
| xxxxxx | xxx | Wound<br>infection | Yes | | DDMMMYYYY<br>(xx) | xxxxx |

See SAP for definition of severe infection at baseline.

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient Program Name:

Date Generated:

<sup>[</sup>a] Relative to the day of first dose of study treatment

Listing 16.2.4.3 Medical History ITT Population

Treatment: Treatment 1

| Center | Patient | System Organ Code (SOC)/<br>Preferred Term[a] | Verbatim | Start Date (Day[b])/<br>Stop Date (Day[b]) | Ongoing? |
|---|---|---|---|---|---|
| xxxxxx | xxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxx | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx) | No |
| xxxxxx | xxx | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | xxxxxxxxxxxxx | DDMMMYYYY (xx)/ | Yes |
| xxxxxx | xxx | None | | | |

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient, SOC and preferred term.

Program Name:

Date Generated:

<sup>[</sup>a] MedDRA Dictionary (Version 18.1) was used for coding.

<sup>[</sup>b] Relative to the day of first dose of study treatment

## Listing 16.2.4.4 Prior and Concomitant Medication ITT Population

Treatment: Treatment 1

| | | | Therapeutic Class Chemical Subgroup | Prior/ | Dose/Unit/<br>Frequency/ | | Reason or<br>Indication/ | Start Date (day)[b]/<br>Stop Date (day)[b]/ |
|---|---|---|---|---|---|---|---|---|
| Center | Patient | CM No. | Generic Term [a] | Concomitant | Route | Antibiotic? | Other, specify | Duration (days) |
| xx | xxx | xx | xxxxxxxxxx<br>xxxxxxxxxxxx | Yes/<br>No | xx/units/<br>xx/ | Yes | xxxxxxxxx/ | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/ |
| | | | (xxxxxxxxxxx) | | XX | | | xx<br>DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/ |
| XX | xxx | xx | xxxxxxxxx<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes/<br>Yes | xx/units/<br>xx/<br>xx | No | Other/<br>xxxxxxxxx | xx<br>DDMMMYYYY (xx)/<br>Ongoing |
| xx | XXX | | None | | | | | |

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient, start date and drug class. Program Name:

Date Generated: Page x of y

<sup>[</sup>a] WHO Drug Dictionary (Version WHODRUG Enhanced 201509, DDEB2) was used for coding.

<sup>[</sup>b] Relative to date of first dose of study treatment

# Listing 16.2.5.1 Study Drug Administration Safety Population

Treatment: Treatment 1

| Center | Patient | Dose No. | Start Date Time<br>(day)[a]/<br>Stop Date Time<br>(day)[a] | Full dose infused? | If no,<br>explain | Volume infused (mL) | Inpatient or<br>Outpatient? |
|---|---|---|---|---|---|---|---|
| xxxxx | xxx | xxx | DDMMMYYYY:HHMM (xx)/ DDMMMYYYY:HHMM (xx) | | xxx | Inpatient | |
| | | xxx | DDMMMYYYY:HHMM (xx)/ DDMMMYYYY:HHMM (xx) | Yes | xxx Outpatient | Outpatient | |

[a] Relative to date of first dose of study treatment

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient

Program Name:

Date Generated:

> Listing 16.2.5.2 Overall Compliance Safety Population

Treatment: Treatment 1

| Center | Patient | Visit | Actual number of | Planned number | Total Compliance | Duration of |
|---|---|---|---|---|---|---|
| | | | doses received | of doses | (%) | Exposure (days) |
| xxxxxx | xxx | ETP | XX | xx | XX.X | XX |
| | | EOT | | | | |
| | | TOC | | | | |

. . .

% compliance for each patient is calculated as 100\*Actual number of doses received / Planned number of doses
Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient
# Listing 16.2.5.3 Population Pharmacokinetic Safety Population

Treatment: Treatment 1

| Center | Patient | Visit | PK Time<br>Point | Was Sample<br>Collected? | Date and Time of Collectin (Day)[a] |
|---|---|---|---|---|---|
| xxxxxx | XXX | | | | DDMMMYYYY:HHMM (xx) |

[a] Relative to the day of first dose of study treatment Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Program Name: Date Generated:

Listing 16.2.6.1
Blood Culture Results
ITT Population

Treatment: Treatment 1

| Center | Patient | Visit | Was a<br>specimen<br>obtained?/<br>If no,<br>specify | Specimen<br>No. | Specimen<br>Type | Was<br>culture<br>performed? | If no,<br>reason/<br>Other,<br>specify | Did the culture grow an organism? | Accession<br>No. | Was the organism a pathogen? | Pathogen<br>Genus/<br>Species | Culture<br>Agent | MIC Panel result (mg/mL)/ Interpre- tation |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx | Baseline | Yes | XXX | Aerobic<br>blood | Yes | | Yes | xx | Yes | xxxxxx/<br>xxxx | xxxxx | 1/<br>Intermediate |
| | | Visit 2 | No/<br>xxxxxx | | | | | | | | | | |
| | | ETP | | | | No | Other/<br>xxxxx | | | | | | |
| | | EOT | | | | | | | | | | | |

. . .

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Program Name: Date Generated:

Listing 16.2.6.2 Signs and Symptoms of ABSSSI ITT Population

Treatment: Treatment 1

| Center | Patient | Visit | Date of<br>Assessment<br>(day)[a] | TEN | ERY | EDE | PUR | FLUC | IND | ULC | NEC | LOC | SWL | CHL | FEV |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | XXX | Baseline | DDMMMYYYY<br>(xx) | | | | | | | | | | | | |
| | | Visit 2 | DDMMMYYYY<br>(xx) | | | | | | | | | | | | |
| | | ETP | DDMMMYYYY<br>(xx) | | | | | | | | | | | | |
| | | Visit 4 | DDMMMYYYY<br>(xx) | | | | | | | | | | | | |
| | | EOT | DDMMMYYYY<br>(xx) | | | | | | | | | | | | |
| | | TOC | DDMMMYYYY<br>(xx) | | | | | | | | | | | | |

TEN=Tender to palpitation, ERY=Erythema, EDE=Edema, PUR=Purulent drainage/ discharge, FLUC=Fluctuance, IND=Induration, ULC=Ulceration, NEC=Necrotic tissue, LOC=Localized pain, SWL=Swelling, CHL=Chills, FEV=Fever.

[a] Relative to the day of first dose of study treatment

Programming Notes:

Repeat for all treatments. Sort by treatment, center and patient

Listing 16.2.6.3 Clinical Efficacy Assessment ITT Population

| Treatment. | Treatment | 7 |
|------------|-----------|---|

| Center | Patient | Visit | Date of<br>Assessment<br>(day) [a] | Total<br>lesion<br>size<br>(cm²) | Change of<br>lesion<br>size from<br>baseline | >=20% reduction in lesion size at ETP | >=90%<br>reduction<br>in lesion<br>size at<br>TOC | Clinical<br>outcome at<br>TOC |
|---|---|---|---|---|---|---|---|---|
| xxxxx | xxx | Baseline | DDMMMYYYY | XX.X | | NA | NA | NA |
| | | | (xx) | | | | | |
| | | ETP | DDMMMYYYY<br>(xx) | XX.X | XX.X | Yes | NA | NA |
| | | EOT | DDMMMYYYY<br>(xx) | xx.x | XX.X | NA | NA | NA |
| | | TOC | DDMMMYYYY<br>(xx) | xx.x | xx.x | NA | Yes | Cure |

[a] Relative to the day of first dose of study treatment

Programming Notes:

Programming notes: Repeat for all treatments. Sort by treatment, center, patient and visit.

# Listing 16.2.6.4.1 Microbiological Assessment - Patient Level ITT Population

Treatment: Treatment 1

| Center | Patient | Visit | Bacteriological |
|--------|---------|-------|-----------------|
| | | | Response |
| XXXXXX | XXX | ETP | XXXXXXX |
| | | EOT | XXXXXX |
| | | TOC | xxxxxx |
| xxxxxx | XXX | ETP | xxxxxx |
| | | EOT | XXXXXX |
| | | TOC | XXXXXX |

Programming Notes:

Programming notes: Repeat for all treatments. Sort by treatment,

center, patient and visit.

Listing 16.2.6.4.2
Microbiological Assessment - Pathogen Level
ITT Population

Treatment: Treatment 1

| Center | Patient | Visit | Pathogen | Bacteriological |
|--------|---------|-------|------------|-----------------|
| | | | | Response |
| XXXXXX | XXX | ETP | pathogen 1 | XXXXXX |
| | | | pathogen 2 | XXXXXX |
| | | EOT | pathogen 1 | XXXXXX |
| | | | pathogen 2 | XXXXXX |
| | | TOC | pathogen 1 | XXXXXX |
| | | | pathogen 2 | XXXXXX |
| XXXXXX | XXX | | | |

Programming Notes:

Programming notes: Repeat for all treatments. Sort by treatment,

center, patient and visit.

Program Name: Date Generated: Page x of y


Listing 16.2.6.5
Microbiological Assessment of Primary Infection Site - Gram Stain Results
ITT Population

Treatment: Treatment 1

| Center | Patient | Specimen No. | Date of<br>Collection<br>(day)[a] | Method of<br>Collection | Result of<br>Gram Stain |
|---|---|---|---|---|---|
| xxxxxx | xxx | XX | DDMMMYYYY (xx) | xxxxxxx | xxxxx |
| | | **** | | ************ | XXXXXX |
| | | | DDMMMYYYY (xx) | xxxxxxx | xxxxxx |
| | | | | | XXXXXX |
| | | | DDMMMYYYY (xx) | XXXXXXX | Not Done |

[a] Relative to the day of first dose of study treatment Programming Notes:

Programming notes: Repeat for all treatments. Sort by treatment, center, patient and visit.

# Listing 16.2.6.6 Significant Surgical Procedures ITT Population

Treatment: Treatment 1

| Center | Patient | Visit | Procedure<br>No. | Significant<br>Procedure | Other, specify | Date performed (day)[a] | Does the need of procedure reflect failure of antimicrobial therapy? |
|---|---|---|---|---|---|---|---|
| xxxxx | xxx | Visit 2<br>ETP<br>Visit 4<br>EOT<br>TOC | xx<br>xx<br>xx<br>xx<br>xx | Debridement<br>No procedure | | DDMMMYYYY (xx) | No |
| XXXXXX | XXX | | | | | | |

[a] Relative to the day of first dose of study treatment

Programming Notes:

Programming notes: Repeat for all treatments. Sort by treatment, center, patient and visit.

Listing 16.2.6.7

Death

ITT Population

Treatment: treatment 1

| Center | Patient | Date of final contact (day)[a] | Date of death<br>(day)[a] | Cause of<br>death | Death within 28<br>days of first<br>dose |
|---|---|---|---|---|---|
| xxxxxx | xxx<br>xxx | DDMMMYYYY (xx) DDMMMYYYY (xx) | DDMMMYYYY (xx) DDMMMYYYY (xx) | XXXXXXX | Yes<br>No |

[a] Relative to the day of first dose of study treatment

> Listing 16.2.6.8.1 Unblinding ITT Population

Treatment: treatment 1

| | | Date and time | Reason of | |
|---|---|---|---|---|
| | | of unblinding | unblinding/ | Unblinded by/ |
| Center | Patient | (day)[a] | Other, specify | Other, specify |
| XXXXXX | XXX | DDMMMYYYY: HHMM | xxxxxxx/ | xxxxxx/ |
| XXXXXX | XXX | DDMMMYYYY:HHMM (xx) | xxxxxxx/<br>xxxxxx | xxxxxx/<br>xxxxxxx |
| xxxxxx | | | * | · |

[a] Relative to the day of first dose of study treatment

> Listing 16.2.6.8.2 Unblinding Dose ITT Population

Treatment: treatment 1

| Center | Patient | Dose No. | Date and Time prepared (Day)[a] | Dosage prepared (mg) | Reason for dose adjustment |
|---|---|---|---|---|---|
| xxxxxx | xxx | xx | DDMMMYYYY:HHMM (xx) | xxx.x | xxxxxx |
| | | XX | DDMMMYYYY:HHMM (xx) | XXX.X | xxxxxx |

. . .

<sup>[</sup>a] Relative to the day of first dose of study treatment

Listing 16.2.7 Adverse Events Safety Population

Treatment: Treatment 1

| Center | Patient | AE No. | System Organ Class/<br>Preferred Term/<br>Verbatim [a] | Onset Date (day)[b]/<br>End Date (day)[b]/<br>Duration (days) | Treatment<br>emergent?/<br>Severity/<br>SAE? | Relationship<br>to Study<br>Drug/<br>ADR? | Treatment required? | Action<br>Taken[c] | Outcome |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxx | XX | *******************/ ***************** | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/<br>xx | Yes/<br>Mild | Not related/<br>No | Yes | xxx | Completely recovered |
| | | | *******************/ ***************** | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx)/<br>xx | Moderate | Probably not<br>related/<br>No | No | xxxx | Death |
| XXXXXX | xxx | xx | xxxxxxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx/<br>xxxxxx | DDMMMYYYY (xx)/<br>Ongoing | Severe | Probably<br>related/<br>Yes | Yes | xxxx | Ongoing |
| | | | | | | Related/<br>Yes | Yes | xxx | Recovered to stability |

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient, start date and SOC.

<sup>[</sup>a] Coded using MedDRA Dictionary (Version 18.1)

<sup>[</sup>b] Relative to the day of first dose of study treatment

### Listing 16.2.8.1 Laboratory Findings in Local Labs at Baseline - Hematology Safety Population

Treatment: Treatment 1

| Center | Patient | Age<br>(years)/<br>Gender | Test | Visit | Collection Date Time (day) [a] | Result | Units | Normal<br>Range | Out of<br>Range<br>[b] | Clinical<br>Significance<br>[b] |
|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX | xx/ Male | Hematocrit | Baseline | DDMMMYYYY<br>HH:MM (xx) | xxx.xxx | XXX | xxx - xxx | Н | CS |

. . .

[a] Relative to the day of first dose of study treatment

Note: Baseline is defined as the last scheduled or unscheduled value obtained prior to the first dose of treatment

[b] B = Baseline; H = Above upper limit of normal; L = Below lower limit of normal;

\* = Unscheduled value, not included in summary tables if post-dose.

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Include all Hematology tests (including C-reactive protein and LFT)

Listing 16.2.8.2

Laboratory Findings in Local Labs at Baseline - Chemistry Safety Population

Treatment: Treatment 1

| Center | Patient | Age<br>(years)/<br>Gender | Test | Visit | Collection<br>Date Time<br>Visit (day) [a] Result Units | | Normal<br>Range | Out of<br>Range<br>[b] | Clinical<br>Significance<br>[b] | |
|---|---|---|---|---|---|---|---|---|---|---|
| xx | XXX | xx/ Male | Albumin | Baseline | DDMMMYYYY<br>HH:MM (xx) | xxx.xxx | XXX | xxx - xxx | Н | CS |

. . .

[a] Relative to the day of first dose of study treatment

Note: Baseline is defined as the last scheduled or unscheduled value obtained prior to the first dose of treatment

[b] B = Baseline; H = Above upper limit of normal; L = Below lower limit of normal;

 $\star$  = Unscheduled value, not included in summary tables if post-dose.

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Include all Clinical Chemistry tests and creatinine clearance

### Listing 16.2.8.3 Laboratory Findings in Local Labs at Baseline - Urinalysis Safety Population

Treatment: Treatment 1

| Center | Patient | Age<br>(years)/<br>Gender | Test | Visit | Collection Date Time (day) [a] | Result | Units | Normal<br>Range | Out of<br>Range<br>[b] | Clinical<br>Significance<br>[b] |
|---|---|---|---|---|---|---|---|---|---|---|
| XX | XXX | xx/ Male | рН | Baseline | DDMMMYYYY<br>HH:MM (xx) | xxx.xxx | XXX | xxx - xxx | Н | CS |

. . .

[a] Relative to the day of first dose of study treatment

Note: Baseline is defined as the last scheduled or unscheduled value obtained prior to the first dose of treatment

[b] B = Baseline; H = Above upper limit of normal; L = Below lower limit of normal;

 $\star$  = Unscheduled value, not included in summary tables if post-dose.

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Include all Urinalysis tests

Listing 16.2.8.4

Laboratory Findings in Central Labs by Visit - Hematology Safety Population

Treatment: Treatment 1

| | | Age<br>(years)/ | | | Collection<br>Date Time | | SI | Normal | Out of<br>Range | Clinical<br>Significance |
|---|---|---|---|---|---|---|---|---|---|---|
| Center | Patient | Gender | Test | Visit | (day) [a] | Result | Units | Range | [b] | [b] |
| XXXXX | XXX | xx/ Male | Hematocrit | Baseline | DDMMMYYYY:HHMM(xx) | xxx.xxx | XXX | xxx - | Н | CS |
| | | | | ETP | DDMMMYYYY:HHMM (xx) | xxx.xxx | XXX | xxx - | L | NCS |
| | | | | Visit 4 | DDMMMYYYY:HHMM (xx) | xxx.xxx | XXX | xxx - | L | NCS |
| | | | | EOT | DDMMMYYYY:HHMM (xx) | xxx.xxx | XXX | xxx - | L | NCS |
| | | | | TOC | DDMMMYYYY:HHMM (xx) | xxx.xxx | XXX | xxx - | L | NCS |

. . .

Note: Baseline is defined as the last scheduled or unscheduled value obtained prior to the first dose of treatment

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Include all Hematology tests (including C-reactive protein and LFT)

<sup>[</sup>a] Relative to the day of first dose of study treatment

<sup>[</sup>b] B = Baseline; H = Above upper limit of normal; L = Below lower limit of normal;

<sup>\* =</sup> Unscheduled value, not included in summary tables if post-dose.

Listing 16.2.8.5
Laboratory Findings in Central Labs by Visit - Chemistry

Safety Population

Treatment: Treatment 1

| | | Age | | | Collection | | | _ | Out of | Clinical |
|---|---|---|---|---|---|---|---|---|---|---|
| | | (years)/ | | | Date Time | | SI | Normal | Range | Significance |
| Center | Patient | Gender | Test | Visit | (day) [a] | Result | Units | Range | [b] | [b] |
| XXXXX | xxx | xx/ Male | Albumin | Baseline | DDMMMYYYY:HHMM(xx) | xxx.xxx | xxx | xxx - xxx | Н | CS |
| | | | | ETP | DDMMMYYYY:HHMM (xx) | xxx.xxx | xxx | XXX - XXX | L | NCS |
| | | | | Visit 4 | DDMMMYYYY:HHMM (xx) | xxx.xxx | xxx | XXX - XXX | L | NCS |
| | | | | EOT | DDMMMYYYY:HHMM (xx) | xxx.xxx | xxx | XXX - XXX | L | NCS |
| | | | | TOC | DDMMMYYYY:HHMM (xx) | xxx.xxx | XXX | XXX - XXX | L | NCS |

. . .

Note: Baseline is defined as the last scheduled or unscheduled value obtained prior to the first dose of treatment

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Include all Clinical Chemistry tests

Program Name: Date Generated:

<sup>[</sup>a] Relative to the day of first dose of study treatment

<sup>[</sup>b] B = Baseline; H = Above upper limit of normal; L = Below lower limit of normal;

<sup>\* =</sup> Unscheduled value, not included in summary tables if post-dose.

Listing 16.2.8.6
Laboratory Findings in Central Labs by Visit - Urinalysis
Safety Population

Treatment: Treatment 1

| | | Age<br>(years)/ | | | Collection<br>Date Time | | SI | Normal | Out of<br>Range | Clinical<br>Significance |
|---|---|---|---|---|---|---|---|---|---|---|
| Center | Patient | Gender | Test | Visit | (day) [a] | Result | Units | Range | [b] | [b] |
| XXXXX | XXX | xx/ Male | рН | Baseline | DDMMMYYYY:HHMM (xx) | xxx.xxx | xxx | xxx - xxx | Н | CS |
| | | | | ETP | DDMMMYYYY:HHMM (xx) | xxx.xxx | xxx | xxx - xxx | L | NCS |
| | | | | Visit 4 | DDMMMYYYY:HHMM (xx) | xxx.xxx | xxx | xxx - xxx | L | NCS |
| | | | | EOT | DDMMMYYYY:HHMM (xx) | xxx.xxx | XXX | xxx - xxx | L | NCS |
| | | | | TOC | DDMMMYYYY:HHMM (xx) | xxx.xxx | XXX | xxx - xxx | L | NCS |

. . .

Note: Baseline is defined as the last scheduled or unscheduled value obtained prior to the first dose of treatment

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Include all Urinalysis tests

<sup>[</sup>a] Relative to the day of first dose of study treatment

<sup>[</sup>b] B = Baseline; H = Above upper limit of normal; L = Below lower limit of normal;

<sup>\* =</sup> Unscheduled value, not included in summary tables if post-dose.

> Listing 16.2.9 Vital Signs Safety Population

Treatment: Treatment 1

| Center | Patient | Visit | Vital Signs | Values |
|--------|---------|-----------|---------------------------|----------|
| xxxxxx | xxx | Baseline | Systolic BP (mm Hq) | Not Done |
| | | 200022110 | Diastolic BP (mm Hg) | Not Done |
| | | | Heart Rate (beat/min) | XX |
| | | | Respiration (breaths/min) | XX |
| | | | Body Temperature (°C) | XX.X |
| | | | Height (cm) | XXX.X |
| | | | Weight (kg) | XX.X |
| | | | BMI (kg/m^2) | XX.X |

<Continue for remaining post-baseline time points>

XXXXXX XXX

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Program Name: Date Generated:

Listing 16.2.10.1 ECG Results Safety Population

Treatment: Treatment 1

| | | | Assessment | | | | |
|---|---|---|---|---|---|---|---|
| Center | Patient | Visit | Date (day)[a] | ECG Measurements | Units | Values | Interpretation |
| XXXXXX | XXX | Baseline | DDMMMYYYY (xx) | Median Heart | beats/min | XXX | |
| | | | | Rate | | | |
| | | | | Median RR | msec | Not Done | |
| | | | | Interval | | | |
| | | | | Median PR | msec | XXX | |
| | | | | Interval | | | |
| | | | | Median QRS | msec | XXX | |
| | | | | Duration | | | |
| | | | | Median QT | msec | XXX | |
| | | | | Interval | | | |
| | | | | Median QTcB [b] | msec | XXX | |
| | | | | Interval | | | |
| | | | | Median QTcF [b] | msec | XXX | |
| | | | | Interval | | | |

<Continue for remaining post-baseline time points>

XXXXXX XXX

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit. Date Generated:

Program Name:

<sup>[</sup>a] Relative to the day of first dose of study treatment

<sup>[</sup>b] QTcB = Bazett corrected QT interval; QTcF = Fridericia corrected QT interval.

Listing 16.2.10.2 ECG Assessment

Safety Population

Treatment: Treatment 1

| TTCGCINC | iic. iicacii | 0110 1 | | | | |
|---|---|---|---|---|---|---|
| Center | Patient | Visit | Assessment<br>Date (day)<br>[a] | Clinical significance [b] | Marked QT/QTc<br>prolongation<br>[c] | Comments |
| xxxxxx | xxx | Baseline | DDMMMYYYY<br>(xx) | Normal | | |
| | | | | Abnormal, NCS<br>Abnormal, CS | Yes | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxx | XXX | | | Not Done | | |

- [a] Relative to the day of first dose of study treatment
- [b] NCS=not clinically significant, CS=clinically significant.
- [c] marked QT/QTc prolongation is defined as median QTcF value >500 msec and/or >60 msec different from the pre-dose baseline value.

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit.

Program Name: Date Generated:

# Listing 16.2.11 Physical Examination Results Safety Population

Treatment: Treatment 1

| Center | Patient | Visit | Assessment Date (day) [a] | Any PE performed? | Body System | Examined? | Reason for no PE exam/ Other, specify | Overall<br>Results |
|---|---|---|---|---|---|---|---|---|
| | | | | | <del>*</del> * | | , 11 1 1 | <del>-</del> |
| xxxxxx | XXX | Baseline | DDMMMYYYY (xx) | Yes | Cardiovascular | Yes | Xxxxxx/ | Abnormal |
| | | | | | Respiratory | No | | |
| | | | | | Gastrointestinal | Yes | | |
| | | | | | Skin (other than | Yes | | |
| | | | | | primary site of | | | |
| | | | | | infection) | | | |
| | | | | | Musculoskeletal | Yes | | |
| | | | | | Endocrine | Yes | | |
| | | | | | Neurological | Yes | | |
| | | | | | HEENT | Yes | | |
| | | | | | Genitourinary | Yes | | |
| | | Visit 2 | | | | | | |

[a] Relative to the day of first dose of study treatment

Programming Notes:

Repeat for all treatments. Sort by treatment, center, patient and visit. Only present abnormal body systems. If all body systems are normal at a visit, output "None" in Body System Abnormalities column for the visit.

| Client Name: | Motif BioSciences | <b>Covance Study ID:</b> | 000000145670 |
|---|---|---|---|
| Client Protocol No.: | ICL-24-ABSSSI2 | Meaningful Date (for eTMF only): | 2 October 2017 |
| <b>Investigator Name</b> | NA | Site No.: | NA |
| Artifact Name: | Plan – SAP | Artifact No: | 01.1.31 |
| Topic: | Pre-unblinding decisions on efficacy analyses | | |

#### **Description:**

This Note to File documents pre-database lock decisions on handling efficacy endpoints with regard to the additional rule in selecting clinical response (Cure, Non-cure) and hard-coding of a patient.

Changes from blinded review of 28 September 2017 are detailed in the attached patient profiles, one for antibiotics of cure patients, one for surgical procedures of cure patients, one for antibiotics of indeterminate/failure patients, and one for surgical procedures of indeterminate/failure patients along with clinical outcome at TOC (without lesion):

- Copy of Motif2\_Antibiotics\_CLONITOC\_Indeterminate\_Failure\_28Sep2017\_PM 28Sep17\_dh.xlsx,
- Copy of Motif2\_Procedures\_CLONITOC\_Indterminate\_Failure\_28Sep2017\_PM 28Sep17 dh.xlsx;
- o Copy of Motif2\_Antibiotics\_CLONITOC\_Cure\_28Sep2017\_PM 28Sep17 dh.xlsx. Columns I to N are those criteria used to derive clinical outcome in the antibiotics spreadsheet.

The clinical outcome has used the most current updated rules from Revive 1 (new added failure rules from Revive 1 NTF).

As a result of the medical review of Copy of

Motif2\_Antibiotics\_CLONITOC\_Cure\_28Sep2017\_PM 28Sep17 dh.xlsx, the criteria for determining efficacy response were refined for programming.

- O Cure to Indeterminate: If subject received more than one dose of a short acting (i.e., q12h dosing or less) systemic antibiotic(s) active against Gram-positive pathogens (Appendix F) within the last 7 days, unless there is documented evidence of treatment failure OR demonstrated resistance of Gram-positive pathogens to the prior antibiotic therapy (antibiotics given for surgical prophylqxis are not included in this), the subject should be categorized as non-cure (see exclusion criteria 6 page 34 of the protocol). Given that the antibiotics are given before study drug, they should be categorized as non-cure (indeterminate).
- O The above rule is complex to implement in programming so a list of subjects who took more than 1 short acting antibiotics within 7 days of randomization was reviewed by Covance medical monitor who determined the patients that would follow the above rule. We used the list in a spreadsheet format to implement Clinical outcome of seleted subjects in programming ADEFF dataset. This process is similar to hardcoding, and the subjects that are changed to 'Indeterminate' are:

| Client Name: | Motif BioSciences | <b>Covance Study ID:</b> | 000000145670 |
|---|---|---|---|
| Client Protocol No.: | ICL-24-ABSSSI2 | Meaningful Date (for eTMF only): | 2 October 2017 |
| <b>Investigator Name</b> | NA | Site No.: | NA |
| Artifact Name: | Plan – SAP | Artifact No: | 01.1.31 |
| Topic: | Pre-unblinding decisions on efficacy analyses | | |

201001135, 201003009, 201003011, 201008010, 234004002, 236006002, 243006011, 243006012, 243006016, 246002021, 246002024, 246002028, 246003017, 254009001, 254009003.

Additionally, for the draft topline of 2 October 2017, Covance performed a hard coding for subject 234003001 (the one with indication=Hand lesion which is not the index of infection). Covance medical monitor suggested adding 'secondary' to the Primary\_secondary spreadsheet, but the programs on both production and QC side still does not output it to Indeterminate, so Covance programmatically pulled hand-lesion indication in order to output it as Indeterminate. This will be updated to not hardcode for final topline by having the Covance medical monitor update the spread sheet with non-infection indications.

#### Documents affected:

- o SAP: Added condition for the response for Indeterminate: If subject received more than one dose of a short acting (i.e., q12h dosing or less) systemic antibiotic(s) active against Gram-positive pathogens (Appendix F) within the last 7 days, unless there is documented evidence of treatment failure OR demonstrated resistance of Gram-positive pathogens to the prior antibiotic therapy (antibiotics given for surgical prophylqxis are not included in this), the subject should be categorized as non-cure (see exclusion criteria 6 page 34 of the protocol). Given that the antibiotics are given before study drug, they should be categorized as non-cure (indeterminate).
- EDC database: Not affected.
- Analysis dataset specification: ADEFF specification will be updated to reflect the above rule. ADEFF will be affected as stated above.
- TFL: Draft Top-line TFL
- Encl: Spreadsheet for determining Indeterminate and Failure responses: Copy of Motif2\_Antibiotics\_CLONITOC\_Cure\_28Sep2017\_PM 28Sep17 dh.xlsx.

| Client Name: | Motif BioSciences | Covance Study ID: | 000000145670 |
|---|---|---|---|
| Client Protocol No.: | ICL-24-ABSSSI2 | Meaningful Date (for eTMF only): | 2 October 2017 |
| <b>Investigator Name</b> | NA | Site No.: | NA |
| Artifact Name: | Plan – SAP | Artifact No: | 01.1.31 |
| Topic: | Pre-unblinding decisions on efficacy analyses | | |

### Note to File approved by:

| Signature | 2 October 2017 Date |
|---|---|
| David Huang, MD, PhD, FACP, FIDSA / Chief Medical Officer | |
| Printed Name/Title | |
| Note to File completed by: | |
| Toyoko Oguri | 2 October 2017 |
| Typed Name | Date |
| Senior Manager, Biostatistics and Statistical Programming | |

#### **Instructions:**

Title

This TMF File Note should only be used to document situations that do not fall under the current CDS procedures for documenting deviations, issues and/or complaints.

The investigator name and site number should match CTMS.

For eTMF studies, when a NTF is written to clarify or support an artifact filed in eTMF, the NTF is uploaded with the same artifact name and meaningful date as the artifact the NTF was written to clarify. In eTMF, if a NTF was written to clarify a process or provide supportive information and is filed at the Trial, Country or Site level, the artifact is filed at the NTF artifact location and the meaningful date is the date of the NTF.

Complete each section. If a section does not apply, write "N/A".

| Client Name: | Motif BioSciences | <b>Covance Study ID:</b> | 000000145670 |
|---|---|---|---|
| Client Protocol No.: | ICL-24-ABSSSI2 | Meaningful Date (for eTMF only): | 6 October 2017 |
| <b>Investigator Name</b> | NA | Site No.: | NA |
| Artifact Name: | Plan – SAP | Artifact No: | 01.1.31 |
| Topic: | Post-unblinding decisions on efficacy analyses | | |

#### **Description:**

This Note to File documents post-database lock decisions on programmatically handling efficacy endpoints with regard to (1) the procedure "dressing change" not to be considered a significant surgical procedure, per the protocol; and (2) hard-coding of a patient.

- 1. Procedures that were checked as significant in EDC (thus picked as Failure of antimicrobial therapy) should have been considered as routine procedure, specifically dressing change. The procedure "DRESSING CHANGE" should not be considered a significant procedure and thus patients with such a procedure should not be considered as Clinical Failure as long as there are no other criteria prohibiting such patients from being a Cure. Such cases were revised programmatically.
- 2. Failure to Indeterminate: Patient 240006002 Covance medical expert confirmed that this patient outcome should be Indeterminate. It was recommend to hard code for this subject. This will be applied to all Clinical Outcome parameters including clinical outcome with lesion size.
  - 1) SAP: Add condition to procedure of DRESSING CHANGE as not a significant procedure.
  - 2) EDC database: Not affected.
  - 3) Analysis dataset specification: ADEFF specification will be updated to reflect the above rule.
  - 4) TFL: Final Top-line TFL
  - 5) Encl: none.

| Client Name: | Motif BioSciences | <b>Covance Study ID:</b> | 000000145670 |
|---|---|---|---|
| Client Protocol No.: | ICL-24-ABSSSI2 | Meaningful Date (for eTMF only): | 6 October 2017 |
| <b>Investigator Name</b> | NA | Site No.: | NA |
| Artifact Name: | Plan – SAP | Artifact No: | 01.1.31 |
| Topic: | Post-unblinding decisions on efficacy analyses | | |

### Note to File approved by:

| Dwly | 10/6/2017 |
|---|---|
| Signature | Date |
| David Huang, MD, PhD, FACP, FIDSA / Chief Medical Officer | |
| Printed Name/Title | |
| Note to File completed by: | |
| Toyoko Oguri | 2 October 2017 |
| Typed Name | Date |
| Senior Manager, Biostatistics and Statistical Programming | |

#### Instructions:

Title

This TMF File Note should only be used to document situations that do not fall under the current CDS procedures for documenting deviations, issues and/or complaints.

The investigator name and site number should match CTMS.

For eTMF studies, when a NTF is written to clarify or support an artifact filed in eTMF, the NTF is uploaded with the same artifact name and meaningful date as the artifact the NTF was written to clarify. In eTMF, if a NTF was written to clarify a process or provide supportive information and is filed at the Trial, Country or Site level, the artifact is filed at the NTF artifact location and the meaningful date is the date of the NTF.

Complete each section. If a section does not apply, write "N/A".

| Client Name: | Motif BioSciences | Covance Study ID : | 000000145670 |
|---|---|---|---|
| Client Protocol No.: | ICL-24-ABSSSI2 | Meaningful Date (for eTMF only): | 6 October 2017 |
| Investigator Name | NA | Site No.: | NA |
| Artifact Name: | Plan – SAP | Artifact No: | 01.1.31 |
| Topic: | Post-unblinding decisions on efficacy analyses | | |

#### **Description:**

This Note to File documents decisions on programmatically handling efficacy endpoints with regard to (1) the procedure "dressing change" not to be considered a significant surgical procedure, per the protocol; and (2) hard-coding of a patient. These decisions were made after review of patient data in a blinded fashion after the database was locked and randomization codes were applied. The patient data did not have any treatment identifying information.

- 1. Procedures that were checked as significant in EDC (thus picked as Failure of antimicrobial therapy) should have been considered as routine procedure, specifically dressing change. The procedure "DRESSING CHANGE" should not be considered a significant procedure and thus patients with such a procedure should not be considered as Clinical Failure as long as there are no other criteria prohibiting such patients from being a Cure. Such cases were revised programmatically.
- 2. Failure to Indeterminate: Patient 240006002 Covance medical expert confirmed that this patient outcome should be Indeterminate. It was recommend to hard code for this subject. This will be applied to all Clinical Outcome parameters including clinical outcome with lesion size.
  - 1) SAP: Add condition to procedure of DRESSING CHANGE as not a significant procedure.
  - 2) EDC database: Not affected.
  - 3) Analysis dataset specification: ADEFF specification will be updated to reflect the above rule.
  - 4) TFL: Final Top-line TFL
  - 5) Encl: none.

| Client Name: | Motif BioSciences | <b>Covance Study ID:</b> | 000000145670 |
|---|---|---|---|
| Client Protocol No.: | ICL-24-ABSSSI2 | Meaningful Date (for eTMF only): | 6 October 2017 |
| <b>Investigator Name</b> | NA | Site No.: | NA |
| Artifact Name: | Plan – SAP | Artifact No: | 01.1.31 |
| Topic: | Post-unblinding decisions on efficacy analyses | | |

### Note to File approved by:

| Dwly | 10/6/2017 |
|-----------------------------------------------------------|----------------|
| \$ignature | Date |
| David Huang, MD, PhD, FACP, FIDSA / Chief Medical Officer | |
| Printed Name/Title | |
| Note to File completed by: | |
| Toyoko Oguri | 2 October 2017 |
| Typed Name | Date |
| Senior Manager, Biostatistics and Statistical Programming | |

Title

#### Instructions:

This TMF File Note should only be used to document situations that do not fall under the current CDS procedures for documenting deviations, issues and/or complaints.

The investigator name and site number should match CTMS.

For eTMF studies, when a NTF is written to clarify or support an artifact filed in eTMF, the NTF is uploaded with the same artifact name and meaningful date as the artifact the NTF was written to clarify. In eTMF, if a NTF was written to clarify a process or provide supportive information and is filed at the Trial, Country or Site level, the artifact is filed at the NTF artifact location and the meaningful date is the date of the NTF.

Complete each section. If a section does not apply, write "N/A".

| Client Name: | Motif BioSciences | Covance Study ID : | 000000145416 |
|---|---|---|---|
| Client Protocol No.: | ICL-23-ABSSSI1 | Meaningful Date (for eTMF only): | 2 Dec 2017 |
| Investigator Name | NA | Site No.: | NA |
| Artifact Name: | Plan - SAP | Artifact No: | 01.1.31 |
| Topic: | Hard coding of mITT population for sensitivity analysis | | |

#### **Description:**

This Note to File contains addition of mITT for Sensitivity Analysis population resulting in 3 additional subjects to be included in the original Microbiological intent-to-treat (mITT) population.

The mITT for Sensitivity Analyis consists of patients meeting mITT criteria who had Gram+baseline pathogen identified in infection site or blood culture.

Subjects 101011133, 101011137 and 137003010 are included in mITT population based on clinical assessment review by Covance medical monitor and sponsor medical expert of blood culture for sensitivity analysis.

| USUBJID | Blood_Cultur | | Infection Culture1 | Infection | Culture2 | Conclusion | Motif Comment |
|---|---|---|---|---|---|---|---|
| ICL-23-ABSSSI1-101011133 | VISIT 4.2 | | | | | questionable | Add |
| ICL-23-ABSSSI1-101011133 | VISIT 4.2 | | | | | | |
| ICL-23-ABSSSI1-101011137 | VISIT 3 | | | | | | Add |
| ICL-23-ABSSSI1-101011137 | VISIT 1 | Υ | | | | | |
| ICL-23-ABSSSI1-137003010 | VISIT 1 | Υ | | | | consider adding | Add |

| Note to File approved by: | |
|---|---|
| Sarty | December 4, 2017 |
| Signature | Date |
| David Huang, MD, PhD, FACP, FIDSA / Chief Medical Officer, Motif BioSciences, | Inc |
| Printed Name/Title | |
| Note to File completed by: | |
| Toyoko Oguri | |
| Typed Name | Date |
| Senior Manager, Biostatistics | |
| Title | |

Date Jol/

| Client Name: | Motif BioSciences | Covance Study ID: | 000000145416 |
|---|---|---|---|
| Client Protocol No.: | ICL-23-ABSSSI1 | Meaningful Date (for eTMF only): | 2 Dec 2017 |
| Investigator Name | NA | Site No.: | NA |
| Artifact Name: | Plan - SAP | Artifact No: | 01.1.31 |
| Topic: | Hard coding of mITT population for sensitivity analysis | | |

### Note to File completed by:

Toyoko Oguri Typed Name

Senior Manager, Biostatistics

| Client Name: | Motif BioSciences | Covance Study ID : | 000000145416 |
|---|---|---|---|
| Client Protocol No.: | ICL-23-ABSSSI1 | Meaningful Date (for eTMF only): | 8 Dec 2017 |
| Investigator Name | NA | Site No.: | NA |
| Artifact Name: | Plan - SAP | Artifact No: | 01.1.31 |
| Topic: | Define microbiological Per-Protocol Population and recurrent infection | | |

#### **Description:**

This Note to File clarifies the definition of microbiological Per-Protocol population (mPP) population in the protocol and the SAP and the definition of bacteriological response of recurrent infection.

The mPP definition from the protocol and SAP was:

All mITT patients who receive at least 80% of their planned doses and provide adequate data for assessment for each of the following time points: ETP, EOT, and TOC.

The mPP definition is clarified to include the criteria for the PP population:

All PP patients who have a Gram-positive baseline bacteria pathogen identified as the cause of ABSSSI.

In addition, the microbiological response definition in the SAP for recurrent infection is clarified to be defined as: A pathogen that is same as the baseline pathogen isolated only after the EOT visit outcome was cure and was either eradication or presumed eradication. This was correctly programmed in the tables as defined.

| N 700 | |
|---|---|
| Note to File approved by: | |
| Saxby | December 8, 2017 |
| Signature | Date |
| David Huang, MD, PhD, FACP, FIDSA / Chief Medical Printed Name/Title | Officer, Motif BioSciences, Inc |
| Note to File completed by: | |
| Toyoko Oguri | |
| • | Date |
| Toyoko Oguri Typed Name Senior Manager, Biostatistics | Date |

| Client Name: | Motif BioSciences | Covance Study ID: | 000000145416 |
|---|---|---|---|
| Client Protocol No.: | ICL-23-ABSSSI1 | Meaningful Date (for eTMF only): | 8 Dec 2017 |
| Investigator Name | NA | Site No.: | NA |
| Artifact Name: | Plan - SAP | Artifact No: | 01.1.31 |
| Topic: | Define microbiological Per-Protocol Population and recurrent infection | | |

#### Description:

This Note to File clarifies the definition of microbiological Per-Protocol population (mPP) population in the protocol and the SAP and the definition of bacteriological response of recurrent infection.

The mPP definition from the protocol and SAP was:

All mITT patients who receive at least 80% of their planned doses and provide adequate data for assessment for each of the following time points: ETP, EOT, and TOC.

The mPP definition is clarified to include the criteria for the PP population:

All PP patients who have a Gram-positive baseline bacteria pathogen identified as the cause of ABSSSI.

In addition, the microbiological response definition in the SAP for recurrent infection is clarified to be defined as: A pathogen that is same as the baseline pathogen isolated only after the EOT visit outcome was cure and was either eradication or presumed eradication. This was correctly programmed in the tables as defined.

### Note to File approved by:

| Signature | Date |
|---|---|
| David Huang, MD, PhD, FACP, FIDSA / Chief Medical Officer, Motif BioScient | nces, Inc |
| Printed Name/Title | |
| Note to File completed by: | |
| Toyoko Oguri Typed Name | 8 Dec 2017 |
| V | Date |
| Senior Manager, Biostatistics | |
| Title | |